### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD

• Adult Patient or • Parent, for Minor Patient

INSTITUTE: National Institute of Child Health and Human Development

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome

Continuing Review Approved by the IRB on 01/24/18

Amendment Approved by the IRB on 07/13/18 (S)

Date Posted to Web: 08/03/18

Standard

### **INTRODUCTION**

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

### Purpose of this Study

Approximately 30% of adults in the US have a body mass index (BMI) over 30 kg/m², and are at greater risk for a number of medical problems, including high blood pressure, high blood cholesterol, high triglyceride levels, high blood sugar (diabetes) and heart disease. It is thought that being overweight leads to a state of low-level inflammation and this inflammation may actually lead to some of the medical problems associated with obesity. The purpose of this study is to find out if a medication called colchicine can improve metabolism in adults who have medical complications of their high body weight (these complications are sometimes called the "metabolic syndrome"), but who have not yet developed high blood sugar (diabetes).

### **PATIENT IDENTIFICATION**

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent (1)

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Colchicine is an anti-inflammatory medication that has been used for centuries in the treatment of gout. From animal studies and human studies there is some evidence that anti-inflammatory medicines like colchicine may improve the pancreas's ability to secrete insulin and the body's ability to regulate sugar. We ask you to join our study, so we can find out whether colchicine can improve sugar regulation and metabolic parameters.

If you qualify and agree to participate, you will be one of 40 people assigned by chance to take either colchicine or placebo capsules by mouth twice a day for 3 months. The colchicine capsules will come in the same dose that is available in pharmacies and is prescribed for a disease called "gout": 0.6 milligrams. The placebo capsules look just like the colchicine capsules, but do not contain any colchicine. You will have a 50% chance of being assigned to take colchicine.

This study is designed to be 'double-blind': neither the doctors nor the study participants will know who is taking colchicine capsules and who is taking placebo. Only the NIH pharmacy will know whether a study participant is receiving colchicine or placebo. Unless it becomes medically necessary, the participants and the doctors will not be told until the study is completed (when no participant is still taking colchicine). The purpose of the 'double blinding' is to make sure we avoid bias on the part of the people involved in the study. When the study is completed, we will send all participants information about the results, and tell them whether they were taking colchicine or placebo capsules.

Study participants will need to come to the NIH Clinical Center for four outpatient visits, with an optional fifth outpatient visit. It is important that participants arrive fasting (no food or beverages besides water) to each of these visits. Participants will be compensated for their time and inconvenience (see below: *Compensation* on page 5).

### **Study Population**

We wish to recruit 40 overweight adults.

### **Who Can Be in This Study**

You may be eligible for this research study if you are greater than 18 years old, have a body mass index that is at least 30 kg/m<sup>2</sup> (calculated by dividing weight in kg by height in meters squared), weigh less than 450 lbs, and are in good general health. You also have to meet certain levels for insulin resistance and inflammation, as measured by lab testing, to participate in the full study. If you are a woman of child-bearing age, you will be asked to use an effective form of birth control before participating in this study.

### Who May Not Be In This Study

You may not be eligible for this study if you have a major medical illness that would interfere with study tests or measurements, such as heart, kidney, liver, lung, blood, gut, or endocrine diseases, or uncontrolled high blood pressure. If you are currently using a medication that affects sugar and fat metabolism or absorption in your body, or a medicine that should not be taken with colchicine, you may not be eligible to participate. Also individuals who are pregnant or nursing, or planning to become pregnant, have had a recent weight change greater than 3% of total body weight, have been using weight reducing medications, have recently used colchicine, have a known allergy to colchicine, or use tobacco or nicotine (e.g. e-cigarettes) products will not be recruited for this study. Individuals with a history of keloid formation (who easily develop scars on their skin after an injury) are advised not to take part in this study.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

### **Procedures of the study**

The study consists of four outpatient visits: an **outpatient screening visit** at the Clinical Center to determine eligibility, a **baseline visit** to study your metabolism before the intervention, a **short outpatient** visit to check how you are feeling, and a **final visit** 3 months after the baseline visit look for changes after the intervention. Upon completing the final visit, you have the option to return 3 months later to come for another **washout visit**. This visit will look to see if the changes from the intervention continue to last even after stopping the study medication. You will be randomized to receive colchicine or placebo on the day you complete the baseline visit.

### **Outpatient Screening Visit**

This visit will take about 3 hours to complete. You will be seen on a weekday in the Clinical Center at the National Institutes of Health. We ask that you remain fasting for 10 hours before coming to the clinic and have nothing to eat or drink except water that morning. During this visit, we will perform the following:

- 1. **Protocol review and signing of consent form**. We will go over the study in detail, and answer any questions. The consent form will need to be signed before you can take part in the study.
- 2. **Complete medical history and physical exam,** with weight, height, and blood pressure measurement.
- 3. An **EKG** will be performed to examine your heart function.
- 4. **Fasting blood tests** to ensure that you are in good health. The analysis will examine blood cell count, liver and kidney function, cholesterol levels, blood sugar and insulin levels, thyroid tests, inflammation level, as well as reserve blood samples to be preserved for additional possible research tests. We will also plan to do tests to find out if you have any differences in genes that may be important for metabolism and body weight. In addition to looking at some genes we already think are important for body weight, we will use new DNA sequencing technology that will look at all the human genes we know about. This is known as exome and genome sequencing. This new technology allows us to look at DNA in great detail.
- 5. **Urine sample collection** to ensure that your kidneys work normally, that you are not taking any illicit drugs, and a pregnancy test (for women of childbearing age).
- 6. **Oral glucose tolerance test**. We will perform a test to examine whether you have diabetes, called a 2-hour glucose tolerance test. You will drink a cup of sugar water and then will have your blood drawn 1 and 2 hours later to look at your blood sugar level.
- 7. **Dual energy x-ray absorptiometry (DEXA)** to look at your body composition. The test involves lying still on a table while a small camera passes over your body. The dose of the x-ray is much less than the amount you would get from a normal chest x-ray. The total amount of time to do this test will be about 20-30 minutes.

### Baseline Visit

PATIENT IDENTIFICATION

If you qualify for participation in the study, you will be scheduled for the baseline visit. We ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink except water that morning</u>. You will be seen on

**MEDICAL RECORD** 

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement. A questionnaire will also be performed.
- 2. **Fasting blood tests** to look at your baseline metabolic and inflammatory levels, as well as reserve blood samples to be preserved for additional possible research tests including a sample for future genetic analysis. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection.** We will obtain two stool samples to save for future experiments. As part of this collection, we will ask you to keep track of your diet for 24 hours on a form that will be provided to you, as diet can affect the results of the stool testing. You will also go over this "food record" in person with a nutritionist.
- 4. **Urine sample collection** as described before. We will also collect urine over your eight hours of testing to save for future experiments.
- 5. **Frequently sampled intravenous glucose tolerance test (FSIVGTT)**. This study tells us a lot about how sugar is used by your body, how well your insulin works, and how sensitive your body is to insulin. The FSIVGTT study is done while you rest in bed. A second IV line will be placed in your arm. We will give you some sugar water into one IV over a 2 minute period. We will then draw blood samples from the other IV at -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes (a total of 3 hours) to measure sugar and insulin levels. Exactly 20 minutes into the test, we will give you a small amount of insulin through the IV. A physician or nurse practitioner will be present during the first hour of the study. You can watch TV during this test.
- 6. **Computed Tomography (CT) Scan** of the abdomen to look at where you tend to store your fat. The test involves lying still on a movable table which passes through a large ring where the camera sits. The test does involve radiation, but because we only need to take a snapshot of your abdomen, the method that will be used minimizes your exposure. The total amount of time to do this test will be about 20-30 minutes.
- 7. **Subcutaneous Fat Biopsy**. To examine the level of certain molecules in your fat tissue, a small sample of fat tissue will be taken from under the skin of your abdomen via a "mini-liposuction" technique. Lidocaine, a local anesthetic, is used to numb the area. A needle will be used to remove a piece of fat tissue measuring about 1 ½ teaspoons. A bandage is then applied to the site of needle insertion. We can give you some mild pain medication such as Tylenol, or stronger medication if needed, after the biopsy. The biopsy will be taken from a place on your body that is normally covered and not easily seen.
- 8. **Dispense Study Medication**. You will be given approximately an 8-week supply of study medication to be taken two times a day (morning and late afternoon/evening) at home. The medication can be taken with or without food. We will give you a reminder alarm to help you remember when to take your medicine. If you forget to take a dose, then take it as soon as you remember. But if it is within 4 hours of the time for your next dose, do not take a double dose. Just skip the missed dose.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

### **Short Outpatient Visit**

To make sure that you doing well taking the medication, you will be seen on a weekday in the Clinical Center at the National Institutes of Health. This visit will take about 2 hours to complete. We ask that you **bring your bottle of pills** with you. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.
- 2. **Fasting blood tests** to ensure that you are in good health, to examine your inflammation levels, as well as reserve blood samples to be preserved for additional possible research tests.
- 3. **Urine sample collection** as described before.
- 4. **Dispense Study Medication**. We will give you another bottle of study medication (about 8 weeks' worth) to last you until the Final (3 month) Visit. As before, if you forget to take a dose, then take it as soon as you remember. But if it is within 4 hours of the time for your next dose, do not take a double dose. Just skip the missed dose.

### Final Visit

We will ask you to bring your bottle with any leftover pills to your final visit appointment. We ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink except water that morning</u>. You will be seen on a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.
- 2. **Fasting blood tests** as described before. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection** as described before.
- 4. **Urine sample collection** as described before.
- 5. Frequently sampled intravenous glucose tolerance test (FSIVGTT) as described before.
- 6. **DEXA Scan** as described before.
- 7. **CT Scan** as described before.
- 8. **Subcutaneous Fat Biopsy** as described before
- 9. **Exit questionnaire** to tell us about your experience of participating in our protocol.

### **Optional Washout Visit**

PATIENT IDENTIFICATION

Because we would like to see if colchicine will continue to have lasting positive effects on your glucose regulation, metabolism, inflammation, and/or cardiovascular health even after you've stopped taking it, we invite patients to return to the NIH Clinical Center 3 months after finishing the study medication for repeat testing.

As before, we ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink</u> <u>except water that morning</u>. You will be seen on a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

2. **Fasting blood tests** as described before. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.

- 3. **Stool sample collection** as described before.
- 4. **Urine sample collection** as described before.
- 5. Frequently sampled intravenous glucose tolerance test (FSIVGTT) as described before.
- 6. **DEXA Scan** as described before.
- 7. **CT Scan** as described before.
- 8. Subcutaneous Fat Biopsy as described before

When the study is complete, you will return to the care of your regular physician. Participation in this study does not commit NIH to your long term care.

### **Results of Tests at the NIH**

We will be measuring many things in your blood during your visits, and it is possible we might uncover a medical problem that requires treatment. You will <u>not</u> be routinely provided treatment for any health condition discovered. However, you will be informed about such findings (e.g., high blood pressure) and any medically important information including blood tests or physical exam results will be forwarded to your primary care physician at your request. Some of these medical problems might prevent you from participating further in the study.

### **Risks and discomforts**

- 1. **Physical examination**. A physician or a nurse practitioner may need to examine you with your clothes off, with appropriate precautions to protect your privacy. Some may find this examination embarrassing.
- 2. **Radiation Exposure**: This research study involves exposure to radiation from three DEXA scans and three CT scans. Please note that this radiation exposure is not necessary for your medical care and is for research purposes only. The NIH Radiation Safety Committee has reviewed the use of radiation in this research study and has approved this use as involving minimal risk and necessary to obtain the research information desired.

Although each organ will receive a different dose, the amount of radiation exposure you will receive yearly from this study is equal to a uniform whole-body exposure of 0.093 rem. This calculated value is known as the "effective dose" and is used to relate the dose received by each organ to a single value. The amount of radiation you will receive in this study is below the dose guideline established by the NIH Radiation Safety Committee for research subjects. This guideline is an effective dose of 5 rem received per year.

For comparison, the average person in the United States receives a radiation exposure of 0.3 rem per year from natural background sources, such as from the sun, outer space, and from radioactive materials that are found naturally in the earth's air and soil. If you would like more information about radiation and examples of exposure levels form the other sources, please ask the investigator for a copy of the pamphlet called, <u>An Introduction to Radiation for NIH Research Subjects.</u>

3. **Blood withdrawal**. The blood withdrawal amount is well below the NIH guideline for a safe amount of blood withdrawal (550 cc every 8 weeks). A small bruise may form at any site where the blood is taken. The risk of infection or fainting is very small. Inflammation or clotting of a vein also may rarely occur.

Some of your blood will be sent to another laboratory within the NIH to examine your inflammation levels. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.

**MEDICAL RECORD** 

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

4. **Stool sample collection** has no risk, and should only take a moment to complete. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.

- 5. **Urine sample collection** has no risk and should only take a moment to complete. If you do test positive for an illicit substance, the result will be part of your NIH Medical Record.
- 6. **Questionnaires** are not risky, but may be inconvenient because of the time necessary to complete them.
- 7. **Oral glucose tolerance test.** This test is inconvenient because of the time it takes to complete. The only risks from this kind of study are those described for any blood draw, as well as developing nausea from the oral glucose. Patients may transiently develop high blood sugar levels from the glucose, but it should normalize within a few hours and should not be clinically significant.
- 8. **Intravenous glucose tolerance test.** This test is inconvenient because of the time it takes to complete. You can watch TV during this test. The only risks from these kinds of studies are those described for any blood draw, the possibility of slight arm tenderness in the arm receiving the sugar infusion, (this tenderness goes away within a few minutes with gentle rubbing of the arm), and the possibility of a low blood sugar during the study. With slightly low blood sugars (less than 50 mg/dL), participants may get hungry, have a headache, feel shaky or dizzy, may become drowsy, or may become sweaty. With very low blood sugars (under 30 mg/dL) participants may have trouble speaking, be difficult to arouse, and even have seizures. However, in the test we are doing, we will be giving you extra sugar to raise your blood sugar above normal, and then we will try to bring it back to normal (95-105 mg/dL) with insulin. To do this, we will measure blood sugar at 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, and 180 minutes (a total of 3 hours). A physician or nurse practitioner will be present during the first hour of your test to make sure everything is working properly. We expect that the chance of even a slightly low blood sugar is very low. If a low blood sugar does not come up on its own quickly, the test will be stopped and you will be given sugar by vein to raise the blood sugar to normal.
- 9. **Fat tissue biopsies.** Possible side effects of the biopsy procedure are pain during and for two to three days after the procedure, although rarely the biopsy site may be tender or sore or have bruising or swelling for 2-3 weeks. Biopsy wounds usually heal with a very small, nearly unnoticeable scar, but sometimes a raised scar (keloid) or visible lump may result. Your risk is slightly higher if you are African American. Lidocaine injection for numbing before fat biopsies may cause some mild burning before the numbing takes effect. Rare adverse effects include infection at the biopsy sites or an allergic reaction to Lidocaine that may lead to a rash and/or swelling of the injected area. If you know you are allergic to Lidocaine, we will change to another local anesthetic. Another risk of the procedure is minor bleeding in the area of the biopsy. Some medications may increase the amount of bleeding from the biopsy. If you are taking medications such as Coumadin, Plavix or aspirin to thin your blood, you WILL NOT have a biopsy. If you are taking aspirin or non-steroidal medications such as Advil for pain you will need to stop taking these medicines for one week before the biopsy is performed.
- 10. **Medication.** The most common adverse effects from the medication used in this study are nausea, vomiting, diarrhea, and abdominal pain. Some rare side effects (< 1%) have been reported including decreased production of red cells (which could make you feel tired), white blood cells (which can make more susceptible to infections), and/or platelets (which may make you more susceptible to bruising or bleeding), tingling (neuropathy), dizziness, muscle pain or weakness, rash, allergic reaction, decreased sperm count, and increased liver enzyme levels. These symptoms usually occur in people with underlying medical problems, or were on certain medications, that predisposed them to having the reaction. In general, these symptoms resolved within a week once the medication was stopped. Although colchicine has been used for about 2000 years for gout, as with any

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

medication, there is always the possibility of unpredicted side effects. We will monitor you for all adverse effects. If (severe) adverse effects develop, we will decrease the dose, temporarily stop, or discontinue the medication.

If you experience any of the following, contact our team right away:

- Muscle weakness or pain
- Numbness or tingling in the fingers or toes
- Unusual bleeding or bruising
- Severe diarrhea or vomiting

There are no adequate well-controlled studies on the use of colchicine in pregnancy. Data from a limited number of published studies found no evidence of an increased risk of miscarriage, stillbirth, or teratogenic effects among pregnant women using colchicine. However, colchicine did demonstrate birth defects in the offspring of pregnant rats. If you think you might become pregnant, we will ask that you not participate in this study.

- Taking certain medicines with colchicine can cause your level of colchicine to be too high, especially if you have kidney or liver problems (refer to "Medication Guide" for more information).
- Even medicines that you take for a short period of time, such as antibiotics, can interact with colchicine and cause serious side effects or death. Please tell us about any new medicine you need to take so we can make sure you can continue using colchicine.
- Avoid drinking grapefruit juice, as it can interfere with your body's ability to breakdown colchicine.

### Keep the medication out of the reach of children.

- 11. **DNA testing.** If you allow us to study your DNA, we will use it for genome sequencing. Genome sequencing is a test that could give us different kinds of results. These include:
  - a. We could identify changes in genes that are related to metabolism and body weight.
  - b. We could identify changes in genes that contribute to other diseases or problems.
  - c. We could identify changes in genes that are not known to cause any disease. These are known as normal variations.
  - d. We could find changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

Not all gene changes will have health implications for your family. Changes in genes that have health implications for your family:

- 1. May have already caused health problems.
- 2. May cause a health problem in the future.

One of the goals of this study is to identify changes in genes that may be involved in obesity. This research may take years. If however we identify a genetic cause or likely cause of obesity, with your permission, we will contact you. Please let us know your preference by initialing one of these two statements:

| about any results related to obesity | I would like to be contacted with information about the progress of this study and contacted about any results related to obesity. I understand that this research will take years and that a specific abnormality might not be identified in me. |
|---|---|
| | Please do not contact me regarding the progress of this study or any specific gene changes related to obesity. |

### MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Cli

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

If we detect a genetic change that might be important for you, then we will have to confirm this result in a certified laboratory. For this confirmation, we will ask for a new sample of DNA from you. In most cases this will involve obtaining a small sample of blood (1-2 teaspoons). In some cases we can obtain enough DNA to confirm a genetic change by swabbing the inside of the cheek. You can decide whether you want to do that later, if we contact you with the information that we have found a possible important genetic difference.

Identifying gene changes that are not related to the condition being studied is known as <u>incidental medical</u> information.

We will find gene changes in everyone that we study, but we are only specifically looking for genes related to metabolism and body weight. We will not analyze your DNA for changes that are not related to metabolism and body weight. Even so, some gene changes not related to metabolism and body weight will be detected.

We will only inform you only of changes that have urgent medical significance and would benefit from early medical treatment. An example of this would be a gene change that causes cancer and where you would benefit from early screening. We will not inform you of all gene changes that have uncertain health implications. For example we will not report gene changes that only predispose individuals to disease. An example of this would be a gene change that influences the risk of heart disease, but where the development of the disease is dependent on many genetic and non-genetic (such as diet and smoking) factors. If we find a change in a gene that is important to your family's health, we will only be able to give you those results if the change has been confirmed in a certified laboratory. To make sure an error has not occurred, we would need to obtain a new sample of DNA from you to confirm the experimental results.

In addition to knowing what we could find, we would like you to know the limitations of the genome sequencing and what we will NOT be able to tell you about the changes that we find.

- **1.** Not all gene changes that cause disease will be detected.
- **2.** Some changes that are not currently known to cause health problems will be found to cause health problems in the future. We cannot promise to be able to tell you about those changes in the future.
- **3.** We will not tell you about gene changes that are not known to have health implications, nor will we tell you about gene changes that have only reproductive consequences.
- **4.** This gene sequencing cannot be substituted for diagnostic testing recommended by another physician.

Please initial all of the following statements to indicate that you understand the extent to which we will inform you about incidental genetic changes that we find:

| I understand that I will be informed only of genetic changes that researchers involved in this study feel are urgently important for my family's health and that knowledge of these changes has the potential to provide a significant benefit for me or my family. |
|---|
| I understand that investigators will not specifically look for gene changes not related to metabolism and body weight, and that identification of other disease-causing genes will only occur by chance depending on the analysis being done. |
| I fully understand that even though they could have health or reproductive consequences, I will not be told about all genetic changes identified that are not related to metabolism and body weight. |

### **CONTINUATION SHEET for either:** MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

CONTINUATION:  pages STUDY NUMBER: 14-CH-0119

If we detect a gene change not related to metabolism and body weight and the investigators feel it meets the requirements of having urgent medical significance so that you would benefit from medical treatment, then you will be given a choice to learn or not learn about a genetic change that we find. You can chose not to be contacted at all if that is your preference. An exception to your ability to choose whether or not to find out about a gene change would be a gene change that investigators feel is of critical importance to your health. An example of this would be a gene change that has a high probability of causing cancer or a disease for which early treatment would be beneficial. Before confirming the result in a clinical laboratory we will contact you to obtain a new sample of DNA.

If you have a gene change with urgent health implications, the NIH will confirm the genetic change present in one member of your family. We will discuss the results with you so that you understand who else in your family could be a carrier for this same change. We can help arrange for this testing to be done, but the NIH cannot promise to perform or pay for the clinical testing necessary to confirm or determine who else in your family may have this change in their DNA.

Once a gene change is confirmed, we will discuss the results with you and make recommendations regarding appropriate medical follow up. The NIH cannot promise to perform or pay for recommended medical tests or evaluations.

It is possible that a gene change will not be confirmed on subsequent testing. This could be due to an error in the DNA sequencing or an error in processing the DNA or cell lines. Although you likely will be glad that we did not confirm a problem, this may cause some anxiety and concern that you otherwise would not have experienced.

Please let us know your preferences by initialing one of the following statements:

| <br>_ I DO want to be re-contacted if genetic variants with urgent health implications are discovered during this research testing. |
|---|
| I DO NOT want to be re-contacted if genetic variants with urgent health implications are discovered during this research testing. I understand that an exception to this choice, as described above, will be made for a gene change of critical medical significance. |

**Emotional and psychological risks from DNA testing.** Identification of gene changes could cause emotional and psychological problems. In some situations psychological counseling could be recommended.

- 1. Learning about disease risk in your family can be distressing.
- 2. Learning that you passed on a gene that does not work to your child can be distressing.
- 3. Other members of your family could be upset to learn that they may be at risk for a disorder because of your participation in this study.

You may be falsely reassured about your health status if we do not report any changes to you.

Other risks of genetic testing. If we confirm a gene change in your DNA in a diagnostic laboratory, this information will become part of your medical record at the NIH. Some people are concerned that information about them from their medical records could be released. Possible problems include insurance or employment discrimination. Measures to protect the confidentiality of your information are described below. These problems may also occur if you disclose information yourself or agree to have your research records released.

P.A.: 09-25-0099

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

There are state and federal laws that protect against genetic discrimination. A federal law called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. According to this law, health insurance companies or group health plans (as of May 21, 2010) cannot request your genetic information or use it to make decisions about your eligibility or premiums; and employers cannot use it in deciding to hire, promote, or fire you or in setting the terms of your employment (as of Nov 21, 2009).

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

The following link contains details on this policy: <a href="http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf">http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf</a>

Please initial one of the following three statements regarding future research:

You may ask your research team for additional information or a copy of The Genetic Information Nondiscrimination Act of 2008 informational document.

Genetic studies can uncover unexpected family relationships. For example, it is possible that we might learn that a family member is not the biological child of the parents with whom she or he lives (for example, because of adoption). We will not ordinarily provide this type of information to any member of the family or to the referring physician. However, we may make exceptions under extraordinary circumstances if this information were required for the medical care of the individuals involved. If we are convinced this is necessary, we will provide the information to the physician providing medical care to the patient.

### Use of stored samples and data

**Future DNA Research.** Currently we plan to sequence known genes. This represents only about 1% of your DNA sequence. In the future we may sequence other parts of your DNA, and eventually, we may completely sequence your DNA. These additional studies may occur years from now. Some of your DNA may be sent to other laboratories for specific tests. If this is done DNA will be coded and not have your name on the sample or the paperwork that goes to the laboratory. Should you withdraw from this study, we will keep your DNA for analysis unless you ask us to destroy the DNA samples.

DNA can be used for other kinds of future health-related research. This research is not limited to studies related to obesity, metabolism and body weight. This testing may be done by research laboratories that are not at the NIH. I authorize use of these samples without my additional consent. I understand I will not be contacted if these samples are used in the future.

I understand that genetic samples collected during these NIH visits will be saved and used for future experimental testing related to obesity, metabolism, and body weight. This testing may be done by research laboratories that are not at the NIH. I do NOT authorize use of these samples for any other purpose without my additional consent. I must be contacted and give consent if these samples are to be

\_ Do not use my DNA for any future studies beyond those described above in this consent form.

used in the future.

### CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

**Future research with blood samples.** Our specific research plans have been summarized in this consent form. In the course of the research, we will obtain blood samples. While we can do some of our tests immediately, we may want to store your blood samples in the freezer for future studies. In addition, certain information will be stored in your medical record. In the future, it is possible that your blood samples or medical records will be used for other research purposes that are not specifically outlined in this consent form. If this is done, samples will be coded, and you will not be identified by name. These samples may be stored at a separate site (called a repository) that specializes in storing clinical samples. You have the option, in the future, of requesting that these samples not be used for any additional testing. In addition, it is possible that some information obtained from these studies will be published in the medical literature. However, your identity will not be included in any publications.

publications.
 Please initial one of the following two statements:
 I understand that samples collected during these NIH visits will be saved and used for future experimental testing related to body weight, and/or metabolism. This testing may be done by research laboratories that are not at the NIH. I authorize other uses of these samples without my additional consent. I understand I will not be contacted if these samples are used in the future.
 I understand that samples collected during these NIH visits will be saved and used for future experimental testing related to body weight, and/or metabolism. This testing may be done by research laboratories that are not at the NIH. I do NOT authorize any other use of these samples without my additional consent. I must be contacted and give consent if these samples are to be used in the future.

All through the process of the study and afterwards, the confidentiality of participants will be protected by using codes and medical record numbers in recording your information and test results. Only medical personnel involved in this study will have access to participants' names, test results, and patient code numbers.

You need to be aware that DNA sequence is like a fingerprint. Theoretically if enough DNA sequence information is available, someone could identify you based on his/her DNA sequence. To facilitate genetic research, your DNA sequence information may be deposited in other databases. In this case, unless we have your permission, we will deposit the data in a manner that would not allow someone to identify you. Please understand that this information cannot be removed once it is deposited.

| Please | initial one of the following boxes. |
|---|---|
| | _ I do not want DNA sequence data to be deposited in any database other than the one associated with this study. |
| | _ My DNA sequence data can be deposited in databases that limit access to IRB (ethics board) approved researchers. |
| | _ My DNA sequence can be deposited in a database that is available only to scientists but that does not<br>require IRB approval of research studies. I understand that someone could theoretically identify me fron<br>this information. |

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

CONTINUATION:  pages STUDY NUMBER: 14-CH-0119

### Potential benefits of participation

We are hopeful that your participation in this study will provide evidence as to whether colchicine will help metabolic parameters in obese individuals. However, you might not benefit directly from participating in this study. Should we find abnormalities in any of your test results, you will be notified and receive a copy to assist you in seeking further medical evaluation. This information may or may not improve your health.

### Right of Withdrawal and Conditions for Early Withdrawal

You may withdraw from the study at any time and for any reason without loss of benefits or privileges to which you are otherwise entitled.

### **Discussion of New Findings with You**

After all participants have completed the study, we will inform you about which medicine you took and, once the study is fully analyzed, let you know if colchicine seemed to help with inflammation and insulin resistance. There is no general plan to share your individual test results with you. However, if any findings suggest you have a medical issue, we will provide this information to you and your primary care provider. You may request a copy of your routine laboratory tests if vou desire.

### **Study Termination**

You may be asked to end your participation in this study at any time if we believe that continuation is not in your best medical interest or if you are unable to comply with the requirements of the study.

### **Alternatives to Participation**

The alternative to this study is not to participate. You may be eligible for other studies in the NIH. You may learn more about them through www.clinicaltrials.gov.

### Compensation

You will be compensated for the time and inconvenience associated with participation according to NIH research volunteer guidelines. Compensation for completing all of the testing described above is \$100 for the outpatient screening visit, \$50 for the safety visit, and \$300 each for the baseline, final, and washout visits. The total amount you could receive for participation if you complete all parts of this study is \$1050.

### **Conflict of Interest**

The NIH and members of this research team have no financial interest related to this research study.

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

### Posting of Research Results on www.ClinicalTrials.gov

| A description of this clinical trial will be available on http://www.Clinicaltrials.gov, as required by U.S. Law. This web | site |
|---|---|
| will not include information that can identify you. At most the Web site will include a summary of the results. You car | 1 |
| search this Web site at any time. | |

\_\_\_\_\_ I have received a copy of the signed consent form.

### **MEDICAL RECORD**

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

Adult Patient or Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

### OTHER PERTINENT INFORMATION

**1. Confidentiality.** When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- **2. Policy Regarding Research-Related Injuries.** The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH quidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Jack A. Yanovski, MD, PhD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686 or Associate Investigator Andrew Demidowich, MD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686.

You may also call the Clinical Center Patient Representative at 301-496-2626.

**5. Consent Document.** Please keep a copy of this document in case you want to read it again.

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | |
|---|---|---|
| A. Adult Patient's Consent I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby consent to take part in this study. | | |
| Signature of Adult Patient/Legal Representative Date | Signature of Parent(s)/Guardian | Date |
| Print Name | Print Name | |
| C. Child's Verbal Assent (If Applicable) | | |
| The information in the above consent was described to my child and my child agrees to participate in the study. | | |
| Signature of Parent(s)/Guardian Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM JANUARY 24, 2018 THROUGH FEBRUARY 24, 2019. | | |
| Signature of Investigator Date | Signature of Witness | Date |
| Print Name | Print Name | |

### **PATIENT IDENTIFICATION**

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

NIH-2514-1 (07-09 P.A.: 09-25-0099

File in Section 4: Protocol Consent

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD ● Adult Patient or ● Parent, for Minor Patient

INSTITUTE: Instituto Nacional de Salud Infantil y Desarrollo Humano (National Institute of Child Health and

Human Development)

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Estudio preliminario de los efectos de la colchicina en adultos no diabéticos con síndrome

metabólico

(Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome)

Date Posted to Web: 08/03/18

Continuing Review Approved by the IRB on 01/24/18 Amendment Approved by the IRB on 07/13/18 (S)

Standard Spanish

### **INTRODUCCIÓN**

Deseamos invitarle a participar en un estudio de investigación en los Institutos Nacionales de Salud (*National Institutes of Health, NIH*).

En primer lugar, queremos que Ud. sepa que:

La participación en una investigación del NIH es totalmente voluntaria.

Usted puede decidir no participar o retirarse del estudio en cualquier momento. En cualquier caso, no perderá ninguna compensación a la que pueda tener derecho. No obstante, para recibir atención médica en el NIH usted debe participar en un estudio o estar en evaluación para participar en uno.

Es posible que no reciba ningún beneficio por su participación. Con la investigación podemos adquirir conocimientos que ayuden a otras personas en el futuro.

En segundo lugar, algunas personas pueden tener creencias personales, religiosas o éticas que limiten los tipos de tratamientos médicos o de investigación que deseen recibir (por ejemplo, transfusiones de sangre). Si usted es una de esas personas, hable al respecto con sus médicos o con el equipo de investigación del NIH antes de acceder a participar en el estudio.

El estudio se describe en las siguientes páginas. Antes de decidir participar, tómese todo el tiempo que necesite para hacer preguntas y hablar del estudio con cualquier persona del NIH, o con su familia, amigos, médico personal o cualquier otro profesional de la salud.

### Propósito de este Estudio

Aproximadamente 30% de los adultos en los EE.UU. tienen un índice de masa corporal (IMC) superior a 30 (kg/m2), y están en mayor riesgo de una serie de problemas médicos, incluyendo la presión arterial alta, colesterol alto en la sangre, niveles altos de triglicéridos, azúcar en la sangre (diabetes) y enfermedades del corazón. Se cree que tener sobrepeso, puede llevar a un estado de inflamación aunque de nivel bajo, y que esta inflamación puede conducir a algunos de los problemas médicos asociados con la obesidad. El propósito de este estudio es investigar si un medicamento llamado colchicine puede mejorar el metabolismo de los adultos que tienen complicaciones médicas debido a su sobrepeso corporal (estas complicaciones son algunas veces llamadas, "síndrome metabólico"), pero que aún no han desarrollado altos niveles de azúcar en la sangre (diabetes).

### **PATIENT IDENTIFICATION**

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (2)

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: CONTINUATION:  pages 14-CH-0119

Colchicine es una medicación anti- inflamatoria que se ha utilizado durante siglos en el tratamiento de la gota. A partir de estudios en animales y estudios en humanos, existe alguna evidencia de que los medicamentos anti-inflamatorios como colchicine pueden mejorar la capacidad del páncreas para secretar insulina y la capacidad del cuerpo para regular el azúcar. Les pedimos que se unan a nuestro estudio, por el cual esperamos averiguar si colchicine puede mejorar la regulación del azúcar y los parámetros metabólicos.

Si califica y está de acuerdo en participar, Ud. será una de 40 personas asignadas al azar para tomar ya sea cápsulas de colchicine o cápsulas de placebo por vía oral, dos veces al día durante 3 meses. Las cápsulas de colchicine vendrán en la misma dosis que está disponible en las farmacias y se prescribe para una enfermedad llamada "gota": 0.6 miligramos. Las cápsulas de placebo se parecen a las cápsulas colchicine, pero no contienen colchicine. Usted tendrá un 50% de probabilidad de ser asignado a tomar colchicine.

Este estudio está diseñado para ser "doble ciego": ni los médicos ni los participantes del estudio sabrán quién está tomando las cápsulas de colchicine y quién está tomando placebo. Sólo la farmacia del NIH sabrá si un participante en el estudio está recibiendo colchicine o placebo. A menos que sea necesario por razones médicas, ni los participantes ni los médicos serán informados de quién esta tomando lo uno o lo otro, hasta que se complete el estudio (hasta cuando todos los participantes terminen de tomar las capsulas). El propósito del estudio "doble ciego" es asegurarse de que no va a existir prejudicio hacia ninguna de las personas involucradas en el estudio. Cuando se haya completado el estudio, le enviaremos cada uno de los participantes información sobre los resultados y les daremos a conocer si estaban tomando colchicine o cápsulas de placebo.

Los participantes del estudio tendrán que venir al Centro Clínico del NIH para cuatro consultas ambulatorias, con una quinta consulta ambulatoria opcional. Es importante que los participantes llegen en ayunas (sin alimentos ni bebidas aparte de aqua) a cada una de estas visitas. Los participantes serán compensados por su tiempo y cualquier inconveniente (ver más abajo: Compensación en la página 5).

### Población de estudio

Deseamos reclutar a 40 adultos con sobrepeso.

### Quién puede participar en este estudio

Usted puede ser elegible para este estudio de investigación si es mayor de 18 años de edad; si tiene un índice de masa corporal mínimo de 30, el cual se calcula dividiendo el peso del individuo en kilogramos, por su altura en metros, al cuadrado, (Kg/m2); pesar menos de 450 libras, y que se encuentre en buen estado de salud general. Usted también tiene que cumplir con ciertos niveles de resistencia a la insulina y a la inflamación, medidas por pruebas de laboratorio, para participar en todo el estudio. Si usted es una mujer en edad de procrear, se le pedirá que use un método efectivo de control de la natalidad antes de participar en este studio.

### Quienes no pueden participar en este estudio

Usted no puede ser elegible para este estudio si tiene una enfermedad médica grave que pudiera interferir con las pruebas o mediciones del estudio, como enfermedades del corazón, riñón, hígado, pulmón, sangre, intestinal o enfermedades endocrinas o presión arterial alta no controlada. Si usted está usando un medicamento que afecta el metabolismo del azúcar y la grasa o la absorción en su cuerpo, o un medicamento que no se debe tomar con colchicine, es posible que no sea elegible para participar. Tampoco son elegibles las mujeres que están embarazadas o lactando, o tienen intención de quedar embarazadas; las personas que han tenido un cambio de peso reciente superior al

NIH-2514-1 (10-84) NIH-2514-2 (10-84)

P.A.: 09-25-0099

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

3% del peso corporal total, han estado utilizando medicamentos para reducir el peso, han usado recientemente la colchicina, tener una alergia conocida a la colchicina, o utilizan productos de tabaco o nicotina (p. ej. e-cigarrillos), no serán reclutadas para este estudio. Se recomienda a las personas con antecedentes de formación de queloides (que fácilmente desarrollan cicatrices en su piel después de una lesión) no participar en este estudio.

### Procedimientos del estudio

PATIENT IDENTIFICATION

El estudio consta de cuatro visitas ambulatorias en el Centro Clínico: **una visita para determinar elegibilidad, una visita inicial** para estudiar su metabolismo antes de la participación, **una corta visita ambulatoria** para comprobar cómo se siente el participante durante el estudio, y **una visita final** 3 meses después de la visita inicial para ver los cambios después de la participación. Al término de la visita final, usted tiene la opción de volver 3 meses después para otra visita en la cual se quiere ver si los cambios observados mientras la participacion en el estudiopermanecen incluso después de suspender la medicación del estudio. Se le asignará al azar para recibir la colchicina o placebo el día de completar la visita inicial.

### Visita Ambulatoria de Selección de Pacientes

Esta visita tomará unas 3 horas para realizarse. Usted será visto en un día de semana en el Centro Clínico del NIH. Le pedimos permanecer en ayunas durante las 10 horas anteriores a su llegada a la clínica y no debe comer o beber nada, excepto agua por la mañana. Durante esta visita, vamos a realizar lo siguiente:

- 1. **Protocolo y firma del formulario de consentimiento**. Vamos a repasar el estudio en detalle y a responder cualquier pregunta. El formulario de consentimiento debe ser firmado antes de poder tomar parte en el estudio.
- 2. **Historia médica completa y un examen físico**, con el peso, la altura, y la medición de la presión arterial.
- 3. Un **ECG** se realizará para examinar la función de su corazón.
- 4. Los análisis de sangre en ayunas para asegurarse de que usted se encuentra en buen estado de salud. El análisis examinará el recuento de células de la sangre, función hepática y renal, niveles de colesterol, los niveles de azúcar e insulina en sangre, pruebas de función tiroidea, nivel de la inflamación, así como muestras de sangre de reserva para ser preservadas para poder examinar durante futuras investigaciónes. También realizaremos pruebas para determinar si usted tiene alguna diferencia en genes que pueden ser importantes para el metabolismo y el peso corporal. Además para buscar algunos genes que ya nosotros pensamos que son importantes para el peso corporal, vamos a utilizar nueva tecnología de secuenciación de DNA que se verá en todos los genes humanos que conocemos. Esto se conoce como "exome" y secuenciación del genoma. Esta nueva tecnología nos permite mirar el ADN en gran detalle.
- 5. **Recogida de muestras de orina** para asegurarse de que sus riñones funcionan normalmente, que no está tomando cualquier droga ilícita, y una prueba de embarazo (para las mujeres en edad fértil).
- 6. **Prueba de tolerancia a la glucosa oral**. Vamos a realizar una prueba para examinar si usted tiene diabetes, la llamamos prueba de tolerancia a la glucosa de 2 horas. Va a tomar una taza de agua con azúcar y luego se tomarán muestras 1 y 2 horas después para mirar su nivel de azúcar en la sangre.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

7. **Absorciometría dual de rayos X (DEXA)** para examinar su composición corporal. La prueba consiste en permanecer inmóvil sobre una mesa mientras una pequeña cámara pasa sobre su cuerpo. La dosis de los rayos X es mucho menor que la cantidad que se obtiene de una radiografía de pecho normal. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos.

### Visita Inicial

PATIENT IDENTIFICATION

Si reúne los requisitos para participar en el estudio, se le cita para la visita inicial. Le pediremos que permanezca en ayunas durante 10 horas antes de llegar a la clínica y no comer o beber nada, excepto agua por la mañana. Usted será visto en un dia entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita tomará alrededor de 8 horas para completarse. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo de historia clínica **y examen físico**, con el peso, la altura, y la medición de la presión arterial. También se completará un cuestionario.
- 2. **Los análisis de sangre en ayunas** para mirar su metabolismo basal y los niveles inflamatorios, así como muestras de sangre de reserva para ser preservados para las pruebas de investigación adicionales posibles, incluyendo una muestra para futuro análisis genético. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener las muestras de sangre.
- 3. Obtención **de muestras de heces**, obtendremos dos muestras de heces para conservar para futuros experimentos. Como parte de esta colección, le pediremos que mantenga un record de su dieta por 24 horas en un formulario que se le entregara a usted, y asi ver como la dieta puede afectar los resultados de las pruebas de heces. Los resultados de este "diario de nutricion" irá con un nutricionista.
- 4. Obtención **de muestras de orina** como se describe antes. También vamos a recoger la orina durante su visita a ahorrar para futuros experimentos.
- 5. **Prueba de tolerancia a la glucosa intravenosa muestreado frecuentes**. Este estudio nos dice mucho acerca de cómo su cuerpo utiliza el azúcar, qué tan bien está funcionando su insulina y cómo es la sensibilidad de su cuerpo a la insulina. El estudio FSIVGTT se hace mientras usted descansa en una cama. Una segunda línea IV se coloca en su brazo. Le daremos un poco de agua de azúcar en una vía intravenosa durante un período de 2 minutos. Entonces vamos a tomar muestras de sangre de la otra IV en -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, y 180 minutos (un total de 3 horas ) para medir los niveles de azúcar e insulina . Exactamente a los 20 minutos en la prueba, le daremos una pequeña cantidad de insulina a través de la IV. Un médico o enfermera practicante estará presente durante la primera hora del estudio. Usted puede ver la televisión durante esta prueba.
- 6. Tomografía Computarizada (TC) del abdomen para observar donde se tiende a almacenar su grasa. La prueba consiste en permanecer quieto en una mesa móvil que pasa por un gran anillo donde esta ubicada la cámara. La prueba implica radiación, pero solo porque tomaremos una foto de su abdomen, el método que se utilizará minimiza su exposición. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos
- 7. Subcutánea Biopsia de grasa. Para examinar el nivel de ciertas moléculas en el tejido graso, se tomará una

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

pequeña muestra de tejido graso de debajo de la piel de su abdomen a través de una técnica de "miniliposucción". Para adormecer el área donde se tomarà la muestra, se utilizará la lidocaína, un anestésico local. Una aguja se utilizará para extraer una porción de tejido graso que mide alrededor de 1 ½ cucharaditas. Un vendaje se aplica entonces al sitio de inserción de la aguja. Podemos darle algún medicamento para el leve dolor, como Tylenol o medicamento más fuerte si es necesario, después de la biopsia. La biopsia se tomará de un lugar del cuerpo que normalmente está cubierto y que no se ve fácilmente.

8. **Los medicamentos de dispensación de Estudio**. Se le dará un suministro de aproximadamente 8 semanas de la medicación del estudio para ser tomado dos veces al día (mañana y tarde/noche) en casa. El medicamento se puede tomar con o sin alimentos. Le daremos una alarma de recordatorio para ayudarle a recordar cuándo tomar su medicamento. Si se olvida de tomar una dosis, tómela tan pronto como lo recuerde. Pero si está dentro de las 4 horas de la hora de su siguiente dosis, no tome una dosis doble. Sólo tome la dosis olvidada.

### Visita Ambulatoria Corta

Para asegurarse de que está tomando bien el medicamento, usted será visto en un día de la semana en el Centro Clínico de los Institutos Nacionales de Salud. Esta visita se tomara alrededor de 2 horas en completarse. Le pedimos que traiga su botella de píldoras con usted. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo de historia clínica **y examen físico**, con el peso, la altura, y la medición de la presión arterial.
- Análisis de sangre en ayunas, para asegurarse de que está en buen estado de salud, para examinar sus niveles de inflamación, así como muestras de sangre de reserva para ser preservado para las pruebas adicionales futuras.
- 3. **Recogida de muestras de orina** como se describe antes.
- 4. **Los medicamentos de dispensación de Estudio**. Le daremos otra botella de la medicación del estudio (para un periodo de cerca de 8 semanas) para que le dure hasta la visita final (3 meses). Al igual que antes, si olvida tomar una dosis, tómela tan pronto como lo recuerde. Pero si está dentro de las 4 horas de la hora de su siguiente dosis, no tome una dosis doble. Omita la dosis olvidada.

### Visita Final

PATIENT IDENTIFICATION

Le pediremos traer su botella con pastillas sobrantes de su anterior visita. Le pedimos permanecer en ayunas durante 10 horas antes de llegar a la clínica y <u>no comer o beber nada excepto agua por la mañana</u>. Usted será visto en un día entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita se llevará alrededor de 8 horas para completar. Durante esta visita vamos a realizar lo siguiente:

- 1. **Intervalo historia clínica y examen físico**, con el peso, la altura, y la medición de la presión arterial
- 2. **Análisis de sangre** en ayuno como se describe anteriormente. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener muestras de sangre.
- 3. **Recogida de muestras de heces** como se describe antes.
- 4. **Recogida de muestras de orina** tal como se describe antes.
- 5. Prueba muestreado frecuentes tolerancia a la glucosa intravenosa (FSIVGTT) como se describe antes.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

- 6. **DEXA Scan** como se describe antes.
- 7. **CT Scan** como se describe antes
- 8. Grasa subcutánea biopsia como se ha descrito antes
- 9. Cuestionario final para contarnos acerca de su experiencia de participar en nuestro protocolo.

### Visita Opcional

Debido a que nos gustaría ver si la colchicina seguirá teniendo efectos positivos duraderos en la regulación del metabolismo de su glucosa, la inflamación, y/o su salud cardiovascular, incluso después de haber dejado de tomarlo, invitamos a los pacientes a volver al Centro Clínico de los NIH 3 meses después de terminar la medicación del estudio para repetir las mismas pruebas.

Al igual que antes, le pedimos que permanecer en ayunas durante 10 horas antes de llegar a la clínica y <u>no comer o beber nada, excepto agua por la mañana</u>. Usted será visto en un día entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita llevará alrededor de 8 horas para completarse. Durante esta visita vamos a realizar lo siguiente:

- 1. **Intervalo historia clínica y examen físico**, con el peso, la altura, y la medición de la presión arterial
- 2. **Análisis de sangre e**l ayuno como se describe anteriormente. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener muestras de sangre.
- 3. Recogida de muestras de heces como se describe antes.
- 4. Recogida de muestras de orina tal como se describe antes.
- 5. **Prueba muestreado frecuente de tolerancia a la glucosa intravenosa (FSIVGTT)** como se describe antes.
- 6. **DEXA Scan** como se describe antes.
- 7. **CT Scan** como se describe antes.
- 8. Grasa subcutánea biopsia como se ha descrito antes

Cuando el estudio se haya completado, volverá al cuidado de su médico de cabecera. La participación en este estudio no compromete al NIH a su cuidado a largo plazo.

### Los resultados de pruebas realizadas en el NIH

Estaremos midiendo muchas cosas en su sangre durante sus visitas, y podríamos descubrir algún problema médico que requiere tratamiento. Ud. no recibirá de forma rutinaria tratamiento para cualquier condición de salud descubierto. Sin embargo, se le informará sobre estos hallazgos (por ejemplo: presión arterial alta) y cualquier información de importancia médica que resulten de análisis de sangre o del examen físico, serán remitidos a su médico de atención primaria en su solicitud. Algunos de estos problemas médicos podrían impedir su participación más en el estudio.

### Riesgos y molestias

PATIENT IDENTIFICATION

- 1. **El examen físico**. Un médico o una enfermera puede tener que le examinar pidiéndole que se quite su ropa, con las precauciones adecuadas para proteger su privacidad. Algunos pueden encontrar este examen vergonzoso.
- 2. Exposición a la radiación: Este estudio de investigación implica la exposición a la radiación de tres imagenes

**MEDICAL RECORD** 

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

DEXA y tres tomografías computarizadas. Tenga en cuenta que esta exposición a la radiación no es necesario para su atención médica y es sólo para fines de investigación. El Comité de Seguridad Radiológica NIH ha revisado el uso de la radiación en este estudio de investigación y ha aprobado este uso ya que implica un riesgo mínimo y necesario para obtener la información de investigación deseada.

Aunque cada órgano recibirá una dosis diferente, la cantidad de exposición a la radiación que recibirá anualmente de este estudio es igual a una exposición uniforme de todo el cuerpo a 0.093 rem. Este valor calculado se conoce como la "dosis efectiva" y se utiliza para relacionar la dosis recibida por cada órgano a un solo valor. La cantidad de radiación que recibirá en este estudio es inferior a la pauta de dosis establecido por el Comité de Seguridad Radiológica NIH para los sujetos de investigación. Esta pauta establece una dosis efectiva de 5 rem recibido por año.

Por comparación, la persona promedio en los Estados Unidos recibe una exposición a la radiación de 0,3 rem por año a partir de fuentes naturales, como el sol, el espacio exterior, y de materiales radiactivos que se encuentran naturalmente en el aire y el suelo. Si desea más información sobre la radiación y los ejemplos de los niveles y forma de exposicion a otras fuentes, por favor pregunte al investigador para obtener una copia del folleto titulado, <u>An Introduction to Radiation for NIH Research Subjects.</u>

3. **La extracción de sangre**. La cantidad de extracción de sangre es muy por debajo de la directriz del NIH para una cantidad segura de extracción de sangre (550 cc cada 8 semanas). Un pequeño moretón se puede formar en

cualquier sitio donde se toma la sangre. El riesgo de infección o desmayo es muy pequeña. La inflamación o coagulación de una vena también pueden ocurrir raramente.

Una parte de su sangre será enviado a otro laboratorio dentro del NIH para examinar sus niveles de inflamación. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras

- 4. **Recogida de muestras de heces** no tiene ningún riesgo, y sólo debe tomar un momento para recogerlas. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras.
- 5. **La recogida de muestras de orina** no tiene ningún riesgo y sólo toma un momento para completar. Si el resultado es positivo para una sustancia ilícita, el resultado será parte de su expediente médico NIH.
- 6. **Los cuestionarios no son peligrosos**, pero pueden ser un inconveniente debido al tiempo necesario para su realización.
- 7. **Prueba oral de tolerancia a la glucosa**. Esta prueba es un inconveniente debido al tiempo que se tarda en completar. Los únicos riesgos de este tipo de estudio son las descritos para cualquier extracción de sangre, así como el desarrollo de las náuseas por la glucosa oral. Algunos pacientes pueden desarrollar de forma transitoria niveles altos de azúcar en la sangre a partir de la glucosa, pero deben normalizarse a las pocas horas y no deben ser clínicamente significativos.
- 8. Prueba de tolerancia a la glucosa intravenosa. Esta prueba es un inconveniente debido al tiempo que se

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

tarda en completar. Usted puede ver la televisión durante esta prueba. Los únicos riesgos de este tipo de estudios son las descritas para cualquier extracción de sangre, la posibilidad de una ligera sensitividad en el brazo al recibir la infusión de azúcar, (esa sensitividad desaparece al cabo de unos minutos con el roce suave del brazo), y la posibilidad de un bajo nivel de azúcar en la sangre durante el estudio. Cuando la azúcar en sangre esta baja (menos de 50 mg/dl), los participantes pueden tener hambre, tener dolor de cabeza, sentirse temblorosos o mareados o pueden llegar a ponerse sudorosos. Con azúcar en la sangre muy bajos (menos de 30 mg/dl) participantes pueden tener problemas para hablar, dificultad para despertar, e incluso tener convulsiones.

Sin embargo, en la prueba que estamos haciendo, le estaremos dando azúcar extra para elevar el azúcar en la sangre por encima de lo normal, y luego vamos a tratar de traerlo de vuelta a la normalidad (95-105 mg / dL) con insulina. Para ello, vamos a medir el azúcar en la sangre a los 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, y 180 minutos (un total de 3 horas). Un médico o enfermera practicante estará presente durante la primera hora de su prueba para asegurarse de que todo funciona correctamente. Esperamos que la posibilidad de un nivel de azúcar en sangre bajo sea muy pequeña. Si un bajo nivel de azúcar en la sangre no sube por sí sola con rapidez, se detendrá la prueba y se le dará el azúcar por vía IV para elevar el azúcar en la sangre a la normalidad

- 9. Biopsias de grasa. Los posibles efectos secundarios de la biopsia son el dolor durante y durante dos o tres días después del procedimiento. Aunque rara vez, la zona de la biopsia puede estar sensible o adolorida o tener moretones o hinchazón durante 2-3 semanas. Heridas biopsia suelen sanar con una cicatriz muy pequeña, casi imperceptible, pero a veces una cicatriz elevada (queloides) o bulto visible puede resultar. Su riesgo es ligeramente mayor si usted es afroamericano. Inyección de lidocaína para adormecer antes de biopsias de grasa puede causar un poco de ardor suave antes de que llegue el entumecimiento. Efectos adversos raros incluyen la infección en los sitios de biopsia o una reacción alérgica a la lidocaína que puede llevar a una erupción y/o hinchazón de la zona de inyección. Si usted sabe que es alérgico a la lidocaína, cambiaremos a otro anestésico local. Otro de los riesgos del procedimiento es sangrado menor en el área de la biopsia. Algunos medicamentos pueden aumentar la cantidad de sangrado de la biopsia. Si está tomando medicamentos como Coumadin, Plavix o aspirina para adelgazar la sangre, usted no tendrá una biopsia. Si está tomando aspirina o medicamentos no esteroides como Advil para el dolor tendrá que dejar de tomar estos medicamentos durante una semana antes de realizar la biopsia.
- 10. **Medicamentos.** Los efectos adversos más comunes de los medicamentos utilizados en este estudio son: náuseas, vómitos, diarrea y dolor abdominal. Se han observado algunos efectos secundarios raros (<1%) son los siguientes: disminución de la producción de glóbulos rojos (que podría hacer que se sienta cansado), glóbulos blancos (que puede hacer más susceptibles a las infecciones), y/o plaquetas (que pueden hacerle más susceptibles a la aparición de moretones o sangrado), hormigueo (neuropatía), mareo, dolor muscular o debilidad, erupción, reacción alérgica, disminución del recuento de espermatozoides , y aumento de los niveles de enzimas hepáticas. Estos síntomas generalmente ocurren en personas con problemas médicos subyacentes, o estaban en ciertos medicamentos, que les predispone a tener la reacción. En general, estos síntomas se resolvieron dentro de una semana una vez que se suspende el medicamento. Aunque la colchicine se ha utilizado durante unos 2000 años para la gota, al igual que con cualquier medicamento, siempre existe la posibilidad de efectos secundarios imprevistos. Le supervisaremos por todos los efectos adversos. Si se desarrollan (severos) efectos adversos, vamos a disminuir la dosis, interrumpir temporalmente o suspender la medicación.

Si usted experimenta cualquiera de los siguientes efectos, póngase en contacto con nuestro equipo de inmediato:

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

- Debilidad muscular o dolor
- El entumecimiento u hormigueo en los dedos o dedos de los pies
- Sangrado o moretones inusuales
- La diarrea grave o vómitos

No hay estudios bien controlados adecuados sobre el uso de colchicine durante el embarazo. Los datos de un número limitado de estudios publicados no encontraron evidencia de un mayor riesgo de aborto involuntario, muerte, o efectos teratogénicos en las mujeres embarazadas que usan colchicina. Sin embargo, la colchicine mostró defectos de nacimiento en las crías de ratas embarazadas. Si usted cree que puede quedar embarazada, le pediremos que no participe en este estudio.

- Tomar ciertos medicamentos con colchicina puede hacer que subir demasiado su nivel de colchicina, especialmente si usted tiene problemas renales o hepáticos (consulte "Guía del Medicamento" para más información).
- Incluso los medicamentos que usted toma por un corto período de tiempo, tales como antibióticos, pueden interactuar con colchicina y causar efectos secundarios graves o la muerte. Por favor díganos acerca de cualquier medicamento que usted necesita tomar para que podamos asegurarnos de que puede seguir utilizando colchicina.
- Evite beber jugo de toronja, ya que puede interferir con la capacidad del cuerpo para desglosar colchicina

### Mantenga el medicamento fuera del alcance de los niños.

- 11. **Las pruebas de ADN.** Si nos permite estudiar su ADN, lo vamos a utilizar para la secuenciación del genoma. La secuenciación del genoma es una prueba que nos podrían dar diferentes tipos de resultados. Estos incluyen:
  - a. Podríamos identificar cambios en los genes que están relacionados con el metabolismo y el peso corporal.
  - b. Podríamos identificar cambios en los genes que contribuyen a otras enfermedades o problemas.
  - c. Podríamos identificar los cambios en los genes que no son conocidos por causar ninguna enfermedad. Estos son conocidos como variaciones normales.
  - d. Podríamos encontrar cambios en los genes que son nuevos y de importancia clínica incierta. Esto significa que no se sabe si podrían causar o contribuir a una enfermedad o si son variaciones normales.

No todos los cambios genéticos tendrán implicaciones para la salud de su familia. Los cambios en los genes que tienen implicaciones para la salud de su familia:

- 1. Ya han causado problemas de salud.
- 2. Pueden causar un problema de salud en el futuro.

Uno de los objetivos de este estudio es identificar los cambios en los genes que pueden estar implicados en la obesidad. Esta investigación puede tomar años. Sin embargo, si se identifica una causa genética o la causa probable de la obesidad , con su permiso, nos pondremos en contacto con usted. Por favor, háganos saber su preferencia con sus iniciales en una de estas dos declaraciones:

\_\_\_\_\_ Me gustaría ser contactado con la información sobre los avances de este estudio y contactado acerca de

### **MEDICAL RECORD**

### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

cualquier resultado relacionado con la obesidad. Entiendo que esta investigación llevará años y que una anormalidad específica no se puede identificar en mí.

Por favor no se contacte conmigo acerca de la marcha de este estudio o cualquier cambio de genes específicos relacionados con la obesidad.

Si detectamos un cambio genético que podría ser importante para usted, entonces vamos a tener que confirmar este resultado en un laboratorio certificado. Por esta confirmación, le pediremos una nueva muestra de ADN a usted. En la mayoría de los casos esto implicará la obtención de una pequeña muestra de sangre (1-2 cucharaditas). En algunos casos podemos obtener suficiente ADN para confirmar un cambio genético por limpiando el interior de la mejilla. Usted puede decidir, si desea hacerlo más adelante, si nos comunicamos con usted con la información de que hemos encontrado una posible diferencia genética importante.

La identificación de cambios genéticos que no están relacionados con la condición que se está estudiando, se conoce como información médica incidental.

Vamos a encontrar cambios genéticos en todo el mundo que estudiamos, pero estamos mirando sólo específicamente para los genes relacionados con el metabolismo y el peso corporal. No vamos a analizar su ADN para los cambios que no están relacionados con el metabolismo y el peso corporal. Aun así, algunos cambios en los genes no relacionados con el metabolismo y el peso corporal se detectarán.

Nosotros sólo le informaremos de los cambios que tienen importancia médica urgente y se beneficiarían de un tratamiento médico temprano. Un ejemplo de esto sería un cambio en el gen que causa cáncer y en la que se beneficiaría de la detección temprana. No le informará de todos los cambios en los genes que tienen inciertas implicaciones para la salud. Por ejemplo no vamos a informar de los cambios genéticos que predisponen a los individuos sólo a la enfermedad. Un ejemplo de esto sería un cambio en el gen que influye en el riesgo de enfermedades del corazón, pero en el que el desarrollo de la enfermedad depende de muchos factores genéticos y no genéticos (tales como la dieta y el tabaquismo). Si nos encontramos con un cambio en un gen que es importante para la salud de su familia, sólo le daremos los resultados si el cambio ha sido confirmado por un laboratorio certificado. Para asegurarse de que no se ha producido un error, tendríamos que obtener una nueva muestra de ADN a partir de que se confirmen los resultados experimentales.

Además de saber lo que encontramos, nos gustaría que conociera las limitaciones de la secuenciación del genoma y lo que no vamos a ser capaces de decirle acerca de los cambios que encontramos.

- 1. No todos los cambios en los genes que causan la enfermedad serán detectados.
- 2. Algunos de los cambios que no se conocen actualmente para causar problemas de salud podrían causar problemas de salud en el futuro. No podemos prometer tener la capacidad de decirle a usted acerca de esos cambios en el futuro.
- 3. No le dirá acerca de cambios en los genes que no se sabe que tienen consecuencias para la salud, ni vamos a informarle sobre cambios en los genes que sólo tienen consecuencias reproductivas.
- 4. Esta secuenciación de genes no puede ser sustituido por las pruebas de diagnóstico recomendado por otro médico.

### **CONTINUATION SHEET for either: MEDICAL RECORD**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: CONTINUATION:  pages 14-CH-0119

| • | sus iniciales en todas las siguientes declaraciones para indicar que usted entiende la medida en os sobre los cambios genéticos accidentales que encontremos: |
|---|---|
| Entiendo, que voy a estar informado sólo de cambios genéticos que los investigado<br>en este estudio piensen que son urgentemente importantes para la salud de mi far<br>conocimiento de estos cambios tiene el potencial de un beneficio significativo para<br>familia. | |
| | _ Entiendo que los investigadores no van a buscar específicamente cambios en los genes no relacionados con el metabolismo y el peso corporal, y que la identificación de otros genes que causan enfermedades sólo ocurrirá por casualidad dependiendo del análisis que se realiza. |
| | _ Entiendo perfectamente que a pesar de que podrían tener consecuencias de salud o reproductivas, no se me hablará de todos los cambios genéticos identificados que no están relacionados con el metabolismo y el peso corporal. |
| <b>6</b> | |

Si se detecta <u>un cambio en el gen no relacionado con el metabolismo y el peso corporal</u> y los investigadores sentimos que cumple con los requisitos de tener importancia médica urgente para que usted se beneficie de un tratamiento médico, a continuación, se le dará la opción para aprender o no aprender acerca del cambio genético encontrado. Usted puede elegir no ser contactado en absoluto si esa es su preferencia. Una excepción a su capacidad de elegir si desea o no saber acerca de un cambio en un gen, sería un cambio en un gen que los investigadores consideran que es de vital importancia para su salud. Un ejemplo de esto sería un cambio en el gen que tiene una alta probabilidad de causar cáncer o una enfermedad para la cual el tratamiento temprano sería beneficioso. Antes de confirmar el resultado en un laboratorio clínico nos pondremos en contacto con usted para obtener una nueva muestra de ADN.

Si usted tiene un cambio en un gen con urgentes implicaciones para la salud, el NIH confirmará el cambio genético presente en uno de los miembros de su familia. Discutiremos los resultados con usted para que pueda saber si alguien más en su familia podría ser un portador de este mismo cambio. Podemos ayudarle a organizar las pruebas que haya que hacer, pero el NIH no podemos prometer realizar o pagar por las pruebas clínicas necesarias para confirmar o determinar quién más en su familia puede tener este cambio en su ADN.

Una vez que se confirma un cambio en un gen, vamos a discutir los resultados con usted y hacer recomendaciones sobre apropiado sequimiento médico. El NIH no puede prometer realizar o pagar por los exámenes médicos recomendados o evaluaciones.

Es posible que un cambio genético no se confirmará en las pruebas posteriores. Esto podría ser debido a un error en la secuenciación de ADN o un error en el procesamiento del ADN o líneas celulares. Aunque es agradable para Ud. que no se confirme el problema, esto puede causar un poco de ansiedad y preocupación que de otra manera no habría experimentado.

| Por favor, háganos saber sus preferencias colocando sus iniciales en una de las siguientes afirmaciones: | |
|---|---|
| Yo QUIERO ser re-contactado si se descubren variantes genéticas con consecuencias urgente | 25 |

### CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-1, Consent to Participate in A Clinical Research Study
NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

para la salud, durante esta prueba de investigación.

NO deseo volver a ser contactado si se descubren variantes genéticas con consecuencias urgentes para la salud durante esta prueba de investigación. Entiendo que una excepción a esta elección, como se describió anteriormente, se hará para un cambio en el gen de importancia médica fundamental.

**Riesgos emocionales y psicológicos de la prueba de ADN**. La identificación de los cambios en los genes puede causar problemas emocionales y psicológicos. En algunas situaciones se podría recomendar asesoría psicológica.

- 1. Aprender sobre el riesgo de enfermedad que en su familia puede ser angustiante.
- 2. Aprender que algo que sucede en un gen suyo, puede no suceder en su hijo, puede ser angustiante.
- 3. Otros miembros de su familia podrían ponerse molestos al saber que ellos pueden estar en riesgo de un trastorno debido a su participación en este estudio.

Ud. Puede permanecer falsamente tranquilo acerca de su estado de salud si nosotros no le reportamos ningún cambio en su caso.

**Otros riesgos de las pruebas genéticas.** Si confirmamos un cambio genetico en su ADN en un laboratorio de diagnóstico, esta información será parte de su expediente médico en el NIH. Algunas personas se preocupan de que la información acerca de ellos de sus registros médicos podrían ser dadas a conocer. Posibles problemas incluyen el seguro o la discriminación laboral. Medidas para proteger la confidencialidad de su información se describen a continuación. Estos problemas también pueden ocurrir si usted divulga su propia información o acepta que sus registros de investigación sean liberados.

Hay leyes estatales y federales que protegen contra la discriminación genética. Una ley federal llamada la Ley de No Discriminación por información Genética (GINA), generalmente hace que sea ilegal que las compañías de seguros de salud, planes de salud de grupo, y la mayoría de los empleadores discriminen contra usted basado en su información genética. Según esta ley, las compañías de seguros de salud o planes de salud de grupo (hasta el 21 de mayo de 2010) no puede solicitar su información genética, o utilizarlo para tomar decisiones sobre su elegibilidad o primas; y los empleadores no pueden utilizarlo en la decisión de contratar, promover, ni puede despedirlo, o en el establecimiento de los términos de su empleo (a fecha de 21 de noviembre 2009).

Tenga en cuenta que esta ley federal no le protege contra la discriminación genética por las compañías que venden seguros de vida, seguro de invalidez, o un seguro de cuidado a largo plazo.

Este enlace contiene detalles sobre esta política:

PATIENT IDENTIFICATION

http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf

Usted puede preguntar a su equipo de investigación para obtener información adicional o una copia de la Ley de Discriminación por Información Genética de 2008 documento informativo.

Los estudios genéticos pueden descubrir relaciones familiares inesperados. Por ejemplo, es posible que podamos enteramos de que un miembro de la familia no es el hijo biológico de los padres con los que él o ella vive (por

### CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1. Consent to Participate in A Cli

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

ejemplo, debido a la adopción). No proporcionaremos normalmente este tipo de información a cualquier miembro de la familia o al médico de referencia. Sin embargo, podemos hacer excepciones en circunstancias extraordinarias si esta información se requiere para la atención médica de las personas involucradas. Si estamos convencidos de que esto es necesario, vamos a proporcionar la información al médico que proporciona la atención médica al paciente

### El uso de muestras almacenadas y datos

**Investigaciones futuras ADN**. Actualmente tenemos la intención de secuenciar los genes conocidos. Esto representa sólo alrededor del 1% de su secuencia de ADN. En el futuro podemos secuenciar otras partes de su ADN, y, finalmente, podemos secuenciar completamente su ADN. Estos estudios adicionales pueden ocurrir años a partir de ahora. Algunas partes de su ADN pueden ser enviadas a otros laboratorios para pruebas específicas. Si esto se hace el ADN será codificado y no tendrá su nombre en la muestra o en el papeleo que va al laboratorio. En caso de retirarse de este estudio, vamos a mantener su ADN para el análisis a menos que usted nos pida destruir las muestras de AND.

\_\_\_\_\_ ADN puede ser utilizado para otros tipos de futuras investigaciones relacionadas con la salud. Esta investigación no se limita a los estudios relacionados con la obesidad, el metabolismo y el peso corporal.

Por favor, coloque su inicial en una de las siguientes tres declaraciones relativas a la investigación futura:

Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. Autorizo el uso de estas muestras sin mi consentimiento adicional. Entiendo que no se pondrán en contacto si se utilizan estas muestras en el futuro.

Entiendo que las muestras genéticas recogidas durante estas visitas NIH serán guardados y utilizados para futuras pruebas experimentales relacionadas con la obesidad, el metabolismo y el peso corporal. Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. NO autorizo el uso de estas muestras para ningún otro fin sin mi consentimiento adicional. Debo ser contactado y dar consentimiento si estas muestras se van a utilizar en el futuro.

\_\_\_\_\_ No utilice mi ADN para futuros estudios más allá de los descritos anteriormente en este formulario de consentimiento.

**Futuras investigaciones con muestras de sangre**. Nuestros planes específicos de investigación se han resumido en este formulario de consentimiento. En el curso de la investigación, vamos a obtener muestras de sangre. Si bien podemos hacer algunas de nuestras pruebas de inmediato, es posible que desee almacenar sus muestras de sangre en el congelador para futuros estudios. Además, cierta información se almacenará en su expediente médico. En el futuro, es posible que sus muestras de sangre o registros médicos serán utilizados para otros fines de investigación que no se describen específicamente en este formulario de consentimiento. Si se hace esto, las muestras serán codificadas, y no serán identificados por su nombre. Estas muestras pueden ser almacenadas en un lugar separado (llamado un repositorio) que se especializa en el almacenamiento de muestras clínicas. Usted tiene la opción, en el futuro, de solicitar que estas muestras no se utilicen para hacer más ensayos. Además, es posible que alguna información obtenida de estos estudios serán publicados en la literatura médica. Sin embargo, su identidad no será incluida en cualquier publicación.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

| | Por favor, coloque su inicial en <u>una</u> de las dos afirmaciones siguientes: |
|---|---|
| | Entiendo que las muestras recogidas durante estas visitas NIH serán guardadas y utilizadas para futuros ensayos experimentales relacionados con el peso corporal, y/o el metabolismo. Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. Autorizo a otros usos de estas muestras sin mi consentimiento adicional. Entiendo que no se pondrán en contacto si se utilizan estas muestras en el futuro. |
| | Entiendo que las muestras recogidas durante estas visitas NIH serán guardadas y utilizadas para futuros ensayos experimentales relacionados con el peso corporal, y/o el metabolismo. Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. NO autorizo cualquier otro uso de estas muestras sin mi consentimiento adicional. Debo ser contactado y dar consentimiento si estas muestras se van a utilizar en el futuro. |
| | Durante todo el proceso de estudio y después, la confidencialidad de los participantes será protegida mediante e uso de códigos y números de historia clínica en la grabación de su información y resultados de pruebas. Sólo el personal médico involucrado en este estudio tendrán acceso a los nombres de los participantes, resultados de exámenes, y los números de código de los pacientes. |
| | Usted tiene que ser consciente de que la secuencia de ADN es como una huella digital. Teóricamente si suficiente información de la secuencia de ADN está disponible, alguien podría identificarlo a Ud. en base a su secuencia de ADN. Para facilitar la investigación genética, la información de su secuencia de ADN se puede depositar en otras bases de datos. En este caso, a menos que tengamos su permiso, vamos a depositar los datos de una manera que no permita que alguien le identifique. Por favor, comprenda que esta información no se puede eliminar una vez que se deposita. |
| Por fav | or, coloque su inicial en <u>una</u> de las siguientes casillas: |
| | <ul> <li>No quiero que los datos de secuencia de ADN sean depositados en cualquier base de datos que no sea la que está asociada con este estudio.</li> <li>Mis datos de secuencias de ADN pueden ser depositados en las bases de datos que limitan el acceso a la IRB (comité de ética) Investigadores aprobados.</li> <li>Mi secuencia de ADN puede ser depositada en una base de datos que está disponible sólo para los</li> </ul> |
| | científicos, pero que no requiere la aprobación del IRB de estudios de investigación. Entiendo que alguier |

### Los beneficios potenciales de la participación

Tenemos la esperanza de que su participación en este estudio proporcionará pruebas acerca de si la colchicina ayudará parámetros metabólicos en individuos obesos. Sin embargo, no puede beneficiarse directamente de participar en este estudio. Al encontrar anomalías en cualquiera de sus resultados de la prueba, se le notificará y recibirá una copia para ayudarle en la búsqueda de una mayor evaluación médica. Esta información puede o no mejorar su salud.

Derecho de revocación y Condiciones de retiro anticipado

teóricamente me podía identificar de esta información.

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Usted puede retirarse del estudio en cualquier momento y por cualquier motivo y sin pérdida de beneficios o privilegios a los que tiene derecho.

### La discusión de los nuevos hallazgos con usted

Después de que todos los participantes hayan completado el estudio, se le informará sobre cual medicina tomó y una vez que el estudio esté totalmente analizado, le permiten saber si la colchicina puede ayudar con la inflamación y la resistencia a la insulina. No hay plan general para compartir los resultados de sus pruebas individuales con usted. Sin embargo, si algún hallazgo sugiere que tiene un problema médico, vamos a proporcionar esta información a usted y a su proveedor de atención primaria. Usted puede solicitar una copia de sus pruebas de laboratorio de rutina si lo desea.

### **Terminación de Estudios**

Se le puede pedir terminar su participación en este estudio en cualquier momento, si creemos que la continuación en él no es lo mejor para su interés médico o si no puede cumplir con los requisitos del estudio.

### Alternativas a la Participación

La alternativa a este estudio es no participar. Usted puede ser elegible para otros estudios en los NIH. Usted puede aprender más sobre ellos a través de www.clinicaltrials.gov.

### **Compensación**

Usted será compensado por el tiempo y los inconvenientes asociados a la participación según las directrices de compensación para voluntarios de investigación del NIH. La compensación para completar todas las pruebas que se han descrito anteriormente es: \$100 por la visita de selección de pacientes ambulatorios, \$50 por la visita de seguridad, y de \$300 por cada una de las visitas inicial, final y la opcional. La cantidad total que usted podría recibir por la participación si completa todas las partes de este estudio es de \$1050.

### **Conflicto de intereses**

El NIH y los miembros de este equipo de investigación no tienen ningún interés financiero en relación con este estudio de investigación.

Publicación de Resultados de Investigación en: www.ClinicalTrials.gov

Una descripción de este ensayo clínico estará disponible en http://www.Clinicaltrials.gov, como lo requiere la ley de Estados Unidos. En esta pagina de web no incluirá información que pueda identificarlo. En la mayor parte del sitio Web incluirá un resumen de los resultados. Usted puede buscar en este sitio web en cualquier momento.

| incluira un resumen de los resultados. Usted puede buscar en este sitio web en cualquier momento. |
|---|
| He recibido una copia del formulario de consentimiento firmado. |

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

**MEDICAL RECORD** 

Adult Patient or Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

### INFORMACIÓN PERTINENTE ADICIONAL

**1. Confidencialidad**. Cuando los resultados de un estudio de investigación del NIH se dan a conocer en revistas médicas o reuniones científicas, no se menciona la identidad de los participantes. En la mayoría de los casos, el NIH no divulgará ninguna información sobre su participación en la investigación a menos que usted otorgue su permiso por escrito. No obstante, si usted firma una autorización de divulgación de información, por ejemplo, a una empresa aseguradora, el NIH le proporcionará a ésta información de su expediente médico. Esta información podría influir (en forma favorable o desfavorable para usted) la disposición de la aseguradora a venderle el seguro.

La Ley Federal de Protección de la Vida Privada (Federal Privacy Act) protege el carácter confidencial de sus expedientes médicos en el NIH. Sin embargo, es importante que sepa que esta ley permite la divulgación de cierta información de su expediente médico sin su autorización, por ejemplo, si lo solicitan la Administración de Alimentos y Medicamentos (FDA), los miembros del Congreso, los agentes encargados del cumplimiento de la ley o las organizaciones autorizadas para efectos de acreditación hospitalaria.

- **2. Normas sobre lesiones relacionadas con la investigación**. El Centro Clínico le dará atención médica a corto plazo para cualquier lesión que se deba a su participación en una investigación que se realice allí. En general, ni los Institutos Nacionales de Salud, ni el Centro Clínico, ni el gobierno federal le darán atención médica a largo plazo ni indemnización económica por lesiones relacionadas con la investigación. Sin embargo, usted tiene derecho a buscar una compensación legal si cree que la lesión justifica dicha medida.
- **3. Pagos**. El monto del pago que reciben los voluntarios de investigación se rige por las normas de los Institutos Nacionales de Salud. En general, a los pacientes no se les paga por participar en los estudios de investigación en los Institutos Nacionales de Salud. Se le ofrecerá el reembolso de gastos de viaje y viáticos según las pautas del NIH.
- **4. Problemas o preguntas**. Si hay algún problema o usted tiene una pregunta con respecto a este estudio, a sus derechos como participante en un estudio de investigación clínica o a cualquier lesión relacionada con la investigación, debe comunicarse con el Investigador Principal, Jack A. Yanovski, MD, PhD; Building (Edificio) 10, Room (Sala) 1-3330, Teléfono: (301) 496-4686 o el Investigador Asociado Principal, Andrew Demidowich, MD; Building 10, Room 1-3330, Teléfono: (301) 496-4686.

También puede llamar al representante de los pacientes del Centro Clínico, al teléfono (301) 496-2626.

**5. Documento de consentimiento.** Le sugerimos que conserve una copia de este documento para consultarla posteriormente.

**PATIENT IDENTIFICATION** 

**CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)** 

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

### **MEDICAL RECORD**

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

| COMPLETE LAS CASILLAS CORRESPONDIENTES A CONTINUACION: | |
|---|---|
| A. Consentimiento de un paciente adulto. | B. Permiso otorgado por el (los) padre(s) de un paciente |
| He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo mi consentimiento para participar en este estudio. | menor de edad. He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo permiso para que mi hijo participe en este estudio. (Anéxese el formulario NIH 2514-2, Asentimiento de un menor de edad, si corresponde.) |
| Firma del paciente adulto o su representante legal Fecha | Firma del (los) padre(s) o del tutor legal Fecha |
| Nombre en letra de imprenta | Nombre en letra de imprenta |
| C. Asentimiento verbal de un niño (si corresponde) Se le explicó a mi hijo la información contenida en el presente documento y mi hijo está de acuerdo en participar en el estudio. | |
| Se le explico a fili filjo la iliformación contenida en el presente documento y | 7 mi mjo esta de acuerdo en participar en el estudio. |
| Firma del (los) padre(s) o del tutor legal Fecha | Nombre en letra de imprenta |
| EL USO DE ESTE DOCUMENTO DE CONSENTIMIENTO ESTÁ APROBADO<br>DESDE EL 24 DE ENERO DE 2018 HASTA EL 24 DE FEBRERO DE 2019. | |
| Firma del Investigador Fecha | Firma del testigo Fecha |
| Nombre en letra de imprenta | Nombre en letra de imprenta |

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD

• Adult Patient or • Parent, for Minor Patient

INSTITUTE: National Institute of Child Health and Human Development

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome

Continuing Review Approved by the IRB on 01/24/18 Amendment Approved by the IRB on 07/13/18 (S)

**Evaluation-only** 

### INTRODUCTION

Date Posted to Web: 08/03/18

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

### **Purpose of this Study**

Fat cells play numerous important roles in our body including storing energy, secreting hormones, and helping regulate our metabolism. Insulin is a hormone that circulates throughout our body and communicates with our fat cells and regulates their function. When insulin's ability to communicate with the rest of the body begins to fail, people become "insulin resistant" and can go on to develop diabetes. However, the specific details of how insulin works at the level of the fat cell are still poorly understood. A purpose of this study is to better understand the timing and mechanisms behind insulin's actions on the fat cell, and possibly identify new factors of why some people are more prone to developing diabetes. We ask you to help us understand how insulin works in the body by undergoing a series of tests. You will not be asked to take the study medicine (colchicine).

### **PATIENT IDENTIFICATION**

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent (3)

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

You will need to come to the NIH Clinical Center for two outpatient visits. It is important that you arrive fasting (no food or beverages besides water) to each of these visits. You will be compensated for their time and inconvenience.

### **Study Population**

We wish to recruit healthy adults and adults with type 2 diabetes treated only with diet.

### **Who Can Be in This Study**

You may be eligible for this research study if you are greater than 18 years old, weigh less than 450 lbs, and are in good general health.

### Who May Not Be In This Study

You may not be eligible for this study if you have a major medical illness that would interfere with study tests or measurements, such as heart, kidney, liver, lung, blood, gut, or endocrine diseases, or uncontrolled high blood pressure. People with type 2 diabetes who are taking medication or have hemoglobin A1c >9%, are not allowed to participate. If you are currently using a medication that affects sugar and fat metabolism or absorption in your body, you may not be eligible to participate. Also individuals who are pregnant or nursing, or planning to become pregnant, have had a recent weight change greater than 3% of total body weight, have been using weight reducing medications, have recently used colchicine, have a known allergy to colchicine, or use tobacco or nicotine (e.g. e-cigarettes) products will not be recruited for this study. Individuals with a history of keloid formation (who easily develop scars on their skin after an injury) also will not be allowed to take part in this study.

### **Procedures of the study**

The study consists of two outpatient visits: an **outpatient screening visit** at the Clinical Center to determine eligibility and a **baseline visit** to study your metabolism.

### **Outpatient Screening Visit**

PATIENT IDENTIFICATION

This visit will take about 3 hours to complete. You will be seen on a weekday in the Clinical Center at the National Institutes of Health. We ask that you remain fasting for 10 hours before coming to the clinic and have nothing to eat or drink except water that morning. During this visit, we will perform the following:

- 1. **Protocol review and signing of consent form**. We will go over the study in detail, and answer any questions. The consent form will need to be signed before you can take part in the study.
- 2. **Complete medical history and physical exam,** with weight, height, and blood pressure measurement.
- 3. An **EKG** will be performed to examine your heart function.
- 4. Fasting blood tests to ensure that you are in good health. The analysis will examine blood cell count, liver and kidney function, cholesterol levels, blood sugar and insulin levels, thyroid tests, inflammation level, as well as reserve blood samples to be preserved for additional possible research tests. We will also plan to do tests to find out if you have any differences in genes that may be important for metabolism and body weight. In addition to looking at some genes we already think are important for body weight, we may use new DNA sequencing

P.A.: 09-25-0099

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

technology that will look at all the human genes we know about. This is known as exome and genome sequencing. This new technology allows us to look at DNA in great detail.

- 5. **Urine sample collection** to ensure that your kidneys work normally, that you are not taking any illicit drugs, and a pregnancy test (for women of childbearing age).
- 6. **Oral glucose tolerance test**. We will perform a test to examine whether you have diabetes, called a 2-hour glucose tolerance test. You will drink a cup of sugar water and then will have your blood drawn 1 and 2 hours later to look at your blood sugar level.
- 7. **Dual energy x-ray absorptiometry (DEXA)** to look at your body composition. The test involves lying still on a table while a small camera passes over your body. The dose of the x-ray is much less than the amount you would get from a normal chest x-ray. The total amount of time to do this test will be about 20-30 minutes.

### **Baseline Visit**

PATIENT IDENTIFICATION

If you qualify for participation in the study, you will be scheduled for the baseline visit. We ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink except water that morning</u>. You will be seen on a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement. A questionnaire will also be performed.
- 2. **Fasting blood tests** to look at your baseline metabolic and inflammatory levels, as well as reserve blood samples to be preserved for additional possible research tests including a sample for future genetic analysis. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection.** We will obtain two stool samples to save for future experiments. As part of this collection, we will ask you to keep track of your diet for 24 hours on a form that will be provided to you, as diet can affect the results of the stool testing. You will also go over this "food record" in person with a nutritionist.
- 4. **Urine sample collection** as described before. We will also collect urine over your eight hours of testing to save for future experiments.
- 5. **Frequently sampled intravenous glucose tolerance test (FSIVGTT)**. This study tells us a lot about how sugar is used by your body, how well your insulin works, and how sensitive your body is to insulin. The FSIVGTT study is done while you rest in bed. A second IV line will be placed in your arm. We will give you some sugar water into one IV over a 2 minute period. We will then draw blood samples from the other IV at -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes (a total of 3 hours) to measure sugar and insulin levels. Exactly 20 minutes into the test, we will give you a small amount of insulin through the IV. A physician or nurse practitioner will be present during the first hour of the study. You can watch TV during this test.
- 6. **Computed Tomography (CT) Scan** of the abdomen to look at where you tend to store your fat. The test involves lying still on a movable table which passes through a large ring where the camera sits. The test does

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

involve radiation, but because we only need to take a snapshot of your abdomen, the method that will be used minimizes your exposure. The total amount of time to do this test will be about 20-30 minutes.

7. **Subcutaneous Fat Biopsy**. To examine the level of certain molecules in your fat tissue, a small sample of fat tissue will be taken from under the skin of your abdomen. Lidocaine, a local anesthetic, is used to numb the area. A needle will be used to remove a piece of fat tissue measuring about 1 ½ teaspoons. A bandage is then applied to the site of needle insertion. We can give you some mild pain medication such as Tylenol, or stronger medication if needed, after the biopsy. The biopsy will be taken from a place on your body that is normally covered and not easily seen.

When the study is complete, you will return to the care of your regular physician. Participation in this study does not commit NIH to your long term care.

### **Results of Tests at the NIH**

We will be measuring many things in your blood during your visits, and it is possible we might uncover a medical problem that requires treatment. You will <u>not</u> be routinely provided treatment for any health condition discovered. However, you will be informed about such findings (e.g., high blood pressure) and any medically important information including blood tests or physical exam results will be forwarded to your primary care physician at your request. Some of these medical problems might prevent you from participating further in the study.

### **Risks and discomforts**

PATIENT IDENTIFICATION

- 1. **Physical examination**. A physician or a nurse practitioner may need to examine you with your clothes off, with appropriate precautions to protect your privacy. Some may find this examination embarrassing.
- 2. **Radiation Exposure**: This research study involves exposure to radiation from one DEXA scan and one CT scan. Please note that this radiation exposure is not necessary for your medical care and is for research purposes only. The NIH Radiation Safety Committee has reviewed the use of radiation in this research study and has approved this use as involving minimal risk and necessary to obtain the research information desired.

Although each organ will receive a different dose, the amount of radiation exposure you will receive yearly from this study is equal to a uniform whole-body exposure of 0.031 rem. This calculated value is known as the "effective dose" and is used to relate the dose received by each organ to a single value. The amount of radiation you will receive in this study is below the dose guideline established by the NIH Radiation Safety Committee for research subjects. This guideline is an effective dose of 5 rem received per year.

For comparison, the average person in the United States receives a radiation exposure of 0.3 rem per year from natural background sources, such as from the sun, outer space, and from radioactive materials that are found naturally in the earth's air and soil. If you would like more information about radiation and examples of exposure levels form the other sources, please ask the investigator for a copy of the pamphlet called, <u>An Introduction to Radiation for NIH Research Subjects.</u>

3. **Blood withdrawal**. The blood withdrawal amount is well below the NIH guideline for a safe amount of blood withdrawal (550 cc every 8 weeks). A small bruise may form at any site where the blood is taken. The risk of infection or fainting is very small. Inflammation or clotting of a vein also may rarely occur.
**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Some of your blood will be sent to other laboratories within the NIH to examine your inflammation levels. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.

- 4. **Stool sample collection** has no risk, and should only take a moment to complete. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.
- 5. **Urine sample collection** has no risk and should only take a moment to complete. If you do test positive for an illicit substance, the result will be part of your NIH Medical Record.
- 6. **Questionnaires** are not risky, but may be inconvenient because of the time necessary to complete them.
- 7. **Oral glucose tolerance test.** This test is inconvenient because of the time it takes to complete. The only risks from this kind of study are those described for any blood draw, as well as developing nausea from the oral glucose. Patients may transiently develop high blood sugar levels from the glucose, but it should normalize within a few hours and should not be clinically significant.
- 8. **Intravenous glucose tolerance test.** This test is inconvenient because of the time it takes to complete. You can watch TV during this test. The only risks from these kinds of studies are those described for any blood draw, the possibility of slight arm tenderness in the arm receiving the sugar infusion, (this tenderness goes away within a few minutes with gentle rubbing of the arm), and the possibility of a low blood sugar during the study. With slightly low blood sugars (less than 50 mg/dL), participants may get hungry, have a headache, feel shaky or dizzy, may become drowsy, or may become sweaty. With very low blood sugars (under 30 mg/dL) participants may have trouble speaking, be difficult to arouse, and even have seizures. However, in the test we are doing, we will be giving you extra sugar to raise your blood sugar above normal, and then we will try to bring it back to normal (95-105 mg/dL) with insulin. To do this, we will measure blood sugar at 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, and 180 minutes (a total of 3 hours). A physician or nurse practitioner will be present during the first hour of your test to make sure everything is working properly. We expect that the chance of even a slightly low blood sugar is very low. If a low blood sugar does not come up on its own quickly, the test will be stopped and you will be given sugar by vein to raise the blood sugar to normal.
- 9. Fat tissue biopsies. Possible side effects of the biopsy procedure are pain during and for two to three days after the procedure, although rarely the biopsy site may be tender or sore or have bruising or swelling for 2-3 weeks. Biopsy wounds usually heal with a very small, nearly unnoticeable scar, but sometimes a raised scar (keloid) or visible lump may result. Your risk is slightly higher if you are African American. Lidocaine injection for numbing before fat biopsies may cause some mild burning before the numbing takes effect. Rare adverse effects include infection at the biopsy sites or an allergic reaction to Lidocaine that may lead to a rash and/or swelling of the injected area. If you know you are allergic to Lidocaine, we will change to another local anesthetic. Another risk of the procedure is minor bleeding in the area of the biopsy. Some medications may increase the amount of bleeding from the biopsy. If you are taking medications such as Coumadin, Plavix or aspirin to thin your blood, you WILL NOT have a biopsy. If you are taking aspirin or non-steroidal medications such as Advil for pain you will need to stop taking these medicines for one week before the biopsy is performed.
- 10. **DNA testing.** If you allow us to study your DNA, we will use it for genome sequencing. Genome sequencing is a test that could give us different kinds of results. These include:
  - a. We could identify changes in genes that are related to metabolism and body weight.
  - b. We could identify changes in genes that contribute to other diseases or problems.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

c. We could identify changes in genes that are not known to cause any disease. These are known as normal variations.

d. We could find changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

One of the goals of this study is to identify changes in genes that may be involved in obesity. This research may take years. If however we identify a genetic cause or likely cause of obesity, with your permission, we will contact you. Please let us know your preference by initialing one of these three statements:

| I would like to be contacted with information about the progress of this study and contacted about any results related to obesity. I understand that this research will take years and that a specific abnormality might not be identified in me. |
|---|
| Please do not contact me regarding the progress of this study or any specific gene changes related to obesity. |
| I do NOT authorize any genetic samples to be collected during these NIH visits. |

Identifying gene changes that are not related to the condition being studied is known as <u>incidental medical information</u>. We will find gene changes in everyone that we study, but currently we are only specifically looking for genes related to metabolism and body weight. Even so, some gene changes not related to metabolism and body weight might be detected.

We will only inform you only of changes that have **urgent medical significance** and would benefit from early medical treatment. An example of this would be a gene change that causes cancer and where you would benefit from early screening. We will not inform you of all gene changes that have uncertain health implications or that only predispose individuals to disease. An example of this would be a gene change that influences the risk of heart disease, but where the development of the disease is dependent on many genetic and non-genetic (such as diet and smoking) factors. Also we will not inform you of gene changes that may have reproductive consequences, such as impotence or infertility.

If we find a gene change of urgent medical significance, we will only be able to give you those results once the change has been confirmed in a certified laboratory. For this confirmation, we will ask for a new sample of DNA from you. In most cases this will involve obtaining a small sample of blood (1-2 teaspoons). Sometimes we can obtain enough DNA to confirm your genetic change by swiping the insides of your cheek.

Once a gene change is confirmed, we will discuss the results with you and make recommendations regarding appropriate medical follow up. The NIH cannot promise to perform or pay for recommended medical tests or evaluations. Also, it is possible that a gene change will not be confirmed on subsequent testing. This could be due to an error in the DNA sequencing or an error in processing the DNA or cell lines. Although you likely will be glad that we did not confirm a problem, this may cause some anxiety and concern that you otherwise would not have experienced.

Please let us know your preferences by initialing one of the following statements (You are allowed to change your mind in the future):

| _ I DO want to be re-contacted if genetic variants with urgent health implications are discovered |
|---|
| during this research testing. |

## CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

\_\_\_\_\_ I DO NOT want to be re-contacted if genetic variants with urgent health implications are discovered during this research testing.

If we find a gene change with urgent health implications, the NIH can confirm the genetic change present in one member of your family. We will discuss the results with you so that you understand who else in your family could be a carrier for this same change. We can help arrange for this testing to be done, but the NIH cannot promise to perform or pay for the clinical testing necessary to confirm or determine who else in your family may have this change in their DNA.

In addition to knowing what we could find, we would like you to know the limitations of the genome sequencing and what we will NOT be able to tell you about the changes that we find.

- 1. Not all gene changes that cause disease will be detected.
- **2.** Some changes that are not currently known to cause health problems will be found to cause health problems in the future. We cannot promise to be able to tell you about those changes in the future.
- **3.** We will not tell you about gene changes that are not known to have health implications, nor will we tell you about gene changes that have only reproductive consequences.
- **4.** This gene sequencing cannot be substituted for diagnostic testing recommended by another physician.

**Emotional and psychological risks from DNA testing.** Identification of gene changes could cause emotional and psychological problems. In some situations psychological counseling could be recommended.

- 1. Learning about disease risk in your family can be distressing.
- 2. Learning that you passed on a gene that does not work to your child can be distressing.
- 3. Other members of your family could be upset to learn that they may be at risk for a disorder because of your participation in this study.

You may be falsely reassured about your health status if we do not report any changes to you.

**Other risks of genetic testing.** If we confirm a gene change in your DNA in a diagnostic laboratory, this information will become part of your medical record at the NIH. Some people are concerned that information about them from their medical records could be released. Possible problems include insurance or employment discrimination. Measures to protect the confidentiality of your information are described below. These problems may also occur if you disclose information yourself or agree to have your research records released.

There are state and federal laws that protect against genetic discrimination. A federal law called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. According to this law, health insurance companies or group health plans (as of May 21, 2010) cannot request your genetic information or use it to make decisions about your eligibility or premiums; and employers cannot use it in deciding to hire, promote, or fire you or in setting the terms of your employment (as of Nov 21, 2009).

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

The following link contains details on this policy:

http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

You may ask your research team for additional information or a copy of The Genetic Information Nondiscrimination Act of 2008 informational document.

#### **Use of stored samples and data**

**Future DNA Research.** Currently we plan to sequence known genes, which is only about 1% of your total DNA. In the future we may sequence other parts of your DNA, and it is possible that we will need to send your DNA to specialized labs outside of the NIH to do these tests. If this is done, your DNA will be coded and will not have your name or any other personally identifying information on the sample. The outside lab will have no way of identifying that the blood sample came from you.

| Please | initial <u>one</u> of the following three statements regarding future research: |
|---|---|
| | I give permission to perform future studies on my DNA without needing my additional consent. I understand I will not be contacted if these samples are used in the future. |
| | I must be contacted and give consent if my DNA samples are to be used in future research studies that are not described above in this consent form. |
| | Do not use my DNA for any future studies beyond those described above in this consent form. |
| the free<br>to send<br>stored<br>our lab<br>identify | e research with tissue samples. We plan to store some of your blood, urine, stool, and tissue samples in ezer for future studies that are not specifically outlined in this consent form. It is possible that we will need I your samples to specialized labs outside of the NIH to do these future tests. Also, these samples may be at a separate site (called a repository) that specializes in storing clinical samples. Any samples that leave will be coded and kept anonymous, and the samples will not have your name or any other personally ring information on them. In addition, it is possible that some information obtained from these studies will lished in the medical literature. However, your identity will not be included in any publications. |
| Please | initial one of the following two statements: |
| | I understand that samples collected during these NIH visits will be saved and used for future experimental testing. I authorize other uses of these samples without my additional consent. I understand I will not be contacted if these samples are used in the future. |
| | I understand that samples collected during these NIH visits will be saved and used for future experimental testing. I must be contacted and give additional consent if these samples are to be used in future studies not described above in this consent form. |

All through the process of the study and afterwards, the confidentiality of participants will be protected by using codes and medical record numbers in recording your information and test results. Only medical personnel involved in this study will have access to participants' names, test results, and patient code numbers. Should you withdraw from this study, we will keep your DNA and tissue for analysis unless you ask us to destroy the samples. You have the option, in the future, of requesting that these samples not be used for any additional testing.

# MEDICAL RECORD MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

**DNA Scientific Databases.** To do more powerful research, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. This "larger pool" of information helps enable scientific breakthroughs.

You need to be aware that DNA sequence is like a fingerprint. Theoretically if enough DNA sequence information is available, someone could identify you based on his/her DNA sequence. To facilitate genetic research, your DNA sequence information may be deposited in other databases. In this case, unless we have your permission, we will deposit the data in a manner that would not allow someone to identify you. Please understand that this information cannot be removed once it is deposited.

| riease | e initial one of the following statements: |
|---|---|
| | _ I do not want DNA sequence data to be deposited in any database other than the one associated with this study. |
| | _ My DNA sequence data can be deposited in databases that limit access to IRB (ethics board) approved-researchers. |
| | _ My DNA sequence can be deposited in a database that is available only to scientists but that does not<br>require IRB approval of research studies. I understand that someone could theoretically identify me from<br>this information. |

#### Potential benefits of participation

We are hopeful that your participation in this study will help us better understand the mechanisms of how insulin works in the body. However, you will not benefit directly from participating in this study. Should we find abnormalities in any of your test results, you will be notified and receive a copy to assist you in seeking further medical evaluation. This information may or may not improve your health.

#### Right of Withdrawal and Conditions for Early Withdrawal

You may withdraw from the study at any time and for any reason without loss of benefits or privileges to which you are otherwise entitled.

#### **Discussion of New Findings with You**

There is no general plan to share your individual test results with you. However, if any findings suggest you have a medical issue, we will provide this information to you and your primary care provider. You may request a copy of your routine laboratory tests if you desire.

#### **Study Termination**

You may be asked to end your participation in this study at any time if we believe that continuation is not in your best medical interest or if you are unable to comply with the requirements of the study.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### **Alternatives to Participation**

The alternative to this study is not to participate. You may be eligible for other studies in the NIH. You may learn more about them through <a href="https://www.clinicaltrials.gov">www.clinicaltrials.gov</a>.

#### **Compensation**

You will be compensated for the time and inconvenience associated with participation according to NIH research volunteer guidelines. Compensation for completing all of the testing described above is \$100 for the outpatient screening visit and \$300 for the baseline visit. The total amount you could receive for participation if you complete all parts of this study is \$400.

#### **Conflict of Interest**

The NIH and members of this research team have no financial interest related to this research study.

#### Posting of Research Results on www.ClinicalTrials.gov

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

| I have | received | a conv | of the | signed | consent | form |
|-----------|----------|--------|-----------|--------|----------|---------|
| <br>THAVE | received | a copy | y Oi tile | Signed | COLISCIT | 101111. |

#### MEDICAL RECORD

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- **2. Policy Regarding Research-Related Injuries.** The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Jack A. Yanovski, MD, PhD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686 or Associate Investigator Andrew Demidowich, MD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686.

You may also call the Clinical Center Patient Representative at 301-496-2626.

**5. Consent Document.** Please keep a copy of this document in case you want to read it again.

| COMPLETE APPROPRIATE ITEM(S) BELOW: | |
|---|---|
| <b>A. Adult Patient's Consent</b> I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby consent to take part in this study. | <b>B. Parent's Permission for Minor Patient.</b> I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby give permission for my child to take part in this study. (Attach NIH 2514-2, Minor's Assent, if applicable.) |
| Signature of Adult Patient/Legal Representative Date | Signature of Parent(s)/Guardian Date |
| Print Name | Print Name |
| C. Child's Verbal Assent (If Applicable) The information in the above consent was described to my child and my consent was described to my consent was descr | Print Name |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM JANUARY 24, 2018 THROUGH FEBRUARY 24, 2019. | |
| Signature of Investigator Date | Signature of Witness Date |
| Print Name | Print Name |

#### **PATIENT IDENTIFICATION**

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

NIH-2514-1 (07-09 P.A.: 09-25-0099

File in Section 4: Protocol Consent

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

INSTITUTE: Instituto Nacional de Salud Infantil y Desarrollo Humano (National Institute of Child Health and

Human Development)

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Estudio preliminario de los efectos de la colchicina en adultos no diabéticos con síndrome

metabólico

Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome)

Date Posted to Web: 08/03/18

Continuing Review Approved by the IRB on 01/24/18 Amendment Approved by the IRB on 07/13/18 (S)

Evaluation Only - Spanish

MEDICAL RECORD

#### INTRODUCCIÓN

Deseamos invitarle a participar en un estudio de investigación en los Institutos Nacionales de Salud (*National Institutes of Health, NIH*).

En primer lugar, queremos que Ud. sepa que:

La participación en una investigación del NIH es totalmente voluntaria.

Usted puede decidir no participar o retirarse del estudio en cualquier momento. En cualquier caso, no perderá ninguna compensación a la que pueda tener derecho. No obstante, para recibir atención médica en el NIH usted debe participar en un estudio o estar en evaluación para participar en uno.

Es posible que no reciba ningún beneficio por su participación. Con la investigación podemos adquirir conocimientos que ayuden a otras personas en el futuro.

En segundo lugar, algunas personas pueden tener creencias personales, religiosas o éticas que limiten los tipos de tratamientos médicos o de investigación que deseen recibir (por ejemplo, transfusiones de sangre). Si usted es una de esas personas, hable al respecto con sus médicos o con el equipo de investigación del NIH antes de acceder a participar en el estudio.

El estudio se describe en las siguientes páginas. Antes de decidir participar, tómese todo el tiempo que necesite para hacer preguntas y hablar del estudio con cualquier persona del NIH, o con su familia, amigos, médico personal o cualquier otro profesional de la salud.

#### Propósito de este Estudio

Las células grasas desempeñan numerosos papeles importantes en nuestro cuerpo, incluyendo el almacenamiento de energía, la secreción de hormonas, y ayudando a regular nuestro metabolismo. La insulina es una hormona que circula por todo el cuerpo y se comunica con las células grasas y regula su función. Cuando la capacidad de la insulina para comunicarse con el resto del cuerpo comienza a fallar, la gente se vuelve "resistente a la insulina" y pueden llegar a desarrollar diabetes. Sin embargo, los detalles específicos de cómo funciona la insulina a nivel de la célula grasa son aún poco conocidos. A propósito de este estudio es comprender mejor el tiempo y los mecanismos detrás de las acciones de la insulina en las células de grasa, y posiblemente identificar nuevos factores de por qué algunas personas son más

#### **PATIENT IDENTIFICATION**

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (4)

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

propensas a desarrollar diabetes. Le pedimos que nos ayude a entender cómo funciona la insulina en el cuerpo al someterse a una serie de pruebas. No se le pedirá que tome el medicamento de estudio (colchicina).

Los participantes del estudio tendrán que venir al Centro Clínico del NIH para dos consultas ambulatorias. Es importante que los participantes llegen en ayunas (sin alimentos ni bebidas aparte de agua) a cada una de estas visitas. Los participantes serán compensados por su tiempo y cualquier inconveniente.

#### Población de estudio

Deseamos reclutar a adultos sanos y adultos con diabetes tipo 2 tratados sólo con dieta.

#### Quién puede participar en este estudio

Usted puede ser elegible para este estudio de investigación si es mayor de 18 años de edad; pesar menos de 450 libras, y que se encuentre en buen estado de salud general.

#### Quienes no pueden participar en este estudio

Usted no puede ser elegible para este estudio si tiene una enfermedad médica grave que pudiera interferir con las pruebas o mediciones del estudio, como enfermedades del corazón, riñón, hígado, pulmón, sangre, intestinal o enfermedades endocrinas o presión arterial alta no controlada. Las personas con diabetes tipo 2 que están tomando medicamentos o tienen hemoglobina A1c> 9%, no pueden participar. Si usted está usando un medicamento que afecta el metabolismo del azúcar y la grasa o la absorción en su cuerpo, es posible que no sea elegible para participar. Tampoco son elegibles las mujeres que están embarazadas o lactando, o tienen intención de quedar embarazadas; las personas que han tenido un cambio de peso reciente superior al 3% del peso corporal total, han estado utilizando medicamentos para reducir el peso, han usado recientemente la colchicina, tener una alergia conocida a la colchicina, o utilizan productos de tabaco o nicotina (p. ej. e-cigarrillos), no serán reclutadas para este estudio. Las personas con antecedentes de formación de queloides (que fácilmente desarrollan cicatrices en su piel después de una lesión) tampoco no pueden participar en este estudio.

#### Procedimientos del estudio

PATIENT IDENTIFICATION

El estudio consta de dos visitas ambulatorias en el Centro Clínico: **una visita para determinar elegibilidad** y **una visita inicial** para estudiar su metabolismo.

Visita Ambulatoria de Selección de Pacientes

Esta visita tomará unas 3 horas para realizarse. Usted será visto en un día de semana en el Centro Clínico del NIH. Le pedimos permanecer en ayunas durante las 10 horas anteriores a su llegada a la clínica y <u>no debe comer o beber nada, excepto aqua por la mañana</u>. Durante esta visita, vamos a realizar lo siguiente:

- 1. **Protocolo y firma del formulario de consentimiento**. Vamos a repasar el estudio en detalle y a responder cualquier pregunta. El formulario de consentimiento debe ser firmado antes de poder tomar parte en el estudio.
- 2. **Historia médica completa y un examen físico**, con el peso, la altura, y la medición de la presión arterial.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

3. Un **ECG** se realizará para examinar la función de su corazón.

- 4. Los análisis de sangre en ayunas para asegurarse de que usted se encuentra en buen estado de salud. El análisis examinará el recuento de células de la sangre, función hepática y renal, niveles de colesterol, los niveles de azúcar e insulina en sangre, pruebas de función tiroidea, nivel de la inflamación, así como muestras de sangre de reserva para ser preservadas para poder examinar durante futuras investigaciónes. También realizaremos pruebas para determinar si usted tiene alguna diferencia en genes que pueden ser importantes para el metabolismo y el peso corporal. Además para buscar algunos genes que ya nosotros pensamos que son importantes para el peso corporal, vamos a utilizar nueva tecnología de secuenciación de DNA que se verá en todos los genes humanos que conocemos. Esto se conoce como "exome" y secuenciación del genoma. Esta nueva tecnología nos permite mirar el ADN en gran detalle.
- 5. **Recogida de muestras de orina** para asegurarse de que sus riñones funcionan normalmente, que no está tomando cualquier droga ilícita, y una prueba de embarazo (para las mujeres en edad fértil).
- 6. **Prueba de tolerancia a la glucosa oral**. Vamos a realizar una prueba para examinar si usted tiene diabetes, la llamamos prueba de tolerancia a la glucosa de 2 horas. Va a tomar una taza de agua con azúcar y luego se tomarán muestras 1 y 2 horas después para mirar su nivel de azúcar en la sangre.
- 7. **Absorciometría dual de rayos X (DEXA)** para examinar su composición corporal. La prueba consiste en permanecer inmóvil sobre una mesa mientras una pequeña cámara pasa sobre su cuerpo. La dosis de los rayos X es mucho menor que la cantidad que se obtiene de una radiografía de pecho normal. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos.

#### Visita Inicial

Si reúne los requisitos para participar en el estudio, se le cita para la visita inicial. Le pediremos que permanezca en ayunas durante 10 horas antes de llegar a la clínica y <u>no comer o beber nada, excepto agua por la mañana</u>. Usted será visto en un dia entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita tomará alrededor de 8 horas para completarse. Durante esta visita vamos a realizar lo siguiente:

- 1. **Intervalo de historia clínica y examen físico**, con el peso, la altura, y la medición de la presión arterial. También se completará un cuestionario.
- 2. **Los análisis de sangre en ayunas** para mirar su metabolismo basal y los niveles inflamatorios, así como muestras de sangre de reserva para ser preservados para las pruebas de investigación adicionales posibles, incluyendo una muestra para futuro análisis genético. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener las muestras de sangre.
- 3. Obtención **de muestras de heces**, obtendremos dos muestras de heces para conservar para futuros experimentos. Como parte de esta colección, le pediremos que mantenga un record de su dieta por 24 horas en un formulario que se le entregara a usted, y asi ver como la dieta puede afectar los resultados de las pruebas de heces. Los resultados de este "diario de nutricion" irá con un nutricionista.
- 4. Obtención **de muestras de orina** como se describe antes. También vamos a recoger la orina durante su visita a ahorrar para futuros experimentos.

## CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

5. **Prueba de tolerancia a la glucosa intravenosa muestreado frecuentes**. Este estudio nos dice mucho acerca de cómo su cuerpo utiliza el azúcar, qué tan bien está funcionando su insulina y cómo es la sensibilidad de su cuerpo a la insulina. El estudio FSIVGTT se hace mientras usted descansa en una cama. Una segunda línea IV se coloca en su brazo. Le daremos un poco de agua de azúcar en una vía intravenosa durante un período de 2 minutos. Entonces vamos a tomar muestras de sangre de la otra IV en -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, y 180 minutos (un total de 3 horas ) para medir los niveles de azúcar e insulina . Exactamente a los 20 minutos en la prueba, le daremos una pequeña cantidad de insulina a través de la IV. Un médico o enfermera practicante estará presente durante la primera hora del estudio. Usted puede ver la televisión durante esta prueba.

- 6. Tomografía Computarizada (TC) del abdomen para observar donde se tiende a almacenar su grasa. La prueba consiste en permanecer quieto en una mesa móvil que pasa por un gran anillo donde esta ubicada la cámara. La prueba implica radiación, pero solo porque tomaremos una foto de su abdomen, el método que se utilizará minimiza su exposición. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos
- 7. **Subcutánea Biopsia de grasa**. Para examinar el nivel de ciertas moléculas en el tejido graso, se tomará una pequeña muestra de tejido graso de debajo de la piel de su abdomen. Para adormecer el área donde se tomarà la muestra, se utilizará la lidocaína, un anestésico local. Una aguja se utilizará para extraer una porción de tejido graso que mide alrededor de 1 ½ cucharaditas. Un vendaje se aplica entonces al sitio de inserción de la aguja. Podemos darle algún medicamento para el leve dolor, como Tylenol o medicamento más fuerte si es necesario, después de la biopsia. La biopsia se tomará de un lugar del cuerpo que normalmente está cubierto y que no se ve fácilmente.

Cuando el estudio se haya completado, volverá al cuidado de su médico de cabecera. La participación en este estudio no compromete al NIH a su cuidado a largo plazo.

#### Los resultados de pruebas realizadas en el NIH

Estaremos midiendo muchas cosas en su sangre durante sus visitas, y podríamos descubrir algún problema médico que requiere tratamiento. Ud. no recibirá de forma rutinaria tratamiento para cualquier condición de salud descubierto. Sin embargo, se le informará sobre estos hallazgos (por ejemplo: presión arterial alta) y cualquier información de importancia médica que resulten de análisis de sangre o del examen físico, serán remitidos a su médico de atención primaria en su solicitud. Algunos de estos problemas médicos podrían impedir su participación más en el estudio.

#### Riesgos y molestias

PATIENT IDENTIFICATION

- 1. **El examen físico**. Un médico o una enfermera puede tener que le examinar pidiéndole que se quite su ropa, con las precauciones adecuadas para proteger su privacidad. Algunos pueden encontrar este examen vergonzoso.
- 2. **Exposición a la radiación**: Este estudio de investigación implica la exposición a la radiación de tres imagenes DEXA y tres tomografías computarizadas. Tenga en cuenta que esta exposición a la radiación no es necesario para su atención médica y es sólo para fines de investigación. El Comité de Seguridad Radiológica NIH ha revisado el uso de la radiación en este estudio de investigación y ha aprobado este uso ya que implica un riesgo mínimo y necesario para obtener la información de investigación deseada.

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Aunque cada órgano recibirá una dosis diferente, la cantidad de exposición a la radiación que recibirá anualmente de este estudio es igual a una exposición uniforme de todo el cuerpo a 0.031 rem. Este valor calculado se conoce como la "dosis efectiva" y se utiliza para relacionar la dosis recibida por cada órgano a un solo valor. La cantidad de radiación que recibirá en este estudio es inferior a la pauta de dosis establecido por el Comité de Seguridad Radiológica NIH para los sujetos de investigación. Esta pauta establece una dosis efectiva de 5 rem recibido por año.

Por comparación, la persona promedio en los Estados Unidos recibe una exposición a la radiación de 0,3 rem por año a partir de fuentes naturales, como el sol, el espacio exterior, y de materiales radiactivos que se encuentran naturalmente en el aire y el suelo. Si desea más información sobre la radiación y los ejemplos de los niveles y forma de exposicion a otras fuentes, por favor pregunte al investigador para obtener una copia del folleto titulado, An Introduction to Radiation for NIH Research Subjects.

3. **La extracción de sangre**. La cantidad de extracción de sangre es muy por debajo de la directriz del NIH para una cantidad segura de extracción de sangre (550 cc cada 8 semanas). Un pequeño moretón se puede formar en cualquier sitio donde se toma la sangre. El riesgo de infección o desmayo es muy pequeña. La inflamación o coagulación de una vena también pueden ocurrir raramente.

Una parte de su sangre será enviada a otros laboratorios dentro del NIH para examinar sus niveles de inflamación. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras

- 4. Recogida de muestras de heces no tiene ningún riesgo, y sólo debe tomar un momento para recogerlas. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras.
- 5. **La recogida de muestras de orina** no tiene ningún riesgo y sólo toma un momento para completar. Si el resultado es positivo para una sustancia ilícita, el resultado será parte de su expediente médico NIH.
- 6. **Los cuestionarios no son peligrosos**, pero pueden ser un inconveniente debido al tiempo necesario para su realización.
- 7. **Prueba oral de tolerancia a la glucosa**. Esta prueba es un inconveniente debido al tiempo que se tarda en completar. Los únicos riesgos de este tipo de estudio son las descritos para cualquier extracción de sangre, así como el desarrollo de las náuseas por la glucosa oral. Algunos pacientes pueden desarrollar de forma transitoria niveles altos de azúcar en la sangre a partir de la glucosa, pero deben normalizarse a las pocas horas y no deben ser clínicamente significativos.
- 8. **Prueba de tolerancia a la glucosa intravenosa**. Esta prueba es un inconveniente debido al tiempo que se tarda en completar. Usted puede ver la televisión durante esta prueba. Los únicos riesgos de este tipo de estudios son las descritas para cualquier extracción de sangre, la posibilidad de una ligera sensitividad en el brazo al recibir la infusión de azúcar, (esa sensitividad desaparece al cabo de unos minutos con el roce suave del brazo), y la posibilidad de un bajo nivel de azúcar en la sangre durante el estudio. Cuando la azúcar en sangre esta baja (menos de 50 mg/dl), los participantes pueden tener hambre, tener dolor de cabeza, sentirse temblorosos o mareados o pueden llegar a ponerse sudorosos. Con azúcar en la sangre muy bajos (menos de 30

# MEDICAL RECORD MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

mg /dl) participantes pueden tener problemas para hablar, dificultad para despertar, e incluso tener convulsiones.

Sin embargo, en la prueba que estamos haciendo, le estaremos dando azúcar extra para elevar el azúcar en la sangre por encima de lo normal, y luego vamos a tratar de traerlo de vuelta a la normalidad (95-105 mg / dL) con insulina. Para ello, vamos a medir el azúcar en la sangre a los 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, y 180 minutos (un total de 3 horas). Un médico o enfermera practicante estará presente durante la primera hora de su prueba para asegurarse de que todo funciona correctamente. Esperamos que la posibilidad de un nivel de azúcar en sangre bajo sea muy pequeña. Si un bajo nivel de azúcar en la sangre no sube por sí sola con rapidez, se detendrá la prueba y se le dará el azúcar por vía IV para elevar el azúcar en la sangre a la normalidad

- 9. Biopsias de grasa. Los posibles efectos secundarios de la biopsia son el dolor durante y durante dos o tres días después del procedimiento. Aunque rara vez, la zona de la biopsia puede estar sensible o adolorida o tener moretones o hinchazón durante 2-3 semanas. Heridas biopsia suelen sanar con una cicatriz muy pequeña, casi imperceptible, pero a veces una cicatriz elevada (queloides) o bulto visible puede resultar. Su riesgo es ligeramente mayor si usted es afroamericano. Inyección de lidocaína para adormecer antes de biopsias de grasa puede causar un poco de ardor suave antes de que llegue el entumecimiento. Efectos adversos raros incluyen la infección en los sitios de biopsia o una reacción alérgica a la lidocaína que puede llevar a una erupción y/o hinchazón de la zona de inyección. Si usted sabe que es alérgico a la lidocaína, cambiaremos a otro anestésico local. Otro de los riesgos del procedimiento es sangrado menor en el área de la biopsia. Algunos medicamentos pueden aumentar la cantidad de sangrado de la biopsia. Si está tomando medicamentos como Coumadin, Plavix o aspirina para adelgazar la sangre, usted no tendrá una biopsia. Si está tomando aspirina o medicamentos no esteroides como Advil para el dolor tendrá que dejar de tomar estos medicamentos durante una semana antes de realizar la biopsia.
- 10. **Las pruebas de ADN.** Si nos permite estudiar su ADN, lo vamos a utilizar para la secuenciación del genoma. La secuenciación del genoma es una prueba que nos podrían dar diferentes tipos de resultados. Estos incluyen:
  - a. Podríamos identificar cambios en los genes que están relacionados con el metabolismo y el peso corporal.
  - b. Podríamos identificar cambios en los genes que contribuyen a otras enfermedades o problemas.
  - c. Podríamos identificar los cambios en los genes que no son conocidos por causar ninguna enfermedad. Estos son conocidos como variaciones normales.
  - d. Podríamos encontrar cambios en los genes que son nuevos y de importancia clínica incierta. Esto significa que no se sabe si podrían causar o contribuir a una enfermedad o si son variaciones normales.

Uno de los objetivos de este estudio es identificar los cambios en los genes que pueden estar implicados en la obesidad. Esta investigación puede tomar años. Sin embargo, si se identifica una causa genética o la causa probable de la obesidad, con su permiso, nos pondremos en contacto con usted. Por favor, háganos saber su preferencia con sus iniciales en una de estas dos declaraciones:

| <br>Me gustaría ser contactado con la información sobre los avances de este estudio y contactado acerca de cualquier resultado relacionado con la obesidad. Entiendo que esta investigación llevará años y que una anormalidad específica no se puede identificar en mí. |
|---|
| <br>Por favor no se contacte conmigo acerca de la marcha de este estudio o cualquier cambio de genes específicos relacionados con la obesidad. |

**MEDICAL RECORD** 

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Yo no autorice ninguna muestras genéticas que se recojan durante estas visitas NIH.

La identificación de cambios genéticos que no están relacionados con la condición que se está estudiando, se conoce como <u>información médica incidental</u>. Vamos a encontrar cambios genéticos en todo el mundo que estudiamos, pero estamos mirando sólo específicamente para los genes relacionados con el metabolismo y el peso corporal. Aun así, algunos cambios en los genes no relacionados con el metabolismo y el peso corporal se detectarán.

Nosotros sólo le informaremos de los cambios que tienen **importancia médica urgente** y se beneficiarían de un tratamiento médico temprano. Un ejemplo de esto sería un cambio en el gen que causa cáncer y en la que se beneficiaría de la detección temprana. No le informará de todos los cambios en los genes que tienen inciertas implicaciones para la salud. No vamos a informar de los cambios genéticos que predisponen a los individuos sólo a la enfermedad. Un ejemplo de esto sería un cambio en el gen que influye en el riesgo de enfermedades del corazón, pero en el que el desarrollo de la enfermedad depende de muchos factores genéticos y no genéticos (tales como la dieta y el tabaquismo). Además, no le informaremos de cambios genéticos que pueden tener consecuencias reproductivas, tales como la impotencia o infertilidad.

Si detectamos un cambio genético que podría ser importante para usted, sólo le daremos los resultados si el cambio ha sido confirmado por un laboratorio certificado. Por esta confirmación, le pediremos una nueva muestra de ADN a usted. En la mayoría de los casos esto implicará la obtención de una pequeña muestra de sangre (1-2 cucharaditas). A veces podemos obtener suficiente ADN para confirmar su cambio genético al golpear el interior de la mejilla.

Una vez que se confirma un cambio en un gen, vamos a discutir los resultados con usted y hacer recomendaciones sobre apropiado seguimiento médico. El NIH no puede prometer realizar o pagar por los exámenes médicos recomendados o evaluaciones. Es posible que un cambio genético no se confirmará en las pruebas posteriores. Esto podría ser debido a un error en la secuenciación de ADN o un error en el procesamiento del ADN o líneas celulares. Aunque es agradable para Ud. que no se confirme el problema, esto puede causar un poco de ansiedad y preocupación que de otra manera no habría experimentado.

Por favor, háganos saber sus preferencias colocando sus iniciales en una de las siguientes afirmaciones:

urgentes para la salud durante esta prueba de investigación.

| Yo QUIERO ser re-contactado si se descubren variantes genéticas con consecuencias urgentes |
|---|
| para la salud, durante esta prueba de investigación. |
| NO deseo volver a ser contactado si se descubren variantes genéticas con consecuencias |

Si usted tiene un cambio en un gen con urgentes implicaciones para la salud, el NIH confirmará el cambio genético presente en uno de los miembros de su familia. Discutiremos los resultados con usted para que pueda saber si alguien más en su familia podría ser un portador de este mismo cambio. Podemos ayudarle a organizar las pruebas que haya que hacer, pero el NIH no podemos prometer realizar o pagar por las pruebas clínicas necesarias para confirmar o determinar quién más en su familia puede tener este cambio en su ADN.

Además de saber lo que encontramos, nos gustaría que conociera las limitaciones de la secuenciación del genoma y lo que no vamos a ser capaces de decirle acerca de los cambios que encontramos.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

1. No todos los cambios en los genes que causan la enfermedad serán detectados.

- 2. Algunos de los cambios que no se conocen actualmente para causar problemas de salud podrían causar problemas de salud en el futuro. No podemos prometer tener la capacidad de decirle a usted acerca de esos cambios en el futuro.
- 3. No le dirá acerca de cambios en los genes que no se sabe que tienen consecuencias para la salud, ni vamos a informarle sobre cambios en los genes que sólo tienen consecuencias reproductivas.
- 4. Esta secuenciación de genes no puede ser sustituido por las pruebas de diagnóstico recomendado por otro médico.

**Riesgos emocionales y psicológicos de la prueba de ADN**. La identificación de los cambios en los genes puede causar problemas emocionales y psicológicos. En algunas situaciones, se podría recomendar asesoría psicológica.

- 1. Aprender sobre el riesgo de enfermedad que en su familia puede ser angustiante.
- 2. Aprender que algo que sucede en un gen suyo, puede no suceder en su hijo, puede ser angustiante.
- 3. Otros miembros de su familia podrían ponerse molestos al saber que ellos pueden estar en riesgo de un trastorno debido a su participación en este estudio.

Ud. Puede permanecer falsamente tranquilo acerca de su estado de salud si nosotros no le reportamos ningún cambio en su caso.

**Otros riesgos de las pruebas genéticas.** Si confirmamos un cambio genetico en su ADN en un laboratorio de diagnóstico, esta información será parte de su expediente médico en el NIH. Algunas personas se preocupan de que la información acerca de ellos de sus registros médicos podrían ser dadas a conocer. Posibles problemas incluyen el seguro o la discriminación laboral. Medidas para proteger la confidencialidad de su información se describen a continuación. Estos problemas también pueden ocurrir si usted divulga su propia información o acepta que sus registros de investigación sean liberados.

Hay leyes estatales y federales que protegen contra la discriminación genética. Una ley federal llamada la Ley de No Discriminación por información Genética (GINA), generalmente hace que sea ilegal que las compañías de seguros de salud, planes de salud de grupo, y la mayoría de los empleadores discriminen contra usted basado en su información genética. Según esta ley, las compañías de seguros de salud o planes de salud de grupo (hasta el 21 de mayo de 2010) no puede solicitar su información genética, o utilizarlo para tomar decisiones sobre su elegibilidad o primas; y los empleadores no pueden utilizarlo en la decisión de contratar, promover, ni puede despedirlo, o en el establecimiento de los términos de su empleo (a fecha de 21 de noviembre 2009).

Tenga en cuenta que esta ley federal no le protege contra la discriminación genética por las compañías que venden seguros de vida, seguro de invalidez, o un seguro de cuidado a largo plazo. Este enlace contiene detalles sobre esta política: http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf

Usted puede preguntar a su equipo de investigación para obtener información adicional o una copia de la Ley de No Discriminación por Información Genética de 2008 documento informativo.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### El uso de muestras almacenadas y datos

**Investigaciones futuras ADN**. Actualmente tenemos la intención de secuenciar los genes conocidos, que representa sólo alrededor del 1% de su secuencia de ADN. En el futuro podemos secuenciar otras partes de su ADN, y es posible que pueden ser enviadas a otros laboratorios para pruebas específicas. Si esto se hace el ADN será codificado y no tendrá su nombre o cualquier otra información de identificación personal en la muestra. El laboratorio externo no tendrá manera de identificar que la muestra de sangre provenía de ti.

| Por favor, coloque su inicial en <u>una</u> de las siguientes tres declaraciones relativas a la investigación futura: |
|---|
| Yo doy permiso para realizar futuros estudios sobre mi ADN sin necesidad de mi consentimiento adicional. Entiendo que no se pondrá en contacto si se utilizan estas muestras en el futuro. |
| Debo ser contactado y dar consentimiento si estas muestras se van a utilizar en futuros estudios de investigación que no se describen más arriba en este formulario de consentimiento. |
| No utilice mi ADN para futuros estudios más allá de los descritos anteriormente en este formulario de consentimiento. |
| Futuras investigaciones con muestras. Tenemos la intención de almacenar algunos muestras de su sangre, orina, heces, y tejidos en el congelador para futuros estudios que no se describen específicamente en este formulario de consentimiento. Es posible que necesitáramos para enviar sus muestras a laboratorios especializados fuera del NIH para hacer estas pruebas futuras. Además, estas muestras pueden almacenarse a u sitio separado (llamado un repositorio) que se especializa en el almacenamiento de muestras clínicas. Cualquier muestra que dejan nuestro laboratorio serán codificados y se mantiene en el anonimato, y las muestras no tendrán su nombre o cualquier otra información de identificación personal sobre ellos. Además, es posible que alguna información obtenida de estos estudios serán publicados en la literatura médica. Sin embargo, su identidad no será incluida en cualquier publicación. |
| Por favor, coloque su inicial en <u>una</u> de las dos afirmaciones siguientes: |
| Entiendo que las muestras recogidas durante estas visitas NIH serán guardadas y utilizadas para futuros ensayos experimentales. Autorizo a otros usos de estas muestras sin mi consentimiento adicional. Entiendo que no se pondrán en contacto si se utilizan estas muestras en el futuro. |
| Entiendo que las muestras recogidas durante estas visitas NIH serán guardadas y utilizadas para futuros ensayos experimentales. Debo ser contactado y dar consentimiento si estas muestras se van a utilizar en en futuros estudios no descritas anteriormente en este formulario de consentimiento. |

Durante todo el proceso de estudio y después, la confidencialidad de los participantes será protegida mediante el uso de códigos y números de historia clínica en la grabación de su información y resultados de pruebas. Sólo el personal médico involucrado en este estudio tendrán acceso a los nombres de los participantes, resultados de exámenes, y los números de código de los pacientes. En caso de retirarse de este estudio, vamos a mantener su ADN para el análisis a menos que usted nos pida destruir las muestras de ADN. Usted tiene la opción, en el futuro, de solicitar que estas muestras no se pueden usar para cualquier prueba adicional.

Bases de datos científicos de ADN. Para hacer la investigación más potente, es de gran ayuda para los

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

investigadores compartan la información que reciben de estudio de muestras humanas. Lo hacen mediante la puesta en una o más bases de datos científicas, donde se almacena junto con la información de otros estudios. Este "grupo más grande" de la información ayuda a permitir avances científicos.

Usted tiene que ser consciente de que la secuencia de ADN es como una huella digital. Teóricamente si suficiente información de la secuencia de ADN está disponible, alquien podría identificarlo a Ud. en base a su secuencia de ADN. Para facilitar la investigación genética, la información de su secuencia de ADN se puede depositar en otras bases de datos. En este caso, a menos que tengamos su permiso, vamos a depositar los datos de una manera que no permita que alguien le identifique. Por favor, comprenda que esta información no se puede eliminar una vez que se deposita.

| Poi Tavoi, coloque su illiciai | en <u>una</u> de las sigulentes casillas. |
|---|---|

| No quiero que los datos de secuencia de ADN sean depositados en cualquier base de datos que no sea la que está asociada con este estudio. |
|---|
| <br>Mis datos de secuencias de ADN pueden ser depositados en las bases de datos que limitan el acceso a la IRB (comité de ética) Investigadores aprobados. |
| Mi secuencia de ADN puede ser depositada en una base de datos que está disponible sólo para los científicos, pero que no requiere la aprobación del IRB de estudios de investigación. Entiendo que alguien teóricamente me podía identificar de esta información. |

#### Los beneficios potenciales de la participación

Day favor and area are initial and the day of a large inviewban and illary

Tenemos la esperanza de que su participación en este estudio nos ayudará a comprender mejor los mecanismos de cómo funciona la insulina en el cuerpo. Sin embargo, no se beneficiará directamente de participar en este estudio. Al encontrar anomalías en cualquiera de sus resultados de la prueba, se le notificará y recibirá una copia para ayudarle en la búsqueda de una mayor evaluación médica. Esta información puede o no mejorar su salud.

#### Derecho de revocación y Condiciones de retiro anticipado

Usted puede retirarse del estudio en cualquier momento y por cualquier motivo y sin pérdida de beneficios o privilegios a los que tiene derecho.

#### La discusión de los nuevos hallazgos con usted

No hay plan general para compartir los resultados de sus pruebas individuales con usted. Sin embargo, si algún hallazgo sugiere que tiene un problema médico, vamos a proporcionar esta información a usted y a su proveedor de atención primaria. Usted puede solicitar una copia de sus pruebas de laboratorio de rutina si lo desea.

#### **Terminación de Estudios**

Es posible que terminamos su participación en este estudio en cualquier momento, si creemos que la continuación en él no es lo mejor para su interés médico o si no puede cumplir con los requisitos del estudio.

#### Alternativas a la Participación

PATIENT IDENTIFICATION

La alternativa a este estudio es no participar. Usted puede ser elegible para otros estudios en los NIH. Usted puede aprender más sobre ellos a través de www.clinicaltrials.gov.

#### Compensación

Usted será compensado por el tiempo y los inconvenientes asociados a la participación según las directrices de compensación para voluntarios de investigación del NIH. La compensación para completar todas las pruebas que se han

P.A.: 09-25-0099

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

descrito anteriormente es: \$100 por la Visita Ambulatoria de Selección de Pacientes, y \$300 por la Visita Inicial. La cantidad total que usted podría recibir por la participación si completa todas las partes de este estudio es de \$400.

#### **Conflicto de intereses**

El NIH y los miembros de este equipo de investigación no tienen ningún interés financiero en relación con este estudio de investigación.

#### Publicación de Resultados de Investigación en: www.ClinicalTrials.gov

Una descripción de este ensayo clínico estará disponible en http://www.Clinicaltrials.gov, como lo requiere la ley de Estados Unidos. En esta pagina de web no incluirá información que pueda identificarlo. En la mayor parte del sitio Web incluirá un resumen de los resultados. Usted puede buscar en este sitio web en cualquier momento.

\_\_\_\_\_ He recibido una copia del formulario de consentimiento firmado.

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

**MEDICAL RECORD** 

Adult Patient or Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### INFORMACIÓN PERTINENTE ADICIONAL

**1. Confidencialidad**. Cuando los resultados de un estudio de investigación del NIH se dan a conocer en revistas médicas o reuniones científicas, no se menciona la identidad de los participantes. En la mayoría de los casos, el NIH no divulgará ninguna información sobre su participación en la investigación a menos que usted otorgue su permiso por escrito. No obstante, si usted firma una autorización de divulgación de información, por ejemplo, a una empresa aseguradora, el NIH le proporcionará a ésta información de su expediente médico. Esta información podría influir (en forma favorable o desfavorable para usted) la disposición de la aseguradora a venderle el seguro.

La Ley Federal de Protección de la Vida Privada (Federal Privacy Act) protege el carácter confidencial de sus expedientes médicos en el NIH. Sin embargo, es importante que sepa que esta ley permite la divulgación de cierta información de su expediente médico sin su autorización, por ejemplo, si lo solicitan la Administración de Alimentos y Medicamentos (FDA), los miembros del Congreso, los agentes encargados del cumplimiento de la ley o las organizaciones autorizadas para efectos de acreditación hospitalaria.

- **2. Normas sobre lesiones relacionadas con la investigación**. El Centro Clínico le dará atención médica a corto plazo para cualquier lesión que se deba a su participación en una investigación que se realice allí. En general, ni los Institutos Nacionales de Salud, ni el Centro Clínico, ni el gobierno federal le darán atención médica a largo plazo ni indemnización económica por lesiones relacionadas con la investigación. Sin embargo, usted tiene derecho a buscar una compensación legal si cree que la lesión justifica dicha medida.
- **3. Pagos**. El monto del pago que reciben los voluntarios de investigación se rige por las normas de los Institutos Nacionales de Salud. En general, a los pacientes no se les paga por participar en los estudios de investigación en los Institutos Nacionales de Salud. Se le ofrecerá el reembolso de gastos de viaje y viáticos según las pautas del NIH.
- **4. Problemas o preguntas**. Si hay algún problema o usted tiene una pregunta con respecto a este estudio, a sus derechos como participante en un estudio de investigación clínica o a cualquier lesión relacionada con la investigación, debe comunicarse con el Investigador Principal, Jack A. Yanovski, MD, PhD; Building (Edificio) 10, Room (Sala) 1-3330, Teléfono: (301) 496-4686 o el Investigador Asociado Principal, Andrew Demidowich, MD; Building 10, Room 1-3330, Teléfono: (301) 496-4686.

También puede llamar al representante de los pacientes del Centro Clínico, al teléfono (301) 496-2626.

**5. Documento de consentimiento.** Le sugerimos que conserve una copia de este documento para consultarla posteriormente.

**PATIENT IDENTIFICATION** 

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

#### MEDICAL RECORD

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119

CONTINUATION:  pages

| COMPLETE LAS CASILLAS CORRESPONDIENTES A CONTINUACION: | |
|---|---|
| A. Consentimiento de un paciente adulto. He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo mi consentimiento para participar en este estudio. | B. Permiso otorgado por el (los) padre(s) de un paciente menor de edad. He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo permiso para que mi hijo participe en este estudio. (Anéxese el formulario NIH 2514-2, Asentimiento de un menor de edad, si corresponde.) |
| Firma del paciente adulto o su representante legal Fecha | Firma del (los) padre(s) o del tutor legal Fecha |
| Nombre en letra de imprenta | Nombre en letra de imprenta |
| C. Asentimiento verbal de un niño (si corresponde) Se le explicó a mi hijo la información contenida en el presente documento y Firma del (los) padre(s) o del tutor legal Fecha | mi hijo está de acuerdo en participar en el estudio. Nombre en letra de imprenta |
| EL USO DE ESTE DOCUMENTO DE CONSENTIMIENTO ESTÁ APROBADO DESDE EL 24 DE ENERO DE 2018 HASTA EL 24 DE FEBRERO DE 2019. Firma del Investigador Fecha Firma del testigo Fecha | |
| Nombre en letra de imprenta | Nombre en letra de imprenta |

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD

• Adult Patient or • Parent, for Minor Patient

INSTITUTE: National Institute of Child Health and Human Development

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome

Continuing Review Approved by the IRB on 01/24/18

Amendment Approved by the IRB on 07/13/18 (S)

Date Posted to Web: 08/03/18

Open-Label Arm

#### **INTRODUCTION**

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

#### Purpose of this Study

Approximately 30% of adults in the US have a body mass index (BMI) over 30 kg/m², and are at greater risk for a number of medical problems, including high blood pressure, high blood cholesterol, high triglyceride levels, high blood sugar (diabetes) and heart disease. It is thought that being overweight leads to a state of low-level inflammation and this inflammation may actually lead to some of the medical problems associated with obesity. The purpose of this study is to find out if a medication called colchicine can improve metabolism in adults who have medical complications of their high body weight (these complications are sometimes called the "metabolic syndrome"), and who have developed high blood sugar (diabetes).

#### **PATIENT IDENTIFICATION**

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent (5)

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Colchicine is an anti-inflammatory medication that has been used for centuries in the treatment of gout. From animal studies and human studies there is some evidence that anti-inflammatory medicines like colchicine may improve the pancreas's ability to secrete insulin and the body's ability to regulate sugar. We ask you to join our study, so we can find out whether colchicine can improve sugar regulation and metabolic parameters.

If you qualify and agree to participate, you will be one of seven people with Type 2 Diabetes (T2DM) assigned to take colchicine tablets by mouth twice a day for 3 months. The colchicine tablets will come in the same dose that is available in pharmacies and is prescribed for a disease called "gout": 0.6 milligrams.

When the study is completed, we will send all participants information about the results, and tell them if taking colchicine helped improve their metabolic syndrome or diabetes.

Study participants will need to come to the NIH Clinical Center for four outpatient visits, with an optional fifth outpatient visit. It is important that participants arrive fasting (no food or beverages besides water) to each of these visits. Participants will be compensated for their time and inconvenience (see below: *Compensation* on page 5).

#### **Study Population**

We wish to recruit seven overweight adults with diet-controlled T2DM.

#### **Who Can Be in This Study**

You may be eligible for this research study if you are greater than 18 years old, have a body mass index that is at least 30 kg/m² (calculated by dividing weight in kg by height in meters squared), weigh less than 450 lbs, and are in good general health. You also have to meet certain levels for insulin resistance and inflammation, as measured by lab testing, and have type 2 diabetes managed with diet to participate in the full study. If you are a woman of child-bearing age, you will be asked to use an effective form of birth control before participating in this study.

#### Who May Not Be In This Study

You may not be eligible for this study if you have a major medical illness that would interfere with study tests or measurements, such as heart, kidney, liver, lung, blood, gut, or endocrine diseases, or uncontrolled high blood pressure. If you are currently using a medication that affects sugar and fat metabolism or absorption in your body, or a medicine that should not be taken with colchicine, you may not be eligible to participate. Also individuals who are pregnant or nursing, or planning to become pregnant, have had a recent weight change greater than 3% of total body weight, have been using weight reducing medications, have recently used colchicine, have a known allergy to colchicine, or use tobacco or nicotine (e.g. e-cigarettes) products will not be recruited for this study. Individuals with a history of keloid formation (who easily develop scars on their skin after an injury) are advised not to take part in this study.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### **Procedures of the study**

The study consists of four outpatient visits: an **outpatient screening visit** at the Clinical Center to determine eligibility, a **baseline visit** to study your metabolism before the intervention, a **short outpatient** visit to check how you are feeling, and a **final visit** 3 months after the baseline visit look for changes after the intervention. Upon completing the final visit, you have the option to return 3 months later to come for another **washout visit**. This visit will look to see if the changes from the intervention continue to last even after stopping the study medication. You will be given the study medication (colchicine) on the day you complete the baseline visit.

#### **Outpatient Screening Visit**

This visit will take about 3 hours to complete. You will be seen on a weekday in the Clinical Center at the National Institutes of Health. We ask that you remain fasting for 10 hours before coming to the clinic and have nothing to eat or drink except water that morning. During this visit, we will perform the following:

- 1. **Protocol review and signing of consent form**. We will go over the study in detail, and answer any questions. The consent form will need to be signed before you can take part in the study.
- 2. **Complete medical history and physical exam,** with weight, height, and blood pressure measurement.
- 3. An **EKG** will be performed to examine your heart function.
- 4. **Fasting blood tests** to ensure that you are in good health. The analysis will examine blood cell count, liver and kidney function, cholesterol levels, blood sugar and insulin levels, thyroid tests, inflammation level, as well as reserve blood samples to be preserved for additional possible research tests. We will also plan to do tests to find out if you have any differences in genes that may be important for metabolism and body weight. In addition to looking at some genes we already think are important for body weight, we will use new DNA sequencing technology that will look at all the human genes we know about. This is known as exome and genome sequencing. This new technology allows us to look at DNA in great detail.
- 5. **Urine sample collection** to ensure that your kidneys work normally, that you are not taking any illicit drugs, and a pregnancy test (for women of childbearing age).
- 6. **Oral glucose tolerance test**. We will perform a test to study how your body handles sugar in the diet, called a 2-hour glucose tolerance test. You will drink a cup of sugar water and then will have your blood drawn over 2 hours to look at your blood sugar levels.
- 7. **Dual energy x-ray absorptiometry (DEXA)** to look at your body composition. The test involves lying still on a table while a small camera passes over your body. The dose of the x-ray is much less than the amount you would get from a normal chest x-ray. The total amount of time to do this test will be about 20-30 minutes.

#### Baseline Visit

PATIENT IDENTIFICATION

If you qualify for participation in the study, you will be scheduled for the baseline visit. We ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink except water that morning</u>. You will be seen on

**MEDICAL RECORD** 

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement. A questionnaire will also be performed.
- 2. **Fasting blood tests** to look at your baseline metabolic and inflammatory levels, as well as reserve blood samples to be preserved for additional possible research tests including a sample for future genetic analysis. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection.** We will obtain two stool samples to save for future experiments. As part of this collection, we will ask you to keep track of your diet for 24 hours on a form that will be provided to you, as diet can affect the results of the stool testing. You will also go over this "food record" in person with a nutritionist.
- 4. **Urine sample collection** as described before. We will also collect urine over your eight hours of testing to save for future experiments.
- 5. **Frequently sampled intravenous glucose tolerance test (FSIVGTT)**. This study tells us a lot about how sugar is used by your body, how well your insulin works, and how sensitive your body is to insulin. The FSIVGTT study is done while you rest in bed. A second IV line will be placed in your arm. We will give you some sugar water into one IV over a 2 minute period. We will then draw blood samples from the other IV at -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes (a total of 3 hours) to measure sugar and insulin levels. Exactly 20 minutes into the test, we will give you a small amount of insulin through the IV. A physician or nurse practitioner will be present during the first hour of the study. You can watch TV during this test.
- 6. **Computed Tomography (CT) Scan** of the abdomen to look at where you tend to store your fat. The test involves lying still on a movable table which passes through a large ring where the camera sits. The test does involve radiation, but because we only need to take a snapshot of your abdomen, the method that will be used minimizes your exposure. The total amount of time to do this test will be about 20-30 minutes.
- 7. **Subcutaneous Fat Biopsy**. To examine the level of certain molecules in your fat tissue, a small sample of fat tissue will be taken from under the skin of your abdomen. Lidocaine, a local anesthetic, is used to numb the area. A needle will be used to remove a piece of fat tissue measuring about 1 ½ teaspoons. A bandage is then applied to the site of needle insertion. We can give you some mild pain medication such as Tylenol, or stronger medication if needed, after the biopsy. The biopsy will be taken from a place on your body that is normally covered and not easily seen.
- 8. **Dispense Study Medication**. You will be given approximately an 8-week supply of colchicine to be taken two times a day (morning and late afternoon/evening) at home. Study medicine will be issued in a pill bottle with a "smart cap" that will record when you take your study medicine. The medication can be taken with or without food. We will give you a reminder alarm to help you remember when to take your medicine. If you forget to take a dose, then take it as soon as you remember. But if it is within 4 hours of the time for your next dose, do not take a double dose. Just skip the missed dose.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### **Short Outpatient Visit**

To make sure that you doing well taking the medication, you will be seen on a weekday in the Clinical Center at the National Institutes of Health. This visit will take about 2 hours to complete. We ask that you **bring your bottle of pills** with you. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.
- 2. **Fasting blood tests** to ensure that you are in good health, to examine your inflammation levels, as well as reserve blood samples to be preserved for additional possible research tests.
- 3. **Urine sample collection** as described before.
- 4. **Dispense Study Medication**. We will give you another bottle of colchicine and "smart cap" (about 8 weeks' worth) to last you until the Final (3 month) Visit. As before, if you forget to take a dose, then take it as soon as you remember. But if it is within 4 hours of the time for your next dose, do not take a double dose. Just skip the missed dose.

#### Final Visit

We will ask you to bring your bottle with any leftover pills to your final visit appointment. We ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink except water that morning</u>. You will be seen on a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.
- 2. **Fasting blood tests** as described before. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection** as described before.
- 4. **Urine sample collection** as described before.
- 5. Frequently sampled intravenous glucose tolerance test (FSIVGTT) as described before.
- 6. **DEXA Scan** as described before.
- 7. **CT Scan** as described before.
- 8. **Subcutaneous Fat Biopsy** as described before
- 9. **Exit questionnaire** to tell us about your experience of participating in our protocol.

#### **Optional Washout Visit**

PATIENT IDENTIFICATION

Because we would like to see if colchicine will continue to have lasting positive effects on your glucose regulation, metabolism, inflammation, and/or cardiovascular health even after you've stopped taking it, we invite patients to return to the NIH Clinical Center 3 months after finishing the study medication for repeat testing.

## MEDICAL RECORD MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

As before, we ask that you remain fasting for 10 hours before coming to the clinic and <u>have nothing to eat or drink</u> <u>except water that morning</u>. You will be seen on a weekday in the Clinical Center at the National Institutes of Health, and the visit will take about 8 hours to complete. During this visit we will perform the following:

- 1. **Interval medical history and physical exam,** with weight, height, and blood pressure measurement.
- 2. **Fasting blood tests** as described before. We will insert a small needle into your vein (an intravenous line or I.V.) in order to obtain blood samples.
- 3. **Stool sample collection** as described before.
- 4. **Urine sample collection** as described before.
- 5. **Frequently sampled intravenous glucose tolerance test (FSIVGTT)** as described before.
- 6. **DEXA Scan** as described before.
- 7. **CT Scan** as described before.
- 8. Subcutaneous Fat Biopsy as described before

When the study is complete, you will return to the care of your regular physician. Participation in this study does not commit NIH to your long term care.

#### Results of Tests at the NIH

We will be measuring many things in your blood during your visits, and it is possible we might uncover a medical problem that requires treatment. You will <u>not</u> be routinely provided treatment for any health condition discovered. However, you will be informed about such findings (e.g., high blood pressure) and any medically important information including blood tests or physical exam results will be forwarded to your primary care physician at your request. Some of these medical problems might prevent you from participating further in the study.

#### **Risks and discomforts**

- 1. **Physical examination**. A physician or a nurse practitioner may need to examine you with your clothes off, with appropriate precautions to protect your privacy. Some may find this examination embarrassing.
- 2. **Radiation Exposure**: This research study involves exposure to radiation from three DEXA scans and three CT scans. Please note that this radiation exposure is not necessary for your medical care and is for research purposes only. The NIH Radiation Safety Committee has reviewed the use of radiation in this research study and has approved this use as involving minimal risk and necessary to obtain the research information desired.

Although each organ will receive a different dose, the amount of radiation exposure you will receive yearly from this study is equal to a uniform whole-body exposure of 0.093 rem. This calculated value is known as the "effective dose" and is used to relate the dose received by each organ to a single value. The amount of radiation you will receive in this study is below the dose guideline established by the NIH Radiation Safety Committee for research subjects. This guideline is an effective dose of 5 rem received per year.

For comparison, the average person in the United States receives a radiation exposure of 0.3 rem per year from natural background sources, such as from the sun, outer space, and from radioactive materials that are found naturally in the earth's air and soil. If you would like more information about radiation and examples of exposure levels form the other sources, please ask the investigator for a copy of the pamphlet called, <u>An Introduction to Radiation for NIH Research Subjects.</u>

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

3. **Blood withdrawal**. The blood withdrawal amount is well below the NIH guideline for a safe amount of blood withdrawal (550 cc every 8 weeks). A small bruise may form at any site where the blood is taken. The risk of infection or fainting is very small. Inflammation or clotting of a vein also may rarely occur.

Some of your blood will be sent to another laboratory within the NIH to examine your inflammation levels. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.

- 4. **Stool sample collection** has no risk, and should only take a moment to complete. The samples will be coded, and only the investigators from this study will have access to the identity of the samples.
- 5. **Urine sample collection** has no risk and should only take a moment to complete. If you do test positive for an illicit substance, the result will be part of your NIH Medical Record.
- 6. **Questionnaires** are not risky, but may be inconvenient because of the time necessary to complete them.
- 7. **Oral glucose tolerance test.** This test is inconvenient because of the time it takes to complete. The only risks from this kind of study are those described for any blood draw, as well as developing nausea from the oral glucose. Patients may transiently develop high blood sugar levels from the glucose, but it should normalize within a few hours and should not be clinically significant.
- 8. **Intravenous glucose tolerance test.** This test is inconvenient because of the time it takes to complete. You can watch TV during this test. The only risks from these kinds of studies are those described for any blood draw, the possibility of slight arm tenderness in the arm receiving the sugar infusion, (this tenderness goes away within a few minutes with gentle rubbing of the arm), and the possibility of a low blood sugar during the study. With slightly low blood sugars (less than 50 mg/dL), participants may get hungry, have a headache, feel shaky or dizzy, may become drowsy, or may become sweaty. With very low blood sugars (under 30 mg/dL) participants may have trouble speaking, be difficult to arouse, and even have seizures. However, in the test we are doing, we will be giving you extra sugar to raise your blood sugar above normal, and then we will try to bring it back to normal (95-105 mg/dL) with insulin. To do this, we will measure blood sugar at 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, and 180 minutes (a total of 3 hours). A physician or nurse practitioner will be present during the first hour of your test to make sure everything is working properly. We expect that the chance of even a slightly low blood sugar is very low. If a low blood sugar does not come up on its own quickly, the test will be stopped and you will be given sugar by vein to raise the blood sugar to normal.
- 9. **Fat tissue biopsies.** Possible side effects of the biopsy procedure are pain during and for two to three days after the procedure, although rarely the biopsy site may be tender or sore or have bruising or swelling for 2-3 weeks. Biopsy wounds usually heal with a very small, nearly unnoticeable scar, but sometimes a raised scar (keloid) or visible lump may result. Your risk is slightly higher if you are African American. Lidocaine injection for numbing before fat biopsies may cause some mild burning before the numbing takes effect. Rare adverse effects include infection at the biopsy sites or an allergic reaction to Lidocaine that may lead to a rash and/or swelling of the injected area. If you know you are allergic to Lidocaine, we will change to another local anesthetic. Another risk of the procedure is minor bleeding in the area of the biopsy. Some medications may increase the amount of bleeding from the biopsy. If you are taking medications such as Coumadin, Plavix or aspirin to thin your blood, you WILL NOT have a biopsy. If you are taking aspirin or non-steroidal medications such as Advil for pain you will need to stop taking these medicines for one week before the biopsy is performed.
- 10. **Smart cap** has no risk and should work no differently than a regular pill bottle cap.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

11. Medication. The most common adverse effects from the medication used in this study are nausea, vomiting, diarrhea, and abdominal pain. Some rare side effects (< 1%) have been reported including decreased production of red cells (which could make you feel tired), white blood cells (which can make more susceptible to infections), and/or platelets (which may make you more susceptible to bruising or bleeding), tingling (neuropathy), dizziness, muscle pain or weakness, rash, allergic reaction, decreased sperm count, and increased liver enzyme levels. These symptoms usually occur in people with underlying medical problems, or were on certain medications, that predisposed them to having the reaction. In general, these symptoms resolved within a week once the medication was stopped. Although colchicine has been used for about 2000 years for gout, as with any medication, there is always the possibility of unpredicted side effects. We will monitor you for all adverse effects. If (severe) adverse effects develop, we will decrease the dose, temporarily stop, or discontinue the medication.</p>

If you experience any of the following, contact our team right away:

- Muscle weakness or pain
- Numbness or tingling in the fingers or toes
- Unusual bleeding or bruising
- Severe diarrhea or vomiting

There are no adequate well-controlled studies on the use of colchicine in pregnancy. Data from a limited number of published studies found no evidence of an increased risk of miscarriage, stillbirth, or teratogenic effects among pregnant women using colchicine. However, colchicine did demonstrate birth defects in the offspring of pregnant rats. If you think you might become pregnant, we will ask that you not participate in this study.

- Taking certain medicines with colchicine can cause your level of colchicine to be too high, especially if you have kidney or liver problems (refer to "Medication Guide" for more information).
- Even medicines that you take for a short period of time, such as antibiotics, can interact with colchicine and cause serious side effects or death. Please tell us about any new medicine you need to take so we can make sure you can continue using colchicine.
- Avoid drinking grapefruit juice, as it can interfere with your body's ability to breakdown colchicine.

#### Keep the medication out of the reach of children.

- 12. **DNA testing.** If you allow us to study your DNA, we will use it for genome sequencing. Genome sequencing is a test that could give us different kinds of results. These include:
  - a. We could identify changes in genes that are related to metabolism and body weight.
  - b. We could identify changes in genes that contribute to other diseases or problems.
  - c. We could identify changes in genes that are not known to cause any disease. These are known as normal variations.
  - d. We could find changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

Not all gene changes will have health implications for your family. Changes in genes that have health implications for your family:

- 1. May have already caused health problems.
- 2. May cause a health problem in the future.

PATIENT IDENTIFICATION

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

One of the goals of this study is to identify changes in genes that may be involved in obesity. This research may take years. If however we identify a genetic cause or likely cause of obesity, with your permission, we will contact you. Please let us know your preference by initialing one of these two statements:

| I would like to be contacted with information about the progress of this study and contacted about any results related to obesity. I understand that this research will take years and that a specific abnormality might not be identified in me. |
|---|
| Please do not contact me regarding the progress of this study or any specific gene changes related to obesity. |

а

If we detect a genetic change that might be important for you, then we will have to confirm this result in a certified laboratory. For this confirmation, we will ask for a new sample of DNA from you. In most cases this will involve obtaining a small sample of blood (1-2 teaspoons). In some cases we can obtain enough DNA to confirm a genetic change by swabbing the inside of the cheek. You can decide whether you want to do that later, if we contact you with the information that we have found a possible important genetic difference.

Identifying gene changes that are not related to the condition being studied is known as <u>incidental medical</u> information.

We will find gene changes in everyone that we study, but we are only specifically looking for genes related to metabolism and body weight. We will not analyze your DNA for changes that are not related to metabolism and body weight. Even so, some gene changes not related to metabolism and body weight will be detected.

We will only inform you only of changes that have urgent medical significance and would benefit from early medical treatment. An example of this would be a gene change that causes cancer and where you would benefit from early screening. We will not inform you of all gene changes that have uncertain health implications. For example we will not report gene changes that only predispose individuals to disease. An example of this would be a gene change that influences the risk of heart disease, but where the development of the disease is dependent on many genetic and non-genetic (such as diet and smoking) factors. If we find a change in a gene that is important to your family's health, we will only be able to give you those results if the change has been confirmed in a certified laboratory. To make sure an error has not occurred, we would need to obtain a new sample of DNA from you to confirm the experimental results.

In addition to knowing what we could find, we would like you to know the limitations of the genome sequencing and what we will NOT be able to tell you about the changes that we find.

**1.** Not all gene changes that cause disease will be detected.

PATIENT IDENTIFICATION

- **2.** Some changes that are not currently known to cause health problems will be found to cause health problems in the future. We cannot promise to be able to tell you about those changes in the future.
- **3.** We will not tell you about gene changes that are not known to have health implications, nor will we tell you about gene changes that have only reproductive consequences.
- **4.** This gene sequencing cannot be substituted for diagnostic testing recommended by another physician.

Please initial all of the following statements to indicate that you understand the extent to which we will inform you about incidental genetic changes that we find:

#### **CONTINUATION SHEET for either: MEDICAL RECORD**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

| STUDY NUMBER: | 14-CH-0119 | CONTINUATION: pages |
|---|---|---|
| | I understand that I will be informed only of genetic changes that researchers study feel are urgently important for my family's health and that knowledge o the potential to provide a significant benefit for me or my family. | |
| _ | metabolism and body | stigators will not specifically look for gene changes not related to weight, and that identification of other disease-causing genes will only nding on the analysis being done. |
| | | even though they could have health or reproductive consequences, I will enetic changes identified that are not related to metabolism and body |
| requiremen<br>will be give<br>contacted a<br>a gene cha<br>of this wou | ts of having urgent medical<br>n a choice to learn or not le<br>t all if that is your preference<br>nge would be a gene chang<br>d be a gene change that ha<br>yould be beneficial. Before o | I to metabolism and body weight and the investigators feel it meets the significance so that you would benefit from medical treatment, then you can about a genetic change that we find. You can chose not to be ce. An exception to your ability to choose whether or not to find out about e that investigators feel is of critical importance to your health. An example as a high probability of causing cancer or a disease for which early confirming the result in a clinical laboratory we will contact you to obtain a |
| one member<br>could be a<br>promise to | er of your family. We will dis<br>carrier for this same change | thealth implications, the NIH will confirm the genetic change present in scuss the results with you so that you understand who else in your family e. We can help arrange for this testing to be done, but the NIH cannot cal testing necessary to confirm or determine who else in your family may |
| | medical follow up. The NIH | will discuss the results with you and make recommendations regarding I cannot promise to perform or pay for recommended medical tests or |
| T1 | | |

It is possible that a gene change will not be confirmed on subsequent testing. This could be due to an error in the DNA sequencing or an error in processing the DNA or cell lines. Although you likely will be glad that we did not confirm a problem, this may cause some anxiety and concern that you otherwise would not have experienced.

Please let us know your preferences by initialing one of the following statements:

| <br>_ I DO want to be re-contacted if genetic variants with urgent health implications are discovered during this research testing. |
|---|
| _ I DO NOT want to be re-contacted if genetic variants with urgent health implications are |
| discovered during this research testing. I understand that an exception to this choice, as |
| described above, will be made for a gene change of critical medical significance. |

**Emotional and psychological risks from DNA testing.** Identification of gene changes could cause emotional and psychological problems. In some situations psychological counseling could be recommended.

1. Learning about disease risk in your family can be distressing.

**PATIENT IDENTIFICATION** 

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

2. Learning that you passed on a gene that does not work to your child can be distressing.

3. Other members of your family could be upset to learn that they may be at risk for a disorder because of your participation in this study.

You may be falsely reassured about your health status if we do not report any changes to you.

**Other risks of genetic testing.** If we confirm a gene change in your DNA in a diagnostic laboratory, this information will become part of your medical record at the NIH. Some people are concerned that information about them from their medical records could be released. Possible problems include insurance or employment discrimination. Measures to protect the confidentiality of your information are described below. These problems may also occur if you disclose information yourself or agree to have your research records released.

There are state and federal laws that protect against genetic discrimination. A federal law called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. According to this law, health insurance companies or group health plans (as of May 21, 2010) cannot request your genetic information or use it to make decisions about your eligibility or premiums; and employers cannot use it in deciding to hire, promote, or fire you or in setting the terms of your employment (as of Nov 21, 2009).

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

The following link contains details on this policy: http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf

You may ask your research team for additional information or a copy of The Genetic Information Nondiscrimination Act of 2008 informational document.

Genetic studies can uncover unexpected family relationships. For example, it is possible that we might learn that a family member is not the biological child of the parents with whom she or he lives (for example, because of adoption). We will not ordinarily provide this type of information to any member of the family or to the referring physician. However, we may make exceptions under extraordinary circumstances if this information were required for the medical care of the individuals involved. If we are convinced this is necessary, we will provide the information to the physician providing medical care to the patient.

#### **Use of stored samples and data**

**Future DNA Research.** Currently we plan to sequence known genes. This represents only about 1% of your DNA sequence. In the future we may sequence other parts of your DNA, and eventually, we may completely sequence your DNA. These additional studies may occur years from now. Some of your DNA may be sent to other laboratories for specific tests. If this is done DNA will be coded and not have your name on the sample or the paperwork that goes to the laboratory. Should you withdraw from this study, we will keep your DNA for analysis unless you ask us to destroy the DNA samples.

Please initial one of the following three statements regarding future research:

\_\_\_\_\_ DNA can be used for other kinds of future health-related research. This research is not limited to studies related to obesity, metabolism and body weight. This testing may be done by research laboratories that

#### **MEDICAL RECORD**

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

| are not at the NIH. I authorize use of these samples without my additional consent. I understand I will not be contacted if these samples are used in the future. |
|---|
| I understand that genetic samples collected during these NIH visits will be saved and used for future experimental testing related to obesity, metabolism, and body weight. This testing may be done by research laboratories that are not at the NIH. I do NOT authorize use of these samples for any other purpose without my additional consent. I must be contacted and give consent if these samples are to be used in the future. |
| Do not use my DNA for any future studies beyond those described above in this consent form. |
| <b>Future research with blood samples.</b> Our specific research plans have been summarized in this consent form. In the course of the research, we will obtain blood samples. While we can do some of our tests immediately, we may want to store your blood samples in the freezer for future studies. In addition, certain information will be stored in your medical record. In the future, it is possible that your blood samples or medical records will be used for other research purposes that are not specifically outlined in this consent form. If this is done, samples will be coded, and you will not be identified by name. These samples may be stored at a separate site (called a repository) that specializes in storing clinical samples. You have the option, in the future, of requesting that these samples not be used for any additional testing. In addition, it is possible that some information obtained from these studies will be published in the medical literature. However, your identity will not be included in any publications. |
| Please initial <u>one</u> of the following two statements: |
| I understand that samples collected during these NIH visits will be saved and used for future experimental testing related to body weight, and/or metabolism. This testing may be done by research laboratories that are not at the NIH. I authorize other uses of these samples without my additional consent. I understand I will not be contacted if these samples are used in the future. |
| I understand that samples collected during these NIH visits will be saved and used for future experimental testing related to body weight, and/or metabolism. This testing may be done by research laboratories that are not at the NIH. I do NOT authorize any other use of these samples without my additional consent. I must be contacted and give consent if these samples are to be used in the future. |
| All through the process of the study and afterwards, the confidentiality of participants will be protected by using codes and medical record numbers in recording your information and test results. Only medical personnel involved in this study will have access to participants' names, test results, and patient code numbers. |
| You need to be aware that DNA sequence is like a fingerprint. Theoretically if enough DNA sequence information is available, someone could identify you based on his/her DNA sequence. To facilitate genetic research, your DNA sequence information may be deposited in other databases. In this case, unless we have your permission, we will deposit the data in a manner that would not allow someone to identify you. Please understand that this information cannot be removed once it is deposited. |
| Please initial one of the following boxes. |
| I do not want DNA sequence data to be deposited in any database other than the one associated with this study. |

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study CONTINUATION:  pages My DNA sequence data can be deposited in databases that limit access to IRB (ethics board) approved-researchers. My DNA sequence can be deposited in a database that is available only to scientists but that does not require IRB approval of research studies. I understand that someone could theoretically identify me from this information.

#### Potential benefits of participation

We are hopeful that your participation in this study will provide evidence as to whether colchicine will help metabolic parameters in obese individuals. However, you might not benefit directly from participating in this study. Should we find abnormalities in any of your test results, you will be notified and receive a copy to assist you in seeking further medical evaluation. This information may or may not improve your health.

#### Right of Withdrawal and Conditions for Early Withdrawal

You may withdraw from the study at any time and for any reason without loss of benefits or privileges to which you are otherwise entitled.

#### **Discussion of New Findings with You**

After all participants have completed the study, we will inform you about which medicine you took and, once the study is fully analyzed, let you know if colchicine seemed to help with inflammation and insulin resistance. There is no general plan to share your individual test results with you. However, if any findings suggest you have a medical issue, we will provide this information to you and your primary care provider. You may request a copy of your routine laboratory tests if you desire.

#### **Study Termination**

You may be asked to end your participation in this study at any time if we believe that continuation is not in your best medical interest or if you are unable to comply with the requirements of the study.

#### **Alternatives to Participation**

PATIENT IDENTIFICATION

The alternative to this study is not to participate. You may be eligible for other studies in the NIH. You may learn more about them through <a href="https://www.clinicaltrials.gov">www.clinicaltrials.gov</a>.

#### **Compensation**

You will be compensated for the time and inconvenience associated with participation according to NIH research volunteer guidelines. Compensation for completing all of the testing described above is \$100 for the outpatient screening visit, \$50 for the safety visit, and \$300 each for the baseline, final, and washout visits. The total amount you could receive for participation if you complete all parts of this study is \$1050.

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### **Conflict of Interest**

The NIH and members of this research team have no financial interest related to this research study.

#### Posting of Research Results on www.ClinicalTrials.gov

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

| I have received a | CODY | of the | cianod | concont | form |
|-------------------|--------|---------|--------|----------|--------|
| I nave received a | і сору | or trie | signed | COHSCHIL | 101111 |

#### **MEDICAL RECORD**

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

Adult Patient or Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### OTHER PERTINENT INFORMATION

**1. Confidentiality.** When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- **2. Policy Regarding Research-Related Injuries.** The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH quidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Jack A. Yanovski, MD, PhD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686 or Associate Investigator Andrew Demidowich, MD; Building 10-CRC Room 1-3330, Telephone: 301-496-4686.

You may also call the Clinical Center Patient Representative at 301-496-2626.

**5. Consent Document.** Please keep a copy of this document in case you want to read it again.

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | |
|---|---|---|
| A. Adult Patient's Consent I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby consent to take part in this study. | <b>B. Parent's Permission for Minor Patient.</b> I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby give permission for my child to take part in this study. (Attach NIH 2514-2, Minor's Assent, if applicable.) | |
| Signature of Adult Patient/Legal Representative Date | Signature of Parent(s)/Guardian | Date |
| Print Name | Print Name | |
| C. Child's Verbal Assent (If Applicable) The information in the above consent was described to my child and my child agrees to participate in the study. | | |
| Signature of Parent(s)/Guardian Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM JANUARY 24, 2018 THROUGH FEBRUARY 24, 2019. Signature of Investigator Date Signature of Witness Date | | |
| Print Name | Print Name | |

#### **PATIENT IDENTIFICATION**

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

**MEDICAL RECORD** 

• Adult Patient or • Parent, for Minor Patient

INSTITUTE: Instituto Nacional de Salud Infantil y Desarrollo Humano (National Institute of Child Health and

Human Development)

STUDY NUMBER: 14-CH-0119 PRINCIPAL INVESTIGATOR: Jack Yanovski, M.D.

STUDY TITLE: Estudio preliminario de los efectos de la colchicina en adultos no diabéticos con síndrome

metabólico

(Pilot Study of the Effects of Colchicine in Non-Diabetic Adults with Metabolic Syndrome)

Continuing Review Approved by the IRB on 01/24/18

Amendment Approved by the IRB on 07/13/18 (S)

Date Posted to Web: 08/07/18

Open-Label Arm Spanish

#### **INTRODUCCIÓN**

Deseamos invitarle a participar en un estudio de investigación en los Institutos Nacionales de Salud (*National Institutes of Health, NIH*).

En primer lugar, queremos que Ud. sepa que:

La participación en una investigación del NIH es totalmente voluntaria.

Usted puede decidir no participar o retirarse del estudio en cualquier momento. En cualquier caso, no perderá ninguna compensación a la que pueda tener derecho. No obstante, para recibir atención médica en el NIH usted debe participar en un estudio o estar en evaluación para participar en uno.

Es posible que no reciba ningún beneficio por su participación. Con la investigación podemos adquirir conocimientos que ayuden a otras personas en el futuro.

En segundo lugar, algunas personas pueden tener creencias personales, religiosas o éticas que limiten los tipos de tratamientos médicos o de investigación que deseen recibir (por ejemplo, transfusiones de sangre). Si usted es una de esas personas, hable al respecto con sus médicos o con el equipo de investigación del NIH antes de acceder a participar en el estudio.

El estudio se describe en las siguientes páginas. Antes de decidir participar, tómese todo el tiempo que necesite para hacer preguntas y hablar del estudio con cualquier persona del NIH, o con su familia, amigos, médico personal o cualquier otro profesional de la salud.

#### Propósito de este Estudio

Aproximadamente 30% de los adultos en los EE.UU. tienen un índice de masa corporal (IMC) superior a 30 (kg/m2), y están en mayor riesgo de una serie de problemas médicos, incluyendo la presión arterial alta, colesterol alto en la sangre, niveles altos de triglicéridos, azúcar en la sangre (diabetes) y enfermedades del corazón. Se cree que tener sobrepeso, puede llevar a un estado de inflamación aunque de nivel bajo, y que esta inflamación puede conducir a algunos de los problemas médicos asociados con la obesidad. El propósito de este estudio es investigar si un medicamento llamado colchicine puede mejorar el metabolismo de los adultos que tienen complicaciones médicas debido a su sobrepeso corporal (estas complicaciones son algunas veces llamadas, "síndrome metabólico"), y han desarrollado altos niveles de azúcar en la sangre (diabetes).

#### **PATIENT IDENTIFICATION**

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (6)
**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Colchicine es una medicación anti- inflamatoria que se ha utilizado durante siglos en el tratamiento de la gota. A partir de estudios en animales y estudios en humanos, existe alguna evidencia de que los medicamentos anti-inflamatorios como colchicine pueden mejorar la capacidad del páncreas para secretar insulina y la capacidad del cuerpo para regular el azúcar. Les pedimos que se unan a nuestro estudio, por el cual esperamos averiguar si colchicine puede mejorar la regulación del azúcar y los parámetros metabólicos.

Si califica y está de acuerdo en participar, Ud. será una de siete personas asignadas al azar para tomar tabletas de colchicine por vía oral, dos veces al día durante 3 meses. Las tabletas de colchicine vendrán en la misma dosis que está disponible en las farmacias y se prescribe para una enfermedad llamada "gota": 0.6 miligramos.

Cuando se haya completado el estudio, le enviaremos cada uno de los participantes información sobre los resultados y les daremos a conocer si la medicación se ayudan.

Los participantes del estudio tendrán que venir al Centro Clínico del NIH para cuatro consultas ambulatorias, con una quinta consulta ambulatoria opcional. Es importante que los participantes llegen en ayunas (sin alimentos ni bebidas aparte de agua) a cada una de estas visitas. Los participantes serán compensados por su tiempo y cualquier inconveniente (ver más abajo: Compensación en la página 5).

#### Población de estudio

PATIENT IDENTIFICATION

Deseamos reclutar a siete adultos con sobrepeso y diabetes, controlada exclusivamente con dieta.

#### Quién puede participar en este estudio

Usted puede ser elegible para este estudio de investigación si es mayor de 18 años de edad; si tiene un índice de masa corporal mínimo de 30, el cual se calcula dividiendo el peso del individuo en kilogramos, por su altura en metros, al cuadrado, (Kg/m2); pesar menos de 450 libras, y que se encuentre en buen estado de salud general. Usted también tiene que cumplir con ciertos niveles de resistencia a la insulina y a la inflamación, medidas por pruebas de laboratorio, y tener diabetes tipo 2 controlada con dieta para participar en todo el estudio. Si usted es una mujer en edad de procrear, se le pedirá que use un método efectivo de control de la natalidad antes de participar en este studio.

#### Quienes no pueden participar en este estudio

Usted no puede ser elegible para este estudio si tiene una enfermedad médica grave que pudiera interferir con las pruebas o mediciones del estudio, como enfermedades del corazón, riñón, hígado, pulmón, sangre, intestinal o enfermedades endocrinas o presión arterial alta no controlada. Si usted está usando un medicamento que afecta el metabolismo del azúcar y la grasa o la absorción en su cuerpo, o un medicamento que no se debe tomar con colchicine, es posible que no sea elegible para participar. Tampoco son elegibles las mujeres que están embarazadas o lactando, o tienen intención de quedar embarazadas; las personas que han tenido un cambio de peso reciente superior al 3% del peso corporal total, han estado utilizando medicamentos para reducir el peso, han usado recientemente la colchicina, tener una alergia conocida a la colchicina, o utilizan productos de tabaco o nicotina (p. ej. e-cigarrillos), no serán reclutadas para este estudio. Se recomienda a las personas con antecedentes de formación de queloides (que fácilmente desarrollan cicatrices en su piel después de una lesión) no participar en este estudio.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

# Procedimientos del estudio

El estudio consta de cuatro visitas ambulatorias en el Centro Clínico: **una visita para determinar elegibilidad, una visita inicial** para estudiar su metabolismo antes de la participación, **una corta visita ambulatoria** para comprobar cómo se siente el participante durante el estudio, y **una visita final** 3 meses después de la visita inicial para ver los cambios después de la participación. Al término de la visita final, usted tiene la opción de volver 3 meses después para otra visita en la cual se quiere ver si los cambios observados mientras la participación en el estudiopermanecen incluso después de suspender la medicación del estudio. Se le dará la medicación del estudio (colchicina) en el día de completar la Visita Inicial.

#### Visita Ambulatoria de Selección de Pacientes

Esta visita tomará unas 3 horas para realizarse. Usted será visto en un día de semana en el Centro Clínico del NIH. Le pedimos permanecer en ayunas durante las 10 horas anteriores a su llegada a la clínica y no debe comer o beber nada, excepto aqua por la mañana. Durante esta visita, vamos a realizar lo siguiente:

- 1. **Protocolo y firma del formulario de consentimiento**. Vamos a repasar el estudio en detalle y a responder cualquier pregunta. El formulario de consentimiento debe ser firmado antes de poder tomar parte en el estudio.
- 2. Historia médica completa y un examen físico, con el peso, la altura, y la medición de la presión arterial.
- 3. Un **ECG** se realizará para examinar la función de su corazón.
- 4. Los análisis de sangre en ayunas para asegurarse de que usted se encuentra en buen estado de salud. El análisis examinará el recuento de células de la sangre, función hepática y renal, niveles de colesterol, los niveles de azúcar e insulina en sangre, pruebas de función tiroidea, nivel de la inflamación, así como muestras de sangre de reserva para ser preservadas para poder examinar durante futuras investigaciónes. También realizaremos pruebas para determinar si usted tiene alguna diferencia en genes que pueden ser importantes para el metabolismo y el peso corporal. Además para buscar algunos genes que ya nosotros pensamos que son importantes para el peso corporal, vamos a utilizar nueva tecnología de secuenciación de DNA que se verá en todos los genes humanos que conocemos. Esto se conoce como "exome" y secuenciación del genoma. Esta nueva tecnología nos permite mirar el ADN en gran detalle.
- 5. **Recogida de muestras de orina** para asegurarse de que sus riñones funcionan normalmente, que no está tomando cualquier droga ilícita, y una prueba de embarazo (para las mujeres en edad fértil).
- 6. **Prueba de tolerancia a la glucosa oral**. Vamos a realizar una prueba para examinar si usted tiene diabetes, la llamamos prueba de tolerancia a la glucosa de 2 horas. Va a tomar una taza de agua con azúcar y luego se tomarán muestras 1 y 2 horas después para mirar su nivel de azúcar en la sangre.
- 7. **Absorciometría dual de rayos X (DEXA)** para examinar su composición corporal. La prueba consiste en permanecer inmóvil sobre una mesa mientras una pequeña cámara pasa sobre su cuerpo. La dosis de los rayos X es mucho menor que la cantidad que se obtiene de una radiografía de pecho normal. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos.

MEDICAL RECORD

PATIENT IDENTIFICATION

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

## Visita Inicial

Si reúne los requisitos para participar en el estudio, se le cita para la visita inicial. Le pediremos que permanezca en ayunas durante 10 horas antes de llegar a la clínica y no comer o beber nada, excepto agua por la mañana. Usted será visto en un dia entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita tomará alrededor de 8 horas para completarse. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo de historia clínica **y examen físico**, con el peso, la altura, y la medición de la presión arterial. También se completará un cuestionario.
- 2. **Los análisis de sangre en ayunas** para mirar su metabolismo basal y los niveles inflamatorios, así como muestras de sangre de reserva para ser preservados para las pruebas de investigación adicionales posibles, incluyendo una muestra para futuro análisis genético. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener las muestras de sangre.
- 3. Obtención **de muestras de heces**, obtendremos dos muestras de heces para conservar para futuros experimentos. Como parte de esta colección, le pediremos que mantenga un record de su dieta por 24 horas en un formulario que se le entregara a usted, y asi ver como la dieta puede afectar los resultados de las pruebas de heces. Los resultados de este "diario de nutricion" irá con un nutricionista.
- 4. Obtención **de muestras de orina** como se describe antes. También vamos a recoger la orina durante su visita a ahorrar para futuros experimentos.
- 5. **Prueba de tolerancia a la glucosa intravenosa muestreado frecuentes**. Este estudio nos dice mucho acerca de cómo su cuerpo utiliza el azúcar, qué tan bien está funcionando su insulina y cómo es la sensibilidad de su cuerpo a la insulina. El estudio FSIVGTT se hace mientras usted descansa en una cama. Una segunda línea IV se coloca en su brazo. Le daremos un poco de agua de azúcar en una vía intravenosa durante un período de 2 minutos. Entonces vamos a tomar muestras de sangre de la otra IV en -15, -10, -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, y 180 minutos (un total de 3 horas ) para medir los niveles de azúcar e insulina . Exactamente a los 20 minutos en la prueba, le daremos una pequeña cantidad de insulina a través de la IV. Un médico o enfermera practicante estará presente durante la primera hora del estudio. Usted puede ver la televisión durante esta prueba.
- 6. **Tomografía Computarizada (TC) del abdomen** para observar donde se tiende a almacenar su grasa. La prueba consiste en permanecer quieto en una mesa móvil que pasa por un gran anillo donde esta ubicada la cámara. La prueba implica radiación, pero solo porque tomaremos una foto de su abdomen, el método que se utilizará minimiza su exposición. La cantidad total de tiempo para realizar esta prueba será de unos 20 a 30 minutos
- 7. **Subcutánea Biopsia de grasa**. Para examinar el nivel de ciertas moléculas en el tejido graso, se tomará una pequeña muestra de tejido graso de debajo de la piel de su abdomen. Para adormecer el área donde se tomarà la muestra, se utilizará la lidocaína, un anestésico local. Una aguja se utilizará para extraer una porción de tejido graso que mide alrededor de 1 ½ cucharaditas. Un vendaje se aplica entonces al sitio de inserción de la aguja. Podemos darle algún medicamento para el leve dolor, como Tylenol o medicamento más fuerte si es necesario, después de la biopsia. La biopsia se tomará de un lugar del cuerpo que normalmente está cubierto y que no se

MEDICAL RECORD

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

ve fácilmente.

8. Los medicamentos de dispensación de Estudio. Se le dará un suministro de aproximadamente 8 semanas de la medicación del estudio para ser tomado dos veces al día (mañana y tarde/noche) en casa. El medicamento del estudio estará en un frasco de tabletas con una "tapa inteligente" que registrará cuando se toma el medicamento de estudio. El medicamento se puede tomar con o sin alimentos. Le daremos una alarma de recordatorio para ayudarle a recordar cuándo tomar su medicamento. Si se olvida de tomar una dosis, tómela tan pronto como lo recuerde. Pero si está dentro de las 4 horas de la hora de su siguiente dosis, no tome una dosis doble. Sólo tome la dosis olvidada.

#### Visita Ambulatoria Corta

Para asegurarse de que está tomando bien el medicamento, usted será visto en un día de la semana en el Centro Clínico de los Institutos Nacionales de Salud. Esta visita se tomara alrededor de 2 horas en completarse. Le pedimos que traiga su botella de píldoras con usted. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo de historia clínica y examen físico, con el peso, la altura, y la medición de la presión arterial.
- Análisis de sangre en ayunas, para asegurarse de que está en buen estado de salud, para examinar sus niveles de inflamación, así como muestras de sangre de reserva para ser preservado para las pruebas adicionales futuras.
- 3. **Recogida de muestras de orina** como se describe antes.
- 4. **Los medicamentos de dispensación de Estudio**. Le daremos otra botella de la medicación del estudio con "tapa inteligente" (para un periodo de cerca de 8 semanas) para que le dure hasta la visita final (3 meses). Al igual que antes, si olvida tomar una dosis, tómela tan pronto como lo recuerde. Pero si está dentro de las 4 horas de la hora de su siguiente dosis, no tome una dosis doble. Omita la dosis olvidada.

#### Visita Final

Le pediremos traer su botella con pastillas sobrantes de su anterior visita. Le pedimos permanecer en ayunas durante 10 horas antes de llegar a la clínica y <u>no comer o beber nada excepto agua por la mañana</u>. Usted será visto en un día entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita se llevará alrededor de 8 horas para completar. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo historia clínica y examen físico, con el peso, la altura, y la medición de la presión arterial
- 2. **Análisis de sangre** en ayuno como se describe anteriormente. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener muestras de sangre.
- 3. Recogida de muestras de heces como se describe antes.
- 4. **Recogida de muestras de orina** tal como se describe antes.
- 5. Prueba muestreado frecuentes tolerancia a la glucosa intravenosa (FSIVGTT) como se describe antes.
- 6. **DEXA Scan** como se describe antes.
- 7. **CT Scan** como se describe antes

PATIENT IDENTIFICATION

- 8. **Grasa subcutánea biopsia** como se ha descrito antes
- 9. **Cuestionario final** para contarnos acerca de su experiencia de participar en nuestro protocolo.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### Visita Opcional

Debido a que nos gustaría ver si la colchicina seguirá teniendo efectos positivos duraderos en la regulación del metabolismo de su glucosa, la inflamación, y/o su salud cardiovascular, incluso después de haber dejado de tomarlo, invitamos a los pacientes a volver al Centro Clínico de los NIH 3 meses después de terminar la medicación del estudio para repetir las mismas pruebas.

Al igual que antes, le pedimos que permanecer en ayunas durante 10 horas antes de llegar a la clínica y <u>no comer o beber nada, excepto agua por la mañana</u>. Usted será visto en un día entre semana en el Centro Clínico de los Institutos Nacionales de Salud, y la visita llevará alrededor de 8 horas para completarse. Durante esta visita vamos a realizar lo siguiente:

- 1. Intervalo historia clínica y examen físico, con el peso, la altura, y la medición de la presión arterial
- 2. **Análisis de sangre e**l ayuno como se describe anteriormente. Vamos a insertar una pequeña aguja en la vena (una vía intravenosa o IV) con el fin de obtener muestras de sangre.
- 3. **Recogida de muestras de heces** como se describe antes.
- 4. Recogida de muestras de orina tal como se describe antes.
- Prueba muestreado frecuente de tolerancia a la glucosa intravenosa (FSIVGTT) como se describe antes.
- 6. **DEXA Scan** como se describe antes.
- 7. **CT Scan** como se describe antes.
- 8. Grasa subcutánea biopsia como se ha descrito antes

Cuando el estudio se haya completado, volverá al cuidado de su médico de cabecera. La participación en este estudio no compromete al NIH a su cuidado a largo plazo.

#### Los resultados de pruebas realizadas en el NIH

Estaremos midiendo muchas cosas en su sangre durante sus visitas, y podríamos descubrir algún problema médico que requiere tratamiento. Ud. no recibirá de forma rutinaria tratamiento para cualquier condición de salud descubierto. Sin embargo, se le informará sobre estos hallazgos (por ejemplo: presión arterial alta) y cualquier información de importancia médica que resulten de análisis de sangre o del examen físico, serán remitidos a su médico de atención primaria en su solicitud. Algunos de estos problemas médicos podrían impedir su participación más en el estudio.

#### Riesgos y molestias

- 1. **El examen físico**. Un médico o una enfermera puede tener que le examinar pidiéndole que se quite su ropa, con las precauciones adecuadas para proteger su privacidad. Algunos pueden encontrar este examen vergonzoso.
- 2. **Exposición a la radiación**: Este estudio de investigación implica la exposición a la radiación de tres imagenes DEXA y tres tomografías computarizadas. Tenga en cuenta que esta exposición a la radiación no es necesario para su atención médica y es sólo para fines de investigación. El Comité de Seguridad Radiológica NIH ha revisado el uso de la radiación en este estudio de investigación y ha aprobado este uso ya que implica un riesgo mínimo y necesario para obtener la información de investigación deseada.

PATIENT IDENTIFICATION

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Aunque cada órgano recibirá una dosis diferente, la cantidad de exposición a la radiación que recibirá anualmente de este estudio es igual a una exposición uniforme de todo el cuerpo a 0.093 rem. Este valor calculado se conoce como la "dosis efectiva" y se utiliza para relacionar la dosis recibida por cada órgano a un solo valor. La cantidad de radiación que recibirá en este estudio es inferior a la pauta de dosis establecido por el Comité de Seguridad Radiológica NIH para los sujetos de investigación. Esta pauta establece una dosis efectiva de 5 rem recibido por año.

Por comparación, la persona promedio en los Estados Unidos recibe una exposición a la radiación de 0,3 rem por año a partir de fuentes naturales, como el sol, el espacio exterior, y de materiales radiactivos que se encuentran naturalmente en el aire y el suelo. Si desea más información sobre la radiación y los ejemplos de los niveles y forma de exposicion a otras fuentes, por favor pregunte al investigador para obtener una copia del folleto titulado, An Introduction to Radiation for NIH Research Subjects.

3. **La extracción de sangre**. La cantidad de extracción de sangre es muy por debajo de la directriz del NIH para una cantidad segura de extracción de sangre (550 cc cada 8 semanas). Un pequeño moretón se puede formar en

cualquier sitio donde se toma la sangre. El riesgo de infección o desmayo es muy pequeña. La inflamación o coagulación de una vena también pueden ocurrir raramente.

Una parte de su sangre será enviado a otro laboratorio dentro del NIH para examinar sus niveles de inflamación. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras

- 4. **Recogida de muestras de heces** no tiene ningún riesgo, y sólo debe tomar un momento para recogerlas. Las muestras serán codificadas, y sólo los investigadores de este estudio tendrán acceso a la identidad de las muestras.
- 5. **La recogida de muestras de orina** no tiene ningún riesgo y sólo toma un momento para completar. Si el resultado es positivo para una sustancia ilícita, el resultado será parte de su expediente médico NIH.
- 6. **Los cuestionarios no son peligrosos**, pero pueden ser un inconveniente debido al tiempo necesario para su realización.
- 7. **Prueba oral de tolerancia a la glucosa**. Esta prueba es un inconveniente debido al tiempo que se tarda en completar. Los únicos riesgos de este tipo de estudio son las descritos para cualquier extracción de sangre, así como el desarrollo de las náuseas por la glucosa oral. Algunos pacientes pueden desarrollar de forma transitoria niveles altos de azúcar en la sangre a partir de la glucosa, pero deben normalizarse a las pocas horas y no deben ser clínicamente significativos.
- 8. **Prueba de tolerancia a la glucosa intravenosa**. Esta prueba es un inconveniente debido al tiempo que se tarda en completar. Usted puede ver la televisión durante esta prueba. Los únicos riesgos de este tipo de estudios son las descritas para cualquier extracción de sangre, la posibilidad de una ligera sensitividad en el brazo al recibir la infusión de azúcar, (esa sensitividad desaparece al cabo de unos minutos con el roce suave del brazo), y la posibilidad de un bajo nivel de azúcar en la sangre durante el estudio. Cuando la azúcar en sangre esta baja (menos de 50 mg/dl), los participantes pueden tener hambre, tener dolor de cabeza, sentirse

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

temblorosos o mareados o pueden llegar a ponerse sudorosos. Con azúcar en la sangre muy bajos (menos de 30 mg/dl) participantes pueden tener problemas para hablar, dificultad para despertar, e incluso tener convulsiones.

Sin embargo, en la prueba que estamos haciendo, le estaremos dando azúcar extra para elevar el azúcar en la sangre por encima de lo normal, y luego vamos a tratar de traerlo de vuelta a la normalidad (95-105 mg / dL) con insulina. Para ello, vamos a medir el azúcar en la sangre a los 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 24, 27, 30, 40, 50, 70, 90, 120, 140, 160, y 180 minutos (un total de 3 horas). Un médico o enfermera practicante estará presente durante la primera hora de su prueba para asegurarse de que todo funciona correctamente. Esperamos que la posibilidad de un nivel de azúcar en sangre bajo sea muy pequeña. Si un bajo nivel de azúcar en la sangre no sube por sí sola con rapidez, se detendrá la prueba y se le dará el azúcar por vía IV para elevar el azúcar en la sangre a la normalidad

9. **Biopsias de grasa.** Los posibles efectos secundarios de la biopsia son el dolor durante y durante dos o tres días después del procedimiento. Aunque rara vez, la zona de la biopsia puede estar sensible o adolorida o tener moretones o hinchazón durante 2-3 semanas. Heridas biopsia suelen sanar con una cicatriz muy pequeña, casi imperceptible, pero a veces una cicatriz elevada (queloides) o bulto visible puede resultar. Su riesgo es ligeramente mayor si usted es afroamericano. Inyección de lidocaína para adormecer antes de biopsias de grasa puede causar un poco de ardor suave antes de que llegue el entumecimiento. Efectos adversos raros incluyen la infección en los sitios de biopsia o una reacción alérgica a la lidocaína que puede llevar a una erupción y/o hinchazón de la zona de inyección. Si usted sabe que es alérgico a la lidocaína, cambiaremos a otro anestésico local. Otro de los riesgos del procedimiento es sangrado menor en el área de la biopsia. Algunos medicamentos

pueden aumentar la cantidad de sangrado de la biopsia. Si está tomando medicamentos como Coumadin, Plavix o aspirina para adelgazar la sangre, usted no tendrá una biopsia. Si está tomando aspirina o medicamentos no esteroides como Advil para el dolor tendrá que dejar de tomar estos medicamentos durante una semanaantes de realizar la biopsia.

- 10. **Tapa inteligente** no tiene riesgo, y debería funcionar igual que una tapa de botella regular.
- 11. **Medicamentos.** Los efectos adversos más comunes de los medicamentos utilizados en este estudio son: náuseas, vómitos, diarrea y dolor abdominal. Se han observado algunos efectos secundarios raros (<1%) son los siguientes: disminución de la producción de glóbulos rojos (que podría hacer que se sienta cansado), glóbulos blancos (que puede hacer más susceptibles a las infecciones), y/o plaquetas (que pueden hacerle más susceptibles a la aparición de moretones o sangrado), hormigueo (neuropatía), mareo, dolor muscular o debilidad, erupción, reacción alérgica, disminución del recuento de espermatozoides , y aumento de los niveles de enzimas hepáticas. Estos síntomas generalmente ocurren en personas con problemas médicos subyacentes, o estaban en ciertos medicamentos, que les predispone a tener la reacción. En general, estos síntomas se resolvieron dentro de una semana una vez que se suspende el medicamento. Aunque la colchicine se ha utilizado durante unos 2000 años para la gota, al igual que con cualquier medicamento, siempre existe la posibilidad de efectos secundarios imprevistos. Le supervisaremos por todos los efectos adversos. Si se desarrollan (severos) efectos adversos, vamos a disminuir la dosis, interrumpir temporalmente o suspender la medicación.

Si usted experimenta cualquiera de los siguientes efectos, póngase en contacto con nuestro equipo de inmediato:

- Debilidad muscular o dolor
- El entumecimiento u hormigueo en los dedos o dedos de los pies

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Sangrado o moretones inusuales

• La diarrea grave o vómitos

No hay estudios bien controlados adecuados sobre el uso de colchicine durante el embarazo. Los datos de un número limitado de estudios publicados no encontraron evidencia de un mayor riesgo de aborto involuntario, muerte, o efectos teratogénicos en las mujeres embarazadas que usan colchicina. Sin embargo, la colchicine mostró defectos de nacimiento en las crías de ratas embarazadas. Si usted cree que puede quedar embarazada, le pediremos que no participe en este estudio.

- Tomar ciertos medicamentos con colchicina puede hacer que subir demasiado su nivel de colchicina, especialmente si usted tiene problemas renales o hepáticos (consulte "Guía del Medicamento" para más información).
- Incluso los medicamentos que usted toma por un corto período de tiempo, tales como antibióticos, pueden interactuar con colchicina y causar efectos secundarios graves o la muerte. Por favor díganos acerca de cualquier medicamento que usted necesita tomar para que podamos asegurarnos de que puede seguir utilizando colchicina.
- Evite beber jugo de toronja, ya que puede interferir con la capacidad del cuerpo para desglosar colchicina

# Mantenga el medicamento fuera del alcance de los niños.

- 11. **Las pruebas de ADN.** Si nos permite estudiar su ADN, lo vamos a utilizar para la secuenciación del genoma. La secuenciación del genoma es una prueba que nos podrían dar diferentes tipos de resultados. Estos incluyen:
  - a. Podríamos identificar cambios en los genes que están relacionados con el metabolismo y el peso corporal.
  - b. Podríamos identificar cambios en los genes que contribuyen a otras enfermedades o problemas.
  - c. Podríamos identificar los cambios en los genes que no son conocidos por causar ninguna enfermedad. Estos son conocidos como variaciones normales.
  - d. Podríamos encontrar cambios en los genes que son nuevos y de importancia clínica incierta. Esto significa que no se sabe si podrían causar o contribuir a una enfermedad o si son variaciones normales.

No todos los cambios genéticos tendrán implicaciones para la salud de su familia. Los cambios en los genes que tienen implicaciones para la salud de su familia:

- 1. Ya han causado problemas de salud.
- 2. Pueden causar un problema de salud en el futuro.

Uno de los objetivos de este estudio es identificar los cambios en los genes que pueden estar implicados en la obesidad. Esta investigación puede tomar años. Sin embargo, si se identifica una causa genética o la causa probable de la obesidad, con su permiso, nos pondremos en contacto con usted. Por favor, háganos saber su preferencia con sus iniciales en una de estas dos declaraciones:

Me gustaría ser contactado con la información sobre los avances de este estudio y contactado acerca de cualquier resultado relacionado con la obesidad. Entiendo que esta investigación llevará años y que una anormalidad específica no se puede identificar en mí.

# MEDICAL RECORD NIH

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

Por favor no se contacte conmigo acerca de la marcha de este estudio o cualquier cambio de genes específicos relacionados con la obesidad.

Si detectamos un cambio genético que podría ser importante para usted, entonces vamos a tener que confirmar este resultado en un laboratorio certificado. Por esta confirmación, le pediremos una nueva muestra de ADN a usted. En la mayoría de los casos esto implicará la obtención de una pequeña muestra de sangre (1-2 cucharaditas). En algunos casos podemos obtener suficiente ADN para confirmar un cambio genético por limpiando el interior de la mejilla. Usted puede decidir, si desea hacerlo más adelante, si nos comunicamos con usted con la información de que hemos encontrado una posible diferencia genética importante.

La identificación de cambios genéticos que no están relacionados con la condición que se está estudiando, se conoce como información médica incidental.

Vamos a encontrar cambios genéticos en todo el mundo que estudiamos, pero estamos mirando sólo específicamente para los genes relacionados con el metabolismo y el peso corporal. No vamos a analizar su ADN para los cambios que no están relacionados con el metabolismo y el peso corporal. Aun así, algunos cambios en los genes no relacionados con el metabolismo y el peso corporal se detectarán.

Nosotros sólo le informaremos de los cambios que tienen importancia médica urgente y se beneficiarían de un tratamiento médico temprano. Un ejemplo de esto sería un cambio en el gen que causa cáncer y en la que se beneficiaría de la detección temprana. No le informará de todos los cambios en los genes que tienen inciertas implicaciones para la salud. Por ejemplo no vamos a informar de los cambios genéticos que predisponen a los individuos sólo a la enfermedad. Un ejemplo de esto sería un cambio en el gen que influye en el riesgo de enfermedades del corazón, pero en el que el desarrollo de la enfermedad depende de muchos factores genéticos y no genéticos (tales como la dieta y el tabaquismo). Si nos encontramos con un cambio en un gen que es importante para la salud de su familia, sólo le daremos los resultados si el cambio ha sido confirmado por un laboratorio certificado. Para asegurarse de que no se ha producido un error, tendríamos que obtener una nueva muestra de ADN a partir de que se confirmen los resultados experimentales.

Además de saber lo que encontramos, nos gustaría que conociera las limitaciones de la secuenciación del genoma y lo que no vamos a ser capaces de decirle acerca de los cambios que encontramos.

- 1. No todos los cambios en los genes que causan la enfermedad serán detectados.
- 2. Algunos de los cambios que no se conocen actualmente para causar problemas de salud podrían causar problemas de salud en el futuro. No podemos prometer tener la capacidad de decirle a usted acerca de esos cambios en el futuro.
- 3. No le dirá acerca de cambios en los genes que no se sabe que tienen consecuencias para la salud, ni vamos a informarle sobre cambios en los genes que sólo tienen consecuencias reproductivas.
- 4. Esta secuenciación de genes no puede ser sustituido por las pruebas de diagnóstico recomendado por otro médico.

Por favor, coloque sus iniciales en todas las siguientes declaraciones para indicar que usted entiende la medida en que le informaremos sobre los cambios genéticos accidentales que encontremos:

14-CH-0119

**MEDICAL RECORD** 

STUDY NUMBER:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

Entiendo, que voy a estar informado sólo de cambios genéticos que los investigadores implicados en este estudio piensen que son urgentemente importantes para la salud de mi familia y que el conocimiento de estos cambios tiene el potencial de un beneficio significativo para mí o mi familia.

> Entiendo que los investigadores no van a buscar específicamente cambios en los genes no relacionados con el metabolismo y el peso corporal, y que la identificación de otros genes que causan enfermedades sólo ocurrirá por casualidad dependiendo del análisis que se realiza.

CONTINUATION:  pages

Entiendo perfectamente que a pesar de que podrían tener consecuencias de salud o reproductivas, no se me hablará de todos los cambios genéticos identificados que no están relacionados con el metabolismo y el peso corporal.

Si se detecta <u>un cambio en el qen no relacionado con el metabolismo y el peso corporal</u> y los investigadores sentimos que cumple con los requisitos de tener importancia médica urgente para que usted se beneficie de un tratamiento médico, a continuación, se le dará la opción para aprender o no aprender acerca del cambio genético encontrado. Usted puede elegir no ser contactado en absoluto si esa es su preferencia. Una excepción a su capacidad de elegir si desea o no saber acerca de un cambio en un gen, sería un cambio en un gen que los investigadores consideran que es de vital importancia para su salud. Un ejemplo de esto sería un cambio en el gen que tiene una alta probabilidad de causar cáncer o una enfermedad para la cual el tratamiento temprano sería beneficioso. Antes de confirmar el resultado en un laboratorio clínico nos pondremos en contacto con usted para obtener una nueva muestra de ADN.

Si usted tiene un cambio en un gen con urgentes implicaciones para la salud, el NIH confirmará el cambio genético presente en uno de los miembros de su familia. Discutiremos los resultados con usted para que pueda saber si alquien más en su familia podría ser un portador de este mismo cambio. Podemos avudarle a organizar las pruebas que haya que hacer, pero el NIH no podemos prometer realizar o pagar por las pruebas clínicas necesarias para confirmar o determinar quién más en su familia puede tener este cambio en su ADN.

Una vez que se confirma un cambio en un gen, vamos a discutir los resultados con usted y hacer recomendaciones sobre apropiado sequimiento médico. El NIH no puede prometer realizar o pagar por los exámenes médicos recomendados o evaluaciones.

Es posible que un cambio genético no se confirmará en las pruebas posteriores. Esto podría ser debido a un error en la secuenciación de ADN o un error en el procesamiento del ADN o líneas celulares. Aunque es agradable para

| Ud. que no se confirme el problema, esto puede causar un p | , , , |
|---|---|
| no habría experimentado. | |
| Por favor, háganos saber sus preferencias colocando sus ini | ciales en una de las siguientes afirmaciones: |

| ., | cas en cas presente concessivo cas iniciares en ana de las elganemes animisationes. |
|---|---|
| | Yo QUIERO ser re-contactado si se descubren variantes genéticas con consecuencias urgentes para la salud, durante esta prueba de investigación. |
| | NO deseo volver a ser contactado si se descubren variantes genéticas con consecuencias urgentes para la salud durante esta prueba de investigación. Entiendo que una excepción a esta elección, como se describió anteriormente, se hará para un cambio en el gen de importancia médica fundamental. |

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: CONTINUATION:  pages 14-CH-0119

Riesgos emocionales y psicológicos de la prueba de ADN. La identificación de los cambios en los genes puede causar problemas emocionales y psicológicos. En algunas situaciones se podría recomendar asesoría psicológica.

- 1. Aprender sobre el riesgo de enfermedad que en su familia puede ser angustiante.
- 2. Aprender que algo que sucede en un gen suyo, puede no suceder en su hijo, puede ser angustiante.
- 3. Otros miembros de su familia podrían ponerse molestos al saber que ellos pueden estar en riesgo de un trastorno debido a su participación en este estudio.

Ud. Puede permanecer falsamente tranquilo acerca de su estado de salud si nosotros no le reportamos ningún cambio en su caso.

Otros riesgos de las pruebas genéticas. Si confirmamos un cambio genetico en su ADN en un laboratorio de diagnóstico, esta información será parte de su expediente médico en el NIH. Algunas personas se preocupan de que la información acerca de ellos de sus registros médicos podrían ser dadas a conocer. Posibles problemas incluyen el seguro o la discriminación laboral. Medidas para proteger la confidencialidad de su información se describen a continuación. Estos problemas también pueden ocurrir si usted divulga su propia información o acepta que sus registros de investigación sean liberados.

Hay leyes estatales y federales que protegen contra la discriminación genética. Una ley federal llamada la Ley de No Discriminación por información Genética (GINA), generalmente hace que sea ilegal que las compañías de seguros de salud, planes de salud de grupo, y la mayoría de los empleadores discriminen contra usted basado en su información genética. Según esta ley, las compañías de seguros de salud o planes de salud de grupo (hasta el 21 de mayo de 2010) no puede solicitar su información genética, o utilizarlo para tomar decisiones sobre su elegibilidad o primas; y los empleadores no pueden utilizarlo en la decisión de contratar, promover, ni puede despedirlo, o en el establecimiento de los términos de su empleo (a fecha de 21 de noviembre 2009).

Tenga en cuenta que esta ley federal no le protege contra la discriminación genética por las compañías que venden seguros de vida, seguro de invalidez, o un seguro de cuidado a largo plazo.

Este enlace contiene detalles sobre esta política:

PATIENT IDENTIFICATION

http://www.genome.gov/Pages/PolicyEthics/GeneticDiscrimination/GINAInfoDoc.pdf

Usted puede preguntar a su equipo de investigación para obtener información adicional o una copia de la Ley de Discriminación por Información Genética de 2008 documento informativo.

Los estudios genéticos pueden descubrir relaciones familiares inesperados. Por ejemplo, es posible que podamos enteramos de que un miembro de la familia no es el hijo biológico de los padres con los que él o ella vive (por ejemplo, debido a la adopción). No proporcionaremos normalmente este tipo de información a cualquier miembro de la familia o al médico de referencia. Sin embargo, podemos hacer excepciones en circunstancias extraordinarias si esta información se requiere para la atención médica de las personas involucradas. Si estamos convencidos de que esto es necesario, vamos a proporcionar la información al médico que proporciona la atención médica al paciente

P.A.: 09-25-0099

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### El uso de muestras almacenadas y datos

**Investigaciones futuras ADN**. Actualmente tenemos la intención de secuenciar los genes conocidos. Esto representa sólo alrededor del 1% de su secuencia de ADN. En el futuro podemos secuenciar otras partes de su ADN, y, finalmente, podemos secuenciar completamente su ADN. Estos estudios adicionales pueden ocurrir años a partir de ahora. Algunas partes de su ADN pueden ser enviadas a otros laboratorios para pruebas específicas. Si esto se hace el ADN será codificado y no tendrá su nombre en la muestra o en el papeleo que va al laboratorio. En caso de retirarse de este estudio, vamos a mantener su ADN para el análisis a menos que usted nos pida destruir las muestras de AND.

ADN puede ser utilizado para otros tipos de futuras investigaciones relacionadas con la salud. Esta investigación no se limita a los estudios relacionados con la obesidad, el metabolismo y el peso corporal. Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. Autorizo el uso de estas muestras sin mi consentimiento adicional. Entiendo que no se pondrán en contacto si se utilizan estas muestras en el futuro.

Entiendo que las muestras genéticas recogidas durante estas visitas NIH serán guardados y utilizados para futuras pruebas experimentales relacionadas con la obesidad, el metabolismo y el peso corporal. Esta prueba puede realizarse por laboratorios de investigación que no se encuentran en el NIH. NO autorizo el uso de estas muestras para ningún otro fin sin mi consentimiento adicional. Debo ser contactado y dar consentimiento si estas muestras se van a utilizar en el futuro.

No utilice mi ADN para futuros estudios más allá de los descritos anteriormente en este formulario de consentimiento.

Por favor, coloque su inicial en una de las siguientes tres declaraciones relativas a la investigación futura:

**Futuras investigaciones con muestras de sangre**. Nuestros planes específicos de investigación se han resumido en este formulario de consentimiento. En el curso de la investigación, vamos a obtener muestras de sangre. Si bien podemos hacer algunas de nuestras pruebas de inmediato, es posible que desee almacenar sus muestras de sangre en el congelador para futuros estudios. Además, cierta información se almacenará en su expediente médico. En el futuro, es posible que sus muestras de sangre o registros médicos serán utilizados para otros fines de investigación que no se describen específicamente en este formulario de consentimiento. Si se hace esto, las muestras serán codificadas, y no serán identificados por su nombre. Estas muestras pueden ser almacenadas en un lugar separado (llamado un repositorio) que se especializa en el almacenamiento de muestras clínicas. Usted tiene la opción, en el futuro, de solicitar que estas muestras no se utilicen para hacer más ensayos. Además, es posible que alguna información obtenida de estos estudios serán publicados en la literatura médica. Sin embargo, su identidad no será incluida en cualquier publicación.

# CONTINUATION SHEET for either: MEDICAL RECORD NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

| 31001 | IT CIT UITS | | continuation: pa | ige 11 of 17 pages | |
|---|---|---|---|---|---|
| | Por favor, coloque su inicial en <u>ı</u> | <u>una</u> de las dos afirmacio | nes siguientes: | | |
| | ensayos experimentales realizarse por laboratori | ras recogidas durante es<br>relacionados con el pes<br>os de investigación que<br>onsentimiento adicional.<br>turo. | o corporal, y/o el met<br>no se encuentran en e | abolismo. Esta prueba p<br>el NIH. Autorizo a otros | ouede<br>usos de |
| | realizarse por laboratori | relacionados con el pes<br>os de investigación que<br>sin mi consentimiento ad | o corporal, y/o el met<br>no se encuentran en e | abolismo. Ésta prueba p<br>el NIH. NO autorizo cual | ouede<br>Iquier otro |
| | Durante todo el proceso de estu<br>uso de códigos y números de hi<br>personal médico involucrado en<br>exámenes, y los números de có | storia clínica en la graba<br>este estudio tendrán ac | ción de su información | n y resultados de prueb | as. Sólo el |
| | Usted tiene que ser consciente on nformación de la secuencia de ADN. Para facilitar la investigacion pases de datos. En este caso, a que no permita que alguien le iduez que se deposita. | ADN está disponible, alg<br>ón genética, la informac<br>menos que tengamos si | uien podría identificar<br>ión de su secuencia do<br>u permiso, vamos a de | lo a Ud. en base a su se<br>e ADN se puede deposit<br>epositar los datos de un | ecuencia de<br>car en otras<br>a manera |
| Por fav | r, coloque su inicial en <u>una</u> de la | as siguientes casillas: | | | |
| | | este estudio.<br>5 de ADN pueden ser de <sub>l</sub><br>ovestigadores aprobados | positados en las bases<br>Ina base de datos que<br>lel IRB de estudios de | de datos que limitan el<br>está disponible sólo pa | l acceso a la<br>ra los |

# Los beneficios potenciales de la participación

Tenemos la esperanza de que su participación en este estudio proporcionará pruebas acerca de si la colchicina ayudará parámetros metabólicos en individuos obesos. Sin embargo, no puede beneficiarse directamente de participar en este estudio. Al encontrar anomalías en cualquiera de sus resultados de la prueba, se le notificará y recibirá una copia para ayudarle en la búsqueda de una mayor evaluación médica. Esta información puede o no mejorar su salud.

# MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

## Derecho de revocación y Condiciones de retiro anticipado

Usted puede retirarse del estudio en cualquier momento y por cualquier motivo y sin pérdida de beneficios o privilegios a los que tiene derecho.

#### La discusión de los nuevos hallazgos con usted

Después de que todos los participantes hayan completado el estudio, se le informará sobre cual medicina tomó y una vez que el estudio esté totalmente analizado, le permiten saber si la colchicina puede ayudar con la inflamación y la resistencia a la insulina. No hay plan general para compartir los resultados de sus pruebas individuales con usted. Sin embargo, si algún hallazgo sugiere que tiene un problema médico, vamos a proporcionar esta información a usted y a su proveedor de atención primaria. Usted puede solicitar una copia de sus pruebas de laboratorio de rutina si lo desea.

## **Terminación de Estudios**

Se le puede pedir terminar su participación en este estudio en cualquier momento, si creemos que la continuación en él no es lo mejor para su interés médico o si no puede cumplir con los requisitos del estudio.

## Alternativas a la Participación

La alternativa a este estudio es no participar. Usted puede ser elegible para otros estudios en los NIH. Usted puede aprender más sobre ellos a través de www.clinicaltrials.gov.

#### Compensación

Usted será compensado por el tiempo y los inconvenientes asociados a la participación según las directrices de compensación para voluntarios de investigación del NIH. La compensación para completar todas las pruebas que se han descrito anteriormente es: \$100 por la visita de selección de pacientes ambulatorios, \$50 por la visita de seguridad, y de \$300 por cada una de las visitas inicial, final y la opcional. La cantidad total que usted podría recibir por la participación si completa todas las partes de este estudio es de \$1050.

#### **Conflicto de intereses**

El NIH y los miembros de este equipo de investigación no tienen ningún interés financiero en relación con este estudio de investigación.

Publicación de Resultados de Investigación en: www.ClinicalTrials.gov

Una descripción de este ensayo clínico estará disponible en http://www.Clinicaltrials.gov, como lo requiere la ley de Estados Unidos. En esta pagina de web no incluirá información que pueda identificarlo. En la mayor parte del sitio Web incluirá un resumen de los resultados. Usted puede buscar en este sitio web en cualquier momento.

| He recibido una copia del formulario de consent | imiento firmado. |
|-------------------------------------------------|------------------|
|-------------------------------------------------|------------------|

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

**MEDICAL RECORD** 

Adult Patient or Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

#### INFORMACIÓN PERTINENTE ADICIONAL

**1. Confidencialidad**. Cuando los resultados de un estudio de investigación del NIH se dan a conocer en revistas médicas o reuniones científicas, no se menciona la identidad de los participantes. En la mayoría de los casos, el NIH no divulgará ninguna información sobre su participación en la investigación a menos que usted otorgue su permiso por escrito. No obstante, si usted firma una autorización de divulgación de información, por ejemplo, a una empresa aseguradora, el NIH le proporcionará a ésta información de su expediente médico. Esta información podría influir (en forma favorable o desfavorable para usted) la disposición de la aseguradora a venderle el seguro.

La Ley Federal de Protección de la Vida Privada (Federal Privacy Act) protege el carácter confidencial de sus expedientes médicos en el NIH. Sin embargo, es importante que sepa que esta ley permite la divulgación de cierta información de su expediente médico sin su autorización, por ejemplo, si lo solicitan la Administración de Alimentos y Medicamentos (FDA), los miembros del Congreso, los agentes encargados del cumplimiento de la ley o las organizaciones autorizadas para efectos de acreditación hospitalaria.

- **2. Normas sobre lesiones relacionadas con la investigación**. El Centro Clínico le dará atención médica a corto plazo para cualquier lesión que se deba a su participación en una investigación que se realice allí. En general, ni los Institutos Nacionales de Salud, ni el Centro Clínico, ni el gobierno federal le darán atención médica a largo plazo ni indemnización económica por lesiones relacionadas con la investigación. Sin embargo, usted tiene derecho a buscar una compensación legal si cree que la lesión justifica dicha medida.
- **3. Pagos**. El monto del pago que reciben los voluntarios de investigación se rige por las normas de los Institutos Nacionales de Salud. En general, a los pacientes no se les paga por participar en los estudios de investigación en los Institutos Nacionales de Salud. Se le ofrecerá el reembolso de gastos de viaje y viáticos según las pautas del NIH.
- **4. Problemas o preguntas**. Si hay algún problema o usted tiene una pregunta con respecto a este estudio, a sus derechos como participante en un estudio de investigación clínica o a cualquier lesión relacionada con la investigación, debe comunicarse con el Investigador Principal, Jack A. Yanovski, MD, PhD; Building (Edificio) 10, Room (Sala) 1-3330, Teléfono: (301) 496-4686 o el Investigador Asociado Principal, Andrew Demidowich, MD; Building 10, Room 1-3330, Teléfono: (301) 496-4686.

También puede llamar al representante de los pacientes del Centro Clínico, al teléfono (301) 496-2626.

**5. Documento de consentimiento.** Le sugerimos que conserve una copia de este documento para consultarla posteriormente.

**PATIENT IDENTIFICATION** 

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

# **MEDICAL RECORD**

#### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 14-CH-0119 CONTINUATION:  pages

| COMPLETE LAS CASILLAS CORRESPONDIENTES A CONTINUACION: | |
|---|---|
| A. Consentimiento de un paciente adulto. He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo mi consentimiento para participar en este estudio. | B. Permiso otorgado por el (los) padre(s) de un paciente menor de edad. He leído la explicación relacionada con este estudio y he tenido la oportunidad de comentarla y hacer preguntas. Por este medio otorgo permiso para que mi hijo participe en este estudio. (Anéxese el formulario NIH 2514-2, Asentimiento de un menor de edad, si corresponde.) |
| Firma del paciente adulto o su representante legal Fecha | Firma del (los) padre(s) o del tutor legal Fecha |
| Nombre en letra de imprenta | Nombre en letra de imprenta |
| C. Asentimiento verbal de un niño (si corresponde) Se le explicó a mi hijo la información contenida en el presente documento y | mi hijo está de acuerdo en participar en el estudio. |
| Firma del (los) padre(s) o del tutor legal Fecha | Nombre en letra de imprenta |
| EL USO DE ESTE DOCUMENTO DE CONSENTIMIENTO ESTÁ APROBADO<br>DESDE EL 24 DE ENERO DE 2018 HASTA EL 24 DE FEBRERO DE 2019. | |
| Firma del Investigador Fecha | Firma del testigo Fecha |
| Nombre en letra de imprenta | Nombre en letra de imprenta |

• Adult Patient or • Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

File in Section 4: Protocol Consent